

# Cover Page

**Official title:** A phase 3 trial comparing the efficacy and safety of LEO 90100 aerosol foam with the aerosol foam vehicle used twice weekly as long-term maintenance therapy in subjects with psoriasis vulgaris.

**LEO Pharma number:** LP0053-1004

NCT number: NCT02899962

Date: 15-Jul-2019

| Trial ID: <b>LP0053-1004</b> | Date: 15-JUL-2019 | Version: 1.0 |
|------------------------------|-------------------|---------------|

# Statistical Analysis Plan

# LEO 90100 twice weekly maintenance regimen for psoriasis vulgaris

A phase 3 trial comparing the efficacy and safety of LEO 90100 aerosol foam with the aerosol foam vehicle used twice weekly as long-term maintenance therapy in subjects with psoriasis vulgaris.

A 12-month, international, multi-centre, randomised, vehicle controlled, double-blind, 2-arm, parallel group trial.

| LEO Pharma A/S | Trial ID: | LP0053-1004 |
|----------------|-----------|-------------|
| | Date: | 15-JUL-2019 |
| | Version: | 1.0 |



|------------------------------|-------------------|---------------|

# 1 Statistical Analysis Plan Approval

# 1.1 Approval Statement

QC Statistician, Biostatistics

On behalf of LEO, the Biostatistics Lead and the Medical Lead, are authorised to approve the Statistical Analysis Plan Update.

The QC statistician has by approving this document confirmed that the statistical information has been subject to statistical quality control.

The following persons have approved this Statistical Analysis Plan Update using electronic signatures as presented on the last page of this document.

| PPD | |
|--------------------|------------------------------|
| Biostatistics Lead | , Global Clinical Operations |
| PPD | |
| Medical Lead, Me | edical Science |
| PPD | |



|------------------------------|-------------------|---------------|

# 2 Statistical Analysis Plan Statements

# 2.1 Compliance with Good Clinical Practice

This Statistical Analysis Plan Update is designed to comply with the standards issued by the International Conference on Harmonisation (ICH) (E3: Structure and Content of Clinical Study Reports, E6: Good Clinical Practice, and E9: Statistical Principles for Clinical Trials).



# **Table of Contents**

| 1 Statistical Analysis Plan | Approval | 2 |
|---|---|---|
| 1.1 Approval Statement | | 2 |
| ** | Statements | |
| - | | |
| | nical Practice | |
| Table of Contents | | 4 |
| 3 List of Abbreviations | | ( |
| 4 Introduction | | - |
| • | | |
| 5.1 Definition of trial periods | | |
| 5.2 Trial Analysis Sets | | 8 |
| 5.3 Baseline Considerations | | 9 |
| 5.3.1 Baseline definition | | ٥ |
| 5.3.2 Disposition of subjects | | 9 |
| 5.3.3 Demographics | | 9 |
| 5.3.4 Compliance | | ( |
| 5.4 Analysis of Efficacy | 1 | ( |
| 5.4.1 Primary Efficacy Endpoi | nt | ( |
| 5.4.2 Secondary Efficacy Endp | points | 2 |
| 5.4.2.1 Proportion of days in a | emission1 | 2 |
| 5.4.2.2 Number of relapses du | ring maintenance phase | ( |
| * | 1 | |
| • | still at risk of first relapse at week 26 and week 52 | |
| | 1 | |
| | sessment of Disease Severity | |
| • | at each visit | |
| | is no longer fulfilled | |
| _ | ecording to m-PASI | |
| | it of relapse | |
| | scores | |
| • | mont days during maintenance phase | |
| | ment days during maintenance phase | |
| J.T.T I anom-Nepolica Gulcon | 100 L | . ' |



| 5.4.4.1 Dermatology Life Quality Index (DLQI) | 21 |
|---------------------------------------------------------------------|----|
| 5.4.4.2 EQ-5D-5L-PSO | 24 |
| 5.4.4.3 WPAI:PSO | 26 |
| 5.4.4.4 Psoriasis Symptom Inventory | 26 |
| 5.4.4.5 Subject's Global Assessment of Disease Severity (SGA) | 28 |
| 5.5 Analysis of Safety | 29 |
| 5.5.1 Exposure | 29 |
| 5.5.2 Drug Accountability | 30 |
| 5.5.3 Adverse Events | 30 |
| 5.5.3.1 Adverse events associated with long term corticosteroid use | 32 |
| 5.5.4 Rebound | 33 |
| 5.5.5 Physician's Assessment of Local Safety and Tolerability | 33 |
| 5.5.6 Subject's Assessment of Local Safety and Tolerability | 34 |
| 5.5.7 ACTH-Challenge Test | 34 |
| 5.5.8 Vital Signs and Physical Findings | 35 |
| 5.5.9 Laboratory Data | 36 |
| 5.6 General Principles | 37 |
| 5.6.1 Pooling of Trial Sites | 37 |
| 5.6.2 Handling of Drop-outs and Missing Values | 38 |
| 5.6.3 Incomplete dates | 38 |
| 5.6.4 Multiplicity adjustment | 38 |
| 5.6.5 Treatment Labels | 39 |
| 5.7 Changes to the analyses described in the protocol | 40 |
| Appendix I | 47 |
| Appendix II | 67 |
| ± ± | |



|------------------------------|-------------------|---------------|

#### 3 List of Abbreviations

ACTH Adrenocorticotropic Hormone

AE Adverse Event

ATC Anatomical Therapeutic Chemical

BSA Body Surface Area

CPM Clinical Project Manager

CPMP Committee for Proprietary Medicinal Products

CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organisation

DK Denmark

DLQI Dermatology Life Quality Index

eCRF Electronic Case Report Form

eDiary Electronic Diary

EU European Union

GCP Good Clinical Practice

ICH International Conference on Harmonisation

IEC Independent Ethics Committee

IMP Investigational Product

IRB Institutional Review Board

m-PASI Modified Psoriasis Area Severity Index

MedDRA Medical Dictionary for Regulatory Activities

MMRM Mixed effect Model Repeat Measurement

ML Maximum Likelihood

PASI Psoriasis Area Severity Index

PASI 75 A 75% reduction in the modified Psoriasis Area Severity Index

PGA Physician's Global Assessment of Disease Severity

PRO Patient Reported Outcome

PSI Psoriasis Symptom Inventory

REML Restricted Maximum Likelihood

SAE Serious Adverse Event



|------------------------------|-------------------|---------------|

| SAP | Statistical Analysis Plan |
|-----|-------------------------------------------------|
| SD | Standard Deviation |
| SGA | Subject's global assessment of disease severity |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| UNS | Unscheduled Visit |

## 4 Introduction

The statistical analysis will be performed as outlined in the Clinical Trial Protocol including amendments. This statistical analysis plan, prepared before the unblinding of the trial, but after the blind review of the data, contains a more technical and detailed elaboration of some points in the statistical analysis described in the Clinical Trial Protocol. Deviations from the planned data presentation and analysis are also described in section 5.7. Furthermore, the analysis sets, which are to be used for the statistical analysis, are presented.

# 5 Statistical Analysis

# 5.1 Definition of trial periods

The trial periods are defined in Table 1.

**Table 1: Definition of trial periods** 

| Trial period | Definition |
|---|---|
| Open-label phase | From the day of enrolment to the day before randomisation. |
| Randomised phase | From the day of randomisation to end of trial, both days included. |
| Maintenance phase | From the day of first exposure to maintenance IMP to the last day of |
| | exposure (rescue or maintenance IMP), both days included. |
| Follow-up phase | From the day after last application of maintenance or rescue IMP to end of trial. |
| Relapse period | Relapse is defined as a PGA score of at least 'mild' during the |
| | maintenance phase, for details on relapse see CTP section 6.14.1. A |
| | relapse period is defined from the relapse start day (included) to the |



|------------------------------|-------------------|---------------|

| | visit date when relapse treatment is discontinued (not included). |
|---|---|
| Remission period | A remission period is a period where the subject is not in a relapse period within the maintenance phase. |
| Visit interval | The interval between two successive scheduled visits. |

# **5.2** Trial Analysis Sets

The trial analysis sets are defined in Table 2. The analysis sets are described in more detail in the Analysis Set Definition Document.

**Table 2: Trial analysis sets** 

| Analysis set | Definition |
|---|---|
| Enrolled subjects | All subjects enrolled (informed consent obtained) in the trial. |
| Open-label safety analysis set | All subjects exposed to LEO 90100 during the open-label phase. |
| Open-label HPA<br>analysis set | All subjects in the open-label safety analysis set who provided consent for the Adrenocorticotropic Hormone (ACTH) challenge test and underwent a Hypothalamic-Pituitary-Adrenal (HPA) axis test. |
| Full analysis set | All subjects randomised who had treatment success at randomisation, defined as PGA score of 'clear' or 'almost clear' with at least a 2-grade improvement from baseline. Subjects randomised without treatment success will be excluded from the full analysis set. This approach is in alignment with the ICH E9, since achieving treatment success is a major randomisation criterion measured prior to randomisation and therefore exclusion of such subjects will not introduce bias. |
| Per protocol<br>analysis set | The per protocol analysis set will be defined by excluding subjects from the full analysis set as described in the protocol and in the Analysis Set Definition Document. |
| Safety analysis | All subjects exposed to IMPs following randomisation and with available |



|------------------------------|-------------------|---------------|

| set | post-randomisation safety evaluations. |
|---|---|
| Randomised subjects | All subjects randomised to the maintenance phase. |
| HPA analysis set | All subjects in the safety analysis set who provided consent for the ACTH challenge test and underwent an HPA axis test. |

#### **5.3** Baseline Considerations

#### **5.3.1** Baseline definition

As described in the protocol, baseline is defined as the measurement taken at screening or visit 1.

The maintenance phase baseline is defined as the last available measurement collected at randomisation (visit 2).

Baseline for rebounds will be handled differently as described in section 5.5.4.

# 5.3.2 Disposition of subjects

The reason for leaving the trial will be presented as described in the protocol.

In addition, cumulative incidence plots of discontinuation by reason for withdrawal will be done for subjects leaving the trial during the open-label phase or the maintenance phase, respectively. The plots for the maintenance phase will be presented by treatment group.

Further details for the tables can be found in Appendix I and Appendix II.

# **5.3.3** Demographics

Demographics and other baseline characteristics will be presented as described in the protocol. Age groups (18-64, >=65) will also be presented for all enrolled subjects and for all randomised subjects by treatment group.

More details for tables for demographics and other baseline characteristics are given in Appendix I and Appendix II.



|------------------------------|-------------------|----------------|

# 5.3.4 Compliance

For the open-label treatment phase, number of subjects in non-compliance with treatment instructions together with percentage of missed daily applications of IMP will be summarised for the open-label safety analysis set.

For the maintenance phase, number of subjects in non-compliance with maintenance treatment instructions (i.e.; excluding relapse periods) will be summarised by treatment group both for each visit interval and for the total maintenance phase for the safety analysis set. The compliance information will be assigned to the visit interval by collection date.

For the relapse periods, number of subjects in non-compliance with rescue treatment instructions and percentage of missed daily applications of rescue IMP will be summarised by treatment group for the safety analysis set.

For an overview of changes as compared to the protocol refer to section 5.7.

## 5.4 Analysis of Efficacy

The assessment of efficacy is done for the maintenance phase. The primary and secondary efficacy endpoints will be analysed for the full analysis set, with the analyses for the per protocol analysis set being supportive. Sensitivity analyses are done for the full analysis set. Trial sites will be pooled as described in section 5.6.4 and will be referred as pooled sites.

# 5.4.1 Primary Efficacy Endpoint

The primary endpoint will be analysed using a cox proportional hazards model with treatment group, pooled sites, and disease severity at maintenance baseline (as determined by the PGA) as factors. Maintenance baseline is used in the model as compared to baseline at visit 1. See section 5.7 for details regarding changes as compared to the protocol.

The survival curves will be estimated using the Kaplan-Meier estimator. A log-log transformation will be applied to the survival function to obtain the pointwise confidence intervals in addition to the confidence intervals for the percentiles of the estimated survival times. The estimated survival curves and the confidence limits will be shown graphically. The percentiles of the estimated survival distribution and 95% confidence limits for the percentiles will be tabulated by treatment group.



|------------------------------|-------------------|----------------|

Number of subjects still at risk of first relapse at timepoints for scheduled visits will be summarised by treatment group.

Further details for tables, figures and listings for the primary endpoint are given in Appendix I and Appendix II.

#### Sensitivity analysis:

In the sensitivity analysis the primary endpoint will be analysed incorporating interval censoring. We will consider three different types of censoring. Subjects who do not encounter a relapse during the trial and subjects who are withdrawn from the trial in the maintenance phase before having a relapse will be right-censored, and the number of days will be treated as a censored observation at the end date of the maintenance phase. Subjects who are confirmed to have a relapse at a scheduled visit are interval censored, and it is assumed that the start of the relapse is between the scheduled visit where the relapse is confirmed and the previous visit where PGA was measured for the subject. For subjects who are confirmed to have a relapse at an unscheduled visit, it is assumed that the relapse starts on the day of this visit. These subjects are assumed to have exact observations. More details are given in Table 3.

The number of subjects without relapse, the number of subjects with relapse confirmed at a scheduled visit, and the number of subjects with relapse confirmed at an unscheduled visit will be summarised by treatment group.

Table 3: Censoring in the sensitivity analysis of primary endpoint

| Relapse | Censoring | | Lower | Upper |
|---|---|---|---|---|
| information | type | Observation type | endpoint | endpoint |
| No relapse | Right-<br>censored | (x, . ], where x is the day the subject completed the trial or withdrew from the trial, and . denotes that this is left missing | х | (missing) |
| Relapse confirmed at scheduled visit | Interval censored | (x, y], where x is the day of the previous visit in which PGA was measured, without relapse, and y is the day of the visit, where relapse is confirmed | х | у |
| Relapse confirmed at unscheduled visit | Exact observation | [x, x], where x is the day of the visit where relapse is confirmed | Х | х |



|------------------------------|-------------------|----------------|

In the sensitivity analysis, time to first relapse during the maintenance phase will be analysed using a proportional hazards model with treatment group, pooled sites, and disease severity at maintenance baseline (determined by the PGA) as factors. The model will incorporate interval censoring. The baseline hazard function is assumed to be a piecewise constant function within ten disjoint intervals. The ten intervals split the time axis such that each interval contains approximately equal number of unique boundary values and imputed middle points. The estimate of the hazard ratio of active treatment group relative to vehicle group together with the 95% confidence interval and p-value will be presented.

Furthermore, survival curves will be estimated using a non-parametric maximum likelihood estimator, namely the Turnbull self-consistency algorithm. Standard errors will be computed using multiple imputation with 1000 samples (seed=39506291). A log-log transformation will be applied to the survival function to obtain the pointwise confidence intervals in addition to the confidence intervals for the percentiles of the estimated survival times. The estimated survival curves and the confidence limits will be shown graphically. The percentiles of the estimated survival distribution and 95% confidence limits for the percentiles will be tabulated by treatment group.

This sensitivity analysis was not specified in the protocol. See section 5.7 for details regarding changes as compared to the protocol.

Further details for tables, figures and listings for the sensitivity analysis are given in Appendix I and Appendix II.

# 5.4.2 Secondary Efficacy Endpoints

Adjustment for multiplicity will be done as described in the protocol. Further details can be found in section 5.6.4.

# **5.4.2.1** Proportion of days in remission

The endpoint is the proportion of days in remission as compared to the number of days in remission described in the protocol section 11.3.3.5. Analysis and sensitivity analysis are also different as compared to the protocol. See section 5.7 for details regarding changes to the protocol.

The number of days in remission will be calculated as the sum of days where the subject is in remission periods as defined in Table 1. The proportion of days in remission will be calculated



|------------------------------|-------------------|----------------|

as the number of days in remission divided by the length of the maintenance phase in days. The proportion of days in remission will be summarised by treatment group.

#### Multiple imputation:

Multiple imputation of data for withdrawn subjects will be done using 100 imputations (seed=20910158). In order not to favour any treatment arm, the imputation approach will depend on whether the subject's reason for withdrawal potentially is related to IMP or not.

For the imputation, the length of the maintenance phase is assumed to be 52 weeks, corresponding to 364 days.

Imputation for subjects withdrawn with reasons 'withdrawal by subject' or 'lost to follow up': This approach assumes that the unobserved remission pattern for withdrawn subjects will be like the pattern observed for subjects in the same treatment group completing the maintenance phase. An example can be found in Figure 1 and the described below.

Figure 1: Example of imputation for a subject withdrawing from trial due to lost to follow-up or withdrawal by subject



#### Imputation steps:

1. For a withdrawn subject the 'number of unobserved days' will be computed as 364 minus the length of the subject's maintenance phase. This 'number of unobserved days' (e.g.; 64) will be used in step 2.



|------------------------------|-------------------|----------------|

- 2. For the sub-set of subjects, that are in the same treatment group as the withdrawn subject and completed their maintenance phase, the proportion of days in remission will be calculated for the last part in their maintenance phase lasting 'number of days unobserved' (e.g.; 64).
- 3. A single proportion of days in remission will be randomly sampled from the proportions calculated in step 2. This will be called the 'sampled proportion' (e.g.; 95%)
- 4. For the withdrawn subject, the number of days in remission for the missing period will be estimated by multiplying the 'sampled proportion' by the 'number of unobserved days' (e.g.; 0.95\*64).
- 5. For the withdrawn subject, the proportion of days in remission will be calculated by summing the observed number of days in remission and the estimated number of days in remission (from step 4) and dividing by 364.
- 6. Steps 1 to 5 will be repeated 100 times for each withdrawn subject to form 100 complete datasets.

Imputation for subjects withdrawn with reasons 'adverse event', 'death', 'lack of efficacy', or 'subject not achieving clear or almost clear after treatment of relapse':

This approach assumes that the unobserved part of the trial for subjects withdrawn due to these reasons, would have been similar to the observed part of the trial for the subjects withdrawing for the same four reasons regardless of treatment arm. An example can be found in Figure 2 and described in the imputation step below.

#### Imputation steps:

- 1. For a withdrawn subject the 'number of unobserved days' (e.g.; 64) will be computed as 364 minus the length of the subject's maintenance phase.
- 2. For the sub-set of subjects withdrawn due to 'adverse event', 'death', 'lack of efficacy', or 'subject not achieving clear or almost clear after treatment of relapse', the proportion of days in remission will be calculated.
- 3. A single proportion of days in remission will be randomly sampled from the proportions in step 2. This will be called the 'sampled proportion' (e.g.; 50%)



|------------------------------|-------------------|----------------|

- 4. For the withdrawn subject, the number of days in remission for the missing period will be estimated by multiplying the 'sampled proportion' by the 'number of unobserved days' (e.g.; 0.50\*64).
- 5. For the withdrawn subject, the proportion of days in remission will be calculated by summing the observed number of days in remission and the estimated number of days in remission (from step 4) and dividing by 364.
- 6. Steps 1 to 5 will be repeated 100 times for each withdrawn subject to form 100 complete datasets.

Figure 2: Example of imputation for a subject withdrawing from trial due to AE, death, lack of efficacy, or subject not clear or almost clear after treatment of relapse



#### Imputation for subjects leaving the trial due to other reasons:

For cases with withdrawal reason specified as 'Other', the details will be revised on a blinded manner, selecting and documenting the imputation approach in the Analysis Set Definition Document.

#### Statistical analysis:

For each of the 100 complete data sets, the difference in proportion of days in remission between treatment groups will be analysed by means of an analysis of variance (ANOVA) model as described in the protocol section 11.3.3.5. The estimates and standard errors from



|------------------------------|-------------------|----------------|

the 100 analyses will be pooled to one estimated treatment difference and associated standard error using Rubin's rule to draw inference. From these pooled estimates, the 95% CI for the treatment difference will be calculated. The p-value for treatment difference will be calculated using a two-tailed Student's t-test based on the pooled estimates.

A histogram with a density curve of proportion of days in remission by treatment group will be presented.

Number of days in remission between relapses will be plotted by treatment group.

#### Sensitivity analysis:

An additional sensitivity analysis will be performed assuming that after the subjects withdrew the pattern of remission will be as if the subject was not treated. This will be done as described above, however in step 2 of the sub-set of subjects will be subjects treated with vehicle.

Further details for tables, figures and listings are given in Appendix I and Appendix II.

# 5.4.2.2 Number of relapses during maintenance phase

The number of relapses will be analysed using a Poisson regression model with treatment group, pooled sites, and disease severity at maintenance baseline as factors, subject as random effect, and time at risk as an offset. REML will be used for estimation. Maintenance baseline is used in the model as compared to baseline at visit 1. See section 5.7 for details regarding changes as compared to the protocol.

Number of relapses will be summarised by treatment group. Rates (number of relapses divided by patient years of exposure multiplied by 100) will also be presented.

In addition, the distribution of the relapse rate by treatment group will be presented.

#### Sensitivity analysis:

The number of relapses will be analysed with a negative binomial regression model with treatment group, pooled sites, and disease severity at maintenance baseline as factors, subject as random effect, and time at risk as an offset. REML will be used for estimation. The purpose of this sensitivity analysis is to account for potential overdispersion in data, which is not adjusted for in the Poisson model.

See section 5.7 for details regarding changes as compared to the protocol.



|------------------------------|-------------------|----------------|

More details for the tables and listings can be found in Appendix I and Appendix II.

# **5.4.3** Exploratory Assessments

The exploratory assessments collected in the maintenance phase will be summarised for the full analysis set and the exploratory assessments collected in the open-label phase will be summarised for the open-label full analysis set. For all exploratory assessments the observations at visit 2 will be used for the purpose of summarising the change from visit 1 in the open-label phase.

# 5.4.3.1 Proportion of subjects still at risk of first relapse at week 26 and week 52

In section 11.3.3.3 of the protocol on the analysis of the primary endpoint, it is described that the proportion of subjects still at risk for a first relapse will be compared between the two treatment groups at 26 weeks and 52 weeks after randomisation. This will be considered as two explorative endpoints on its own. The comparison will be done by using an unpaired z-test. In addition, a binomial test will be done. The proportions and the corresponding standard errors will be obtained from the estimated survival curves for the primary endpoint. The estimates of proportions, the 95% confidence intervals and p-value will be presented.

More details for the tables and listings can be found in Appendix I and Appendix II.

#### 5.4.3.2 m-PASI

#### Open-label phase:

m-PASI will be summarised by visit. Change and percent change in m-PASI from visit 1 to visit 2 will also be summarised.

#### Maintenance phase:

m-PASI when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment group.

m-PASI collected when the subject is initiating a relapse period will be summarised by visit and visit intervals and by treatment group.

m-PASI collected when the subject is ending a relapse period will be summarised by visit and visit intervals and by treatment.



|------------------------------|-------------------|----------------|

Change and percent change in m-PASI from start of relapse to end of relapse will be summarised by visit for start of relapse and by treatment group.

m-PASI collected at visits where the subject is in a relapse period, will be listed only.

See section 5.7 for details regarding changes as compared to the protocol.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.4.3.3 Physician's Global Assessment of Disease Severity

#### Open-label phase:

Physician's global assessment of disease severity (PGA) will be summarised by visit. A shift table for categories of PGA at visit 1 versus the category at visit 2 will also be done.

#### Maintenance phase:

PGA collected when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment group.

PGA collected when the subject is initiating a relapse period will be summarised by visit and visit intervals and by treatment group.

PGA collected when the subject is ending a relapse period will be summarised by visit and visit intervals and by treatment group.

A shift table for categories of PGA at start of relapse versus the category at end of relapse will also be done by visit for start of relapse and by treatment group.

PGA collected at visits in the maintenance phase, when the subject is in a relapse period will be listed only.

See section 5.7 for details regarding changes as compared to the protocol.

More details for the tables and listings can be found in Appendix I and Appendix II.

## 5.4.3.4 Subjects in remission at each visit

The number of subjects in remission will be summarised as described in the protocol section 11.3.4.2 for scheduled visits.

A stack plot over subjects in remission by scheduled visits will be presented.



|------------------------------|-------------------|----------------|

Further details for the table can be found in Appendix I and Appendix II.

## 5.4.3.5 Time to when PASI75 is no longer fulfilled

The endpoint will not be analysed. See section 5.7 regarding details of changes as compared to the protocol.

# 5.4.3.6 Time to first relapse according to m-PASI

The endpoint will not be analysed. See section 5.7 regarding details of changes as compared to the protocol.

# 5.4.3.7 Efficacy after treatment of relapse

Efficacy after treatment of relapse is defined as the proportion of subjects with 'clear' or 'almost clear' according to the PGA after treatment of relapse. The endpoint will be summarised as described in section 11.3.4.5 of the protocol.

A stack plot over proportion of subjects with 'clear' or 'almost clear' according to the PGA after treatment of relapse by treatment group and relapse number will be presented.

More details for the table can be found in Appendix I and Appendix II.

# **5.4.3.8** Target lesion/location scores

#### Open-label phase:

Target lesion/location will be summarised by visit. A shift table for categories of target lesion/location scores at visit 1 versus the category at visit 2 will also be done.

#### Maintenance phase:

Target lesion/location scores collected when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment group.

Target lesion/location scores collected when the subject is initiating a relapse period will be summarised by visit and visit intervals and by treatment group.

Target lesion/location scores collected when the subject is ending a relapse period will be summarised by visit and visit intervals and by treatment group.



|------------------------------|-------------------|----------------|

A shift table for categories of target lesion/location scores at start of relapse versus the category at end of relapse will also be done by visit for start of relapse and by treatment group.

Target lesion/location scores collected when the subject is in a relapse period will be listed only.

See section 5.7 for details regarding changes as compared to the protocol.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.4.3.9 Body Surface Area

Body surface area (BSA) should be interpreted as the percentage of BSA affected by psoriasis.

#### Open-label phase:

The percentage of BSA affected by psoriasis will be summarised by visit. Change and percent change in the affected BSA from visit 1 to visit 2 will also be summarised.

#### Maintenance phase:

The percentage of BSA affected by psoriasis collected when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment group.

The percentage of BSA affected by psoriasis collected when the subject is initiating a relapse period will be summarised by visit and visit intervals and by treatment group.

The percentage of BSA affected by psoriasis collected when the subject is ending a relapse period, will be summarised by visit and visit intervals and by treatment group.

Change and percent change in the affected BSA from start of relapse to end of relapse will be summarised by visit for start of relapse and by treatment group.

The percentage of BSA affected by psoriasis collected when the subject is in a relapse period, will be listed only.

See section 5.7 for details regarding changes as compared to the protocol.

More details for the tables and listings can be found in Appendix I and Appendix II.



|------------------------------|-------------------|----------------|

## 5.4.3.10 Number of active treatment days during maintenance phase

The number of active treatment days during maintenance phase will be normalised by time of exposure and summarised by treatment group.

For the active treatment group, the number of active treatment days is calculated as the sum of days where treated with maintenance treatment (twice weekly) and days where treated with rescue IMP. A day in relapse where treated with both maintenance medication and rescue IMP will count as one active treatment day.

For the vehicle group, the number of active treatment days during the maintenance phase is calculated as the sum of days where treated with rescue IMP.

The number of active treatment days during maintenance phase will also be listed.

More details for the tables and listings can be found in Appendix I and Appendix II.

# **5.4.4 Patient-Reported Outcomes**

Patient reported outcomes collected in the maintenance phase will be analysed for the full analysis set. Patient reported outcomes collected in the open-label phase will be analysed for the open-label full analysis set.

# 5.4.4.1 Dermatology Life Quality Index (DLQI)

#### Open-label phase:

Dermatology life quality index (DLQI) will be summarised by visit. Change and percent change in DLQI from visit 1 to visit 2 will also be summarised.

#### Maintenance phase:

DLQI collected when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment group.

DLQI collected when the subject is initiating a relapse period will be summarised by visit and visit intervals and by treatment group.

DLQI collected when the subject is ending a relapse period will be summarised by visit and visit intervals and by treatment group.



|------------------------------|-------------------|----------------|

Change and percent change in DLQI from start of relapse to end of relapse will be summarised by visit for start of relapse and by treatment group.

DLQI collected when the subject is in a relapse period will be listed only.

See section 5.7 for details regarding changes as compared to the protocol.

#### Details on total DLQI scores calculation:

The total DLQI score will be presented in all above mentioned tables. The total DLQI score is calculated by summing the score of each question. If one question is left unanswered, this is scored 0, and the total score is calculated as usual. If two or more questions are left unanswered, no total score is calculated. The questions 1-6 and 8-10 are scored as described in Table 4. Question 7 is scored as described in Table 5. The total DLQI score ranges from 0 (no quality of life impairment) to 30 (maximal quality of life impairment).

Table 4: Scoring of DLQI question 1-6 and 8-10

| Answer | Score |
|--------------|-------|
| Very much | 3 |
| A lot | 2 |
| A little | 1 |
| Not at all | 0 |
| Not relevant | 0 |
| Unanswered | 0 |

**Table 5: Scoring of DLQI question 7** 

| Answer | | Score |
|-------------------------|-----------------------|-------|
| Main part of question 7 | Subpart of question 7 | |
| Yes | Unanswered | 3 |
| Not relevant | Unanswered | 0 |
| No | A lot | 2 |
| No | A little | 1 |
| No | Not at all | 0 |
| No | Unanswered | 0 |

If the main part of question 7 is answered with 'Yes', and the subpart is not left unanswered, the score will remain 3. If the main part of question 7 is answered with 'Not relevant', and the



|------------------------------|-------------------|----------------|

subpart of the question is answered with 'A lot' or 'A little', the score will be 2 or 1 respectively.

#### Multiple imputation:

Missing DLQI total scores will be imputed using multiple imputation with 100 copies (seed=70309491) described in the steps below.

Missing assessment of the DLQI total score in-between non-missing assessments in the maintenance phase will not be imputed. The imputation step will depend on whether the reason for withdrawal for the subject to be imputed could potentially be related to IMP or not.

Imputation for subjects withdrawn with reasons 'withdrawal by subject' or 'lost to follow up': This approach assumes that in the unobserved part of maintenance phase, the subject will behave similar to the observed part of the maintenance phase for subjects in the same treatment group completing the maintenance phase.

#### Imputation steps:

- 1. DLQI data and relapse status from one subject in the sub-set of subjects that completed their maintenance phase and are in the same treatment group as the withdrawn subject will be randomly selected. This will be referred as 'sampled data' in step 2.
- 2. Missing visits for the withdrawn subject will be inputted using the relevant visits from the sampled data.
- 3. Steps 1 and 2 will be repeated 100 times for each withdrawn subject to form 100 complete datasets

Imputation subjects withdrawn with reasons 'adverse event', 'death', 'lack of efficacy', or 'subject not achieving clear or almost clear after treatment of relapse':

This approach assumes that the subjects behave similarly in the unobserved part of the trial as the observed part for subjects leaving the trial for the same reasons independent of treatment group.

#### Imputation steps:

1. Total DLQI scores and corresponding relapse status from subjects withdrawn from the trial due to 'adverse event', 'death', 'lack of efficacy', or 'subject not achieving clear or almost clear after treatment of relapse' will be collected as one set of data.



| Trial ID: LP0053-1004 | Date: 15-JUL-2019 | Version: 1.0 |
|-----------------------|-------------------|----------------|

- 2. A total DLQI scores will be sampled for each scheduled visit from the above collection of data (step 1).
- 3. Steps 1 and 2 will be repeated 100 times for each withdrawn subject to form 100 complete datasets

#### <u>Imputation for subjects leaving the trial due to other reasons:</u>

For cases with withdrawal reason specified as 'Other', the details will be revised on a blinded manner, selecting and documenting the imputation approach in the Analysis Set Definition Document.

#### Statistical analysis:

For each of the 100 complete datasets the total DLQI scores will be analysed using a Mixed effect Model Repeated Measurement (MMRM) with treatment group, visit (scheduled), interaction between treatment and visit, relapse status, and maintenance baseline total DLQI score as fixed factors and subject as random effect. Repeated measurements within subject is modelled using an unstructured variance structure. REML will be used for estimation.

The estimates and standard errors from the 100 analyses will be pooled into estimated least squares means for each treatment group and estimated treatment difference with associated standard errors using Rubin's rule to draw inference. From these pooled treatment estimates, the 95% CI for the treatment difference will be calculated. The p-value for treatment difference will be calculated using a two-tailed Student's t-test based on the pooled estimate. Pooled treatment estimates together with treatment difference, 95% CI and p-value will be presented by visit. Furthermore, the pooled treatment estimates will be plotted by visit.

See section 5.7 for details regarding changes as compared to the protocol.

More details for the tables and listings can be found in Appendix I and Appendix II.

#### 5.4.4.2 EQ-5D-5L-PSO

#### Open-label phase:

EQ-5D-5L-PSO dimensions, the index score and health on VAS score will be summarised by visit.

A shift table for the category for each of the EQ-5D-5L-PSO dimensions at visit 1 versus the category at visit 2 will be done.

Change and percent change in EQ-5D-5L-PSO index score and health on VAS score from visit 1 to visit 2 will be summarised.



|------------------------------|-------------------|----------------|

#### Maintenance phase:

EQ-5D-5L-PSO dimensions, the index score and health on VAS score collected when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment group.

EQ-5D-5L-PSO dimensions, the index score and health on VAS score collected when the subject is initiating a relapse period will be summarised by visit and visit intervals and by treatment group.

EQ-5D-5L-PSO dimensions, the index score and health on VAS score collected when the subject is ending a relapse period will be summarised by visit and visit intervals and by treatment group.

A shift table for the category for each of the EQ-5D-5L-PSO dimensions at start of relapse versus the category at end of relapse will also be done by visit for start of relapse and by treatment group.

Change and percent change in EQ-5D-5L-PSO index score and health on VAS score from start of relapse to end of relapse will be summarised by visit for start of relapse and by treatment group.

EQ-5D-5L-PSO dimensions, the index score and health on VAS score collected when the subject is in a relapse period, will be listed only.

See section 5.7 for details regarding changes as compared to the protocol.

More details for the tables and listings can be found in Appendix I and Appendix II.

The index score will be calculated calculated according to:

https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/valuation-standard-value-sets/crosswalk-index-value-calculator/.

The UK value sets will be used. In this way, each possible EQ-5D health state is assigned a weight representing the utility or value of that state, on a scale with a maximum value of 1, representing full health, and an anchor of 0, representing equivalent to being death. Values lower than 0 represent states regarded as worse than being death.



|------------------------------|-------------------|----------------|

#### 5.4.4.3 **WPAI:PSO**

The WPAI:PSO questionnaire will be presented by impairment percentages with high number indicating greater impairment. Four derived domains will be constructed from the WPAI:PSO questions (Q1-Q6) as described in Table 6.

Table 6: Scoring of WPAI:PSO question 1-6

| Impairment percentage | Score |
|---|---|
| Absenteeism | Q2/(Q2+Q4) |
| Presenteeism | Q5/10 |
| Total work productivity impairment (TWPI) | Q2/(Q2+Q4)+(1-Q2/(Q2+Q4))x(Q5/10) |
| Total activity impairment (TAI) | Q6/10 |

## Open-label phase:

The WPAI:PSO scores will be summarised by visit.

Change and percent change in each WPAI:PSO questions from visit 1 to visit 2 will also be summarised.

## Maintenance phase:

The WPAI:PSO scores will be summarised by visit, by treatment group and by whether the subject is on rescue IMP or not. As the WPAI:PSO questionnaire is based on experiences with psoriasis during the past 7 days, a subject will be summarised in the rescue IMP category if the subject has been on rescue IMP in at least one of the past 7 days prior to the visit. WPAI:PSO scores collected at unscheduled visits will be listed only.

More details for the tables and listings can be found in Appendix I and Appendix II.

## 5.4.4.4 Psoriasis Symptom Inventory

The total PSI score is calculated by summing the individual item score of each of the eight symptoms. If one question is left unanswered, this is scored 0, and the total score is calculated as usual. If two or more questions are left unanswered, no total score is calculated. The answers are scored as described in Table 7. The total PSI score ranges from 0 (not at all severe psoriasis symptoms) to 32 (very severe psoriasis symptoms).

**Table 7: Scoring of PSI questions** 

| Answer | Score |
|-------------|-------|
| Very severe | 4 |



|------------------------------|-------------------|----------------|

| Answer | Score |
|------------|-------|
| Severe | 3 |
| Moderate | 2 |
| Mild | 1 |
| Not at all | 0 |
| Unanswered | 0 |

#### Open-label phase:

The AUC for total PSI scores will be calculated. Change and percent change in total PSI score from visit 1 to visit 2 will also be summarised.

The AUC for the PSI total score will be calculated for each subject using the standard trapezoidal rule where trial day is used for the x-axis of the curve and total PSI score is used for the y-axis of the curve. The AUC will be normalised by dividing with the time period from visit 1 to visit 2. The normalisation converts the AUC to the original scale of the total PSI score.

#### Maintenance phase:

The AUC for the total PSI scores (from randomisation to 28 weeks after randomisation) will be calculated. The AUC for the total PSI score collected in time in remission and time in relapse, respectively, will be summarised by treatment group.

The AUC for the PSI total score for time in remission will be calculated for each subject by summing AUC over the time intervals where the subject is in remission. The AUC will be normalised by the total time the subject is in remission.

Likewise, the AUC for the PSI total score for time in relapse will be calculated for each subject by summing AUC over time intervals where the subject is in relapse. The AUC will be normalised by the total time the subject is in relapse. Missing assessment of the PSI total score in-between non-missing assessments in the maintenance phase will not be imputed, which corresponds to linear interpolation between non-missing assessments of the PSI total score.

#### Multiple imputation:

Missing DLQI total scores will be imputed using multiple imputation with 100 copies (seed=70309491). The imputation method and the imputation steps are the same as described for DLQI in section 5.4.4.1, however the imputation is done by week and not by visit.



|------------------------------|-------------------|----------------|

#### Statistical analysis:

For each of the 100 complete data sets, the total PSI scores will be analysed using a Mixed effect Model Repeat Measurement (MMRM) with treatment group, week (from randomisation), interaction between treatment and week, relapse status, and maintenance baseline total PSI score as fixed factors and subject as random effect. Repeated measurements within subject is modelled using an unstructured variance structure. REML will be used for estimation.

The estimates and standard errors from the 100 analyses will be pooled into estimated least squares means for each treatment group and estimated treatment difference with associated standard errors using Rubin's rule to draw inference. From these pooled treatment estimates, the 95% CI for the treatment difference will be calculated. The p-value for treatment difference will be calculated using a two-tailed Student's t-test based on the pooled estimate. Pooled treatment estimates together with treatment difference, 95% CI and p-value will be presented by week. Furthermore, the pooled treatment estimates will be plotted by week.

Subjects are supposed to complete the PSI questionnaire on a weekly basis the first 28 weeks of the maintenance phase and the 2 last weeks of the maintenance phase (Week 54 to 56) which is only applicable for completers. However, during blind review of data, it is observed that subjects in general forget to complete the questionnaire the last 2 weeks which implies that limited data are available for this period. For this reason, the analysis of the PSI total score will be based on the first 28 weeks of the maintenance phase.

The analysis of PSI will be done for full analysis set.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.4.4.5 Subject's Global Assessment of Disease Severity (SGA)

#### Open-label phase:

Subject's global assessment of disease severity (SGA) will be summarised by visit. A shift table for categories of subject's global assessment of disease severity at visit 1 versus the category at visit 2 will also be done.

#### Maintenance phase:

SGA collected when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment.



|------------------------------|-------------------|----------------|

SGA collected when the subject is initiating a relapse period, will be summarised by visit and visit intervals and by treatment.

SGA collected when the subject is ending a relapse period will be summarised by visit and visit intervals and by treatment group.

A shift table for categories of SGA at start of relapse versus the category at end of relapse will also be done by visit for start of relapse and by treatment group.

SGA collected when the subject is in a relapse period will be listed only.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.5 Analysis of Safety

The analyses of safety is done for the open-label safety analysis set and the safety analysis set.

# 5.5.1 Exposure

Duration of exposure will be summarised as described in the protocol section 11.3.3.1. If the date of last application of IMP is missing, the date of last visit attended by the subject will be used instead.

Patient years of exposure during a trial phase will be calculated as exposure during the relevant phase (accounting for both maintenance and rescue IMP as relevant) divided by 365.25.

The amount of IMP used will be summarised for the open-label treatment phase. For each subject the amount of IMP used will be normalised by the length of the open-label phase.

The total amount of IMP used, and the amount of rescue IMP used will be summarised by treatment group for the maintenance phase. For each subject the total amount of IMP and the amount of IMP used will be normalised by the length of maintenance phase or the total time in relapse, respectively.

The amount of IMP used, and the amount of rescue will not be summarised for each visit interval as described in the protocol. Instead a cumulative plot of the amount of IMP used over time during the maintenance phase by each subject together with an average cumulative amount curve will be done for the safety analysis set. The cumulative amount of IMP for each subject will be normalised by time in the maintenance phase (in days). The cumulative



|------------------------------|-------------------|----------------|

amount of IMP used up to each scheduled visit and the corresponding number of subjects contributing to these amounts will be tabulated by treatment group.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.5.2 Drug Accountability

For each subject, the weight of IMP used for a given trial period will be calculated as the difference between the weight of a set of full cans dispensed and the weight of the returned cans. The weight of cans dispensed to a subject will be the mean weight of a full can multiplied by the number of dispensed cans. The mean weight of a full can is 195.52 g based on the weight of 20 cans. The weight of IMP used will be multiplied by a correction factor of 0.41 to account for the propellant gasses.

If cans are returned with their seal unbroken, the weight of IMP used from that bottle will be assigned a value of zero. If a returned can weigh more than the estimated mean weight of a full can, it will be assumed that zero grams were used from that can.

If cans are returned at a wrong visit the amount of IMP used from these cans will be assumed to be used in the period from the cans being dispensed to the cans being returned. If some cans are not returned at all, these are cans are assumed to be emptied by the subjects. The amount of IMP used for that bottle will be assigned a value of 60 g, which is the approved amount of IMP contained in an individual can.

In the case where cans are not returned due to the subjects being lost to follow up after the cans is dispensed, the amount of IMP used from these cans will not be calculated, as the subject is assumed to end the treatment with IMP after withdrawal from the trial.

#### **5.5.3** Adverse Events

The adverse events (AEs) will be assigned to a specific period (e.g. open-label phase or randomised phase) based on the onset date the AE.

The long-term safety of LEO 90100 will be evaluated based on data from the randomised phase.

For treatment emergent adverse events (hereafter referred to as AEs) occurring in the randomised phase the following tables will be done:



|------------------------------|-------------------|----------------|

An overall summary of AEs, SAEs, premature discontinuation from the trial due to AEs, treatment related AEs, severity of AEs, action taken with IMP and outcome of AEs will be presented. The summary will include number of events, number (percentage) of subjects and exposure rates.

The number of AEs, the number and percentage of subjects experiencing each type of AE, and the exposure rate will be tabulated by SOC and preferred term. The tabulation will be done for all treatment emergent AEs, for each type of severity separately, for related AEs, for serious AEs (SAEs), for non-serious adverse events, and for frequent AEs (>= 1% in any treatment group).

All above tables will be done for the safety analysis set by treatment for the first 28 weeks of the randomised phase, and for the remaining 32 weeks of the randomised phase separately. In addition, the tables will be done for the safety analysis set by randomised treatment and rescue IMP for the total randomised phase, for the first 28 weeks of the randomised phase, and for the remaining 32 weeks of the randomised phase separately.

Further details for the tables can be found in Appendix I and Appendix II.

#### Open-label phase:

For completeness, AEs for the open-label phase will be summarised separately as follows:

An overall summary of AEs, SAEs, AEs leading to withdrawal, treatment related AEs, severity of AEs, action taken with IMP and outcome of AEs will be presented. The summary will include number of events, number (percentage) of subjects and exposure rates.

The number of AEs, the number and percentage of subjects experiencing each type of AE, and the exposure rate will be tabulated by SOC and preferred term. The tabulation will be done for all treatment emergent AEs, for each type of severity separately, for related AEs, for serious AEs (SAEs), for non-serious adverse events, and for frequent AEs (>= 1%).

The causal relationship to trial medication for each type of AE will be tabulated by SOC and preferred term.

All above tables will be done for the open-label safety analysis set.

#### Additional summaries in the maintenance phase:

Tables exploring safety profile while in remission or relapse will be presented based on the treatment emergent adverse events occurring in the maintenance phase.



|------------------------------|-------------------|----------------|

For AEs from the maintenance phase the following tables will be done:

The number of AEs, the number and percentage of subjects experiencing each type of AE, and the exposure rate will be tabulated by SOC and preferred term. The tabulation will be done for all treatment emergent AEs, for each type of severity separately, for related AEs, for serious AEs (SAEs), for non-serious adverse events, and for frequent AEs (>= 1% in any treatment group). The causal relationship to treatment regimen for each type of AE will be tabulated by SOC and preferred term.

All above tables will be done for the safety analysis set by treatment for the first 28 weeks of the maintenance phase, and for the remaining 24 weeks of the maintenance phase separately. In addition, the tables will be done for the safety analysis set by randomised treatment and rescue IMP for the total maintenance phase, for the first 28 weeks of the maintenance phase, and for the remaining 24 weeks of the maintenance phase separately.

All non-treatment emergent AEs will be listed.

Further details for listings can be found in Appendix I.

#### **Statistical tests:**

In the protocol it is described that the percentage of subjects with any AE or with any related AE will be compared between treatment groups by a chi-square test or Fisher's exact test (if expected cell count < 5). However, this analysis will most likely be biased towards different drop-out between the treatment groups. The longer a subject is followed, the greater is the chance of observing an AE for the subject. As the number of early withdrawals might differ considerably between the two treatment groups, statistical tests performed on the percentage of subjects with any AE or with any related AE is not appropriate in this set up. Hence, no statistical testing will be done for AEs.

#### Calculation of AE rate:

The AE rate will be calculated as number of AEs divided by patient years of exposure in the different phases multiplied by 100.

# 5.5.3.1 Adverse events associated with long term corticosteroid use

Adverse events associated with long term corticosteroid use will be presented as described in the protocol.



|------------------------------|-------------------|----------------|

#### 5.5.4 Rebound

Rebounds will be defined as described in the protocol. The baseline value will be the m-PASI value measured at the start of the rebound follow-up period. A rebound follow-up period is defined as either (i) 2 months after discontinuation of open-label phase treatment, (ii) 2 months after discontinuation of relapse treatment, or (iii) 2 months after discontinuation of maintenance treatment (up to Visit FU3).

Number of rebounds occurring within the first 2 months after discontinuation of the openlabel phase treatment, and number of rebounds occurring within 2 months after discontinuation of relapse treatment will be summarised by treatment group.

Number of rebounds occurring within two months after discontinuation of maintenance treatment will be summarised by treatment group.

Cases of rebounds will be listed.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.5.5 Physician's Assessment of Local Safety and Tolerability

#### Open-label phase:

Physician's assessment of local safety and tolerability will be summarised by visit. A shift table for categories of physician's assessment of local safety and tolerability at visit 1 versus the category at visit 2 will also be done.

#### Maintenance phase:

Physician's assessment of local safety and tolerability when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment group.

Physician's assessment of local safety and when the subject is initiating a relapse period will be summarised by visit and visit intervals and by treatment group.

Physician's assessment of local safety and tolerability when the subject is ending a relapse period will be summarised by visit and visit intervals and by treatment group.

A shift table for categories of physician's assessment of local safety and tolerability at start of relapse versus the category at end of relapse will also be done by visit for start of relapse and by treatment group.



|------------------------------|-------------------|----------------|

Physician's assessment of local safety and tolerability collected when subject is in a relapse period, will be listed only.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.5.6 Subject's Assessment of Local Safety and Tolerability

#### Open-label phase:

Subject's assessment of local safety and will be summarised by visit. A shift table for categories of subject's assessment of local safety and tolerability at visit 1 versus the category at visit 2 will also be done.

#### Maintenance phase:

Subject's assessment of local safety and tolerability collected when the subject is not initiating, ending or in a relapse period will be summarised by visit and by treatment group.

Subject's assessment of local safety and tolerability collected when the subject is initiating a relapse period will be summarised by visit and visit intervals and by treatment group.

Subject's assessment of local safety and tolerability collected when the subject is ending a relapse period will be summarised by visit and visit intervals and by treatment group.

A shift table for categories of subject's assessment of local safety and tolerability at start of relapse versus the category at end of relapse will also be done by visit for start of relapse and by treatment group.

Subject's assessment of local safety and tolerability collected when the subject is in a relapse period, will be listed only.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.5.7 ACTH-Challenge Test

#### Open-label phase:

For the group of subjects undergoing the ACTH-challenge test, the number and percentages of subjects with serum-cortisol concentration values ≤18 mcg/dl at 30 minutes and 60 minutes after the ACTH-challenge test will be summarised by visit.

The serum-cortisol concentration at time 0 (just before the ACTH-challenge test) and at 30 and 60 minutes after ACTH-challenge at visit 1 and visit 2 will be summarised.



|------------------------------|-------------------|----------------|

Individual data for subjects with serum cortisol concentration values ≤18 mcg/dl at either 30 or at 60 minutes after ACTH-challenge in the open-label phase will be tabulated.

A mean plot of the serum-cortisol concentration at time 0, and at 30 and 60 minutes after the ACTH-challenge test for visit 1 and visit 2 will be done.

#### Maintenance phase:

The number and percentages of subjects with serum-cortisol concentration values  $\leq$ 18 mcg/dl at 30 minutes and 60 minutes after the ACTH-challenge test will be summarised by visit and by treatment group.

The serum-cortisol concentration at time 0 and at 30 and 60 minutes after ACTH-challenge tests will be summarised by visit and treatment group.

Individual data for subjects with serum cortisol concentration values  $\leq$ 18 mcg/dl at either 30 or at 60 minutes after ACTH-challenge will be tabulated.

A mean plot of the serum-cortisol concentration at time 0, and at 30 and 60 minutes after the ACTH-challenge test by treatment group will be done.

Results from ACTH-tests performed at early termination visits will be listed only and are not included in the above-mentioned tables and figures.

More details for the tables and listings can be found in Appendix I and Appendix II.

# 5.5.8 Vital Signs and Physical Findings

#### Open-label phase:

The change in vital signs (blood pressure, heart rate) from baseline to end of open-label treatment phase will be summarised.

#### Maintenance phase:

The change in vital signs (blood pressure, heart rate) from randomisation to end of trial will be summarised.

In addition, the change in vital signs from randomisation to end of maintenance phase for subjects discontinuing before 6 months after randomisation, the change in vital signs from randomisation to end maintenance phase for subjects discontinuing on or after 6 months after


|------------------------------|-------------------|----------------|

randomisation, and the change in vital signs from randomisation to visit 15 will be summarised.

If more than one vital sign value is reported for the same visit and time point, the latest value will be used in summary statistics and analyses.

If vital sign measurements are missing for a subject at baseline or at randomisation the change from baseline or randomisation to a specific visit will not be calculated.

Further details for the tables can be found in Appendix I and Appendix II.

Findings from physical examinations and vital signs data will be listed. More details can be found in Appendix I.

#### 5.5.9 Laboratory Data

For the laboratory values, if the value is below the lower limit of quantification, half of the lower limit will be used for quantitative summaries. If the value is above the upper limit of quantification, the upper limit value will be used. If more than one laboratory value is reported for the same visit, the latest value will be used in summary statistics and analyses.

If laboratory parameters are missing for a subject at baseline or at randomisation the change from baseline or randomisation to a specific visit will not be calculated.

Laboratory parameters will be categorised as described in the protocol.

#### Open-label phase:

The change in each of the laboratory parameters from baseline to end of open-label treatment phase will be summarised. A shift table for categories of laboratory parameters at visit 1 versus the category at visit 2 will also be done.

#### Maintenance phase:

The change in laboratory parameters from randomisation to end of maintenance phase for subjects discontinuing before 6 months after randomisation, the change in laboratory parameters from randomisation to end of maintenance phase for subjects discontinuing on or after 6 months after randomisation, and the change in laboratory parameters from randomisation to visit 15 will be summarised.



|------------------------------|-------------------|----------------|

Shift tables showing the categories at randomisation against those at end of maintenance phase for subjects discontinuing before 6 months after randomisation, for subjects discontinuing the trial on or after 6 months after randomisation, and for subjects completing the maintenance phase will be produced.

For subjects with at least one clinically significant value of albumin corrected serum calcium, similar shift tables as described above will be produced.

All laboratory data will be listed. Additionally, subjects with laboratory parameters outside the reference range will be listed in a separate listing.

Further details for the tables and listings can be found in Appendix I and Appendix II.

# **5.6** General Principles

## 5.6.1 Pooling of Trial Sites

As many centres randomises only a few subjects, the centres will be pooled together. For the United States, due to the large geographical area and diverse climatic conditions, centres will be pooled with neighbouring centres based on graphical location and climatic zones to form two pooled centres. The pooling of sites is shown in Table 8.

**Table 8: Pooling of trial sites** 

| Country | Number of subjects randomised | Pooled sites |
|---|---|---|
| Canada | 132 | CAN140, CAN142, CAN143, CAN144, CAN145,<br>CAN146, CAN147, CAN148, CAN149, CAN150,<br>CAN152, CAN154 |
| France | 55 | FRA160, FRA161, FRA162, FRA165, FRA167 |
| Germany | 52 | DEU183, DEU185, DEU186, DEU187, DEU188, DEU189, DEU193 |
| Great Britain | 68 | GBR200, GBR201, GBR202, GBR203, GBR207,<br>GBR209, GBR210 |



|------------------------------|-------------------|----------------|

| Poland | 56 | POL220, POL221, POL222, POL224 |
|---|---|---|
| United States (1) | 68 | USA103, USA106, USA109, USA112, USA122 |
| United States (2) | 114 | USA100, USA102, USA104, USA107, USA108, USA110, USA111, USA113, USA115, USA116, USA117, USA118, USA119, USA120, USA121 |

## 5.6.2 Handling of Drop-outs and Missing Values

The methods of dealing with drop-outs and missing values for primary and secondary endpoints are specified in the relevant sections of the statistical analysis plan, where the analyses of the endpoints are described. If nothing is specified in these sections, missing data and drop-outs are not an issue of concern for the analyses of the endpoint and nothing will be done.

## **5.6.3** Incomplete dates

For incomplete start dates of adverse events in data, the following rules apply:

- If a start day is missing, but start month and year is not missing, it will be assumed that the start date of the adverse event is the date of last contact with the subject in that month, if available, and otherwise it will be the first day of the month.
- If both start day and month is missing, it will be assumed that the start date of the adverse event is the date of the last contact with the subject before the end date of the adverse event.

The adverse events will be assigned to rescue medication and randomised treatment as described in section 5.5.3 based on the imputed dates derived from the above rules.

# 5.6.4 Multiplicity adjustment

To control the overall type 1 error rate, the analyses of the primary and secondary endpoints will follow the hierarchical testing procedure outlined in Figure 3. The hypotheses relating to the two secondary endpoints cannot be rejected unless the hypothesis relating to the primary endpoint is also rejected.



|------------------------------|-------------------|----------------|

Figure 3: Testing procedure for primary and secondary endpoints



The procedure will be as follows:

Time to first relapse between LEO 90100 and vehicle is evaluated at a 5% significance level. If the test is significant, the significance level will be split between the analyses of the two secondary endpoints using the Holm Bonferroni method to adjust for multiplicity. Hence the proportion of days in remission and the number of relapses during the maintenance phase between LEO 90100 and vehicle will be tested in parallel at a 2.5% significance level.

#### **5.6.5** Treatment Labels

The treatment labels for the clinical trial report text and tables are shown in Table 9.

Table 9: Treatment labels for the clinical trial report text and tables

| Label Used in Text | Label Used in Tables | Order in Table |
|--------------------------------|----------------------|----------------|
| LEO 90100 aerosol foam | LEO 90100 | 1 |
| LEO 90100 aerosol foam vehicle | Vehicle | 2 |



|------------------------------|-------------------|----------------|

# 5.7 Changes to the analyses described in the protocol

The following changes have been done to the analyses described in the protocol:

| SAP section | Endpoint/Assessment | Description of change |
|---|---|---|
| Section 5.3.4 | Compliance | Data captured in the eDiary will not allow the computation of percentage |
| | | missed application in the maintenance phase as described in the protocol |
| | | (section 11.3.3.2). |
| | | Number of subjects in non-compliance with maintenance treatment |
| | | instructions (i.e.; excluding relapse periods) will be summarised by |
| | | treatment group. |
| Section 5.4.1 | Time to first relapse (primary endpoint) | The analysis described in the protocol includes disease severity at baseline |
| | | (visit 1) as a covariate and trial site as a factor in the model (section |
| | | 11.3.3.3). |
| | | In the SAP the disease severity at maintenance baseline and pooled sites |
| | | are included in the model instead. |
| | | A sensitivity analysis is added in the SAP, where the primary endpoint will |
| | | be analysed incorporating interval censoring. As compared to the primary |
| | | analysis assuming that the start of relapse is known, the sensitivity analysis |
| | | assumes the relapse starts between two visits. |
| | | The analysis of subjects who are still at risk for a first relapse at week 26 |



|------------------------------|-------------------|----------------|

| Section 5.4.2.2 | Number of relapses during the maintenance phase. | The analysis described in the protocol includes disease severity at baseline (visit 1) as a covariate and trial site as a factor in the model (section |
|---|---|---|
| | | In the SAP a multiple imputation method is described instead. See section 5.4.2.1 for details. |
| | | The imputation method described in the protocol section 11.3.3.6 is not done, since if the withdrawal rate is higher in the vehicle arm (due to lower efficacy), the approach would favour the active treatment arm. |
| Section 5.4.2.1 | Proportion of days in remission | Analysis of number of days in remission is described in the protocol (section 11.3.3.6). The length of the maintenance phase will vary from subject to subject and will influence the number of days in remission. Due to this reason, the endpoint in SAP has been changed to the proportion of days in remission. |
| Section 5.4.3.1 | Proportion of subjects who are still at risk of a first relapse at week 26. Proportion of subjects who are still at risk of a first relapse at week 52. | and 52 mentioned in the protocol section 11.3.3.3 are described as two addition exploratory efficacy endpoints in section 5.4.3.1. These two endpoints where mentioned in section 11.3.3.3 of the protocol. In the SAP they are added as exploratory endpoints. |



|------------------------------|-------------------|----------------|

| | | 11 2 2 () |
|---|---|---|
| | | 11.3.3.6). |
| | | In the SAP the disease severity at maintenance baseline and pooled sites |
| | | are included in the model instead. |
| | | Sensitivity analysis: |
| | | The analysis described in the protocol (section 11.3.3.6) will not be done |
| | | as it conditions on future events by excluding subjects who at some point |
| | | do not achieve 'clear' or 'almost' clear according to PGA after treatment of |
| | | relapse. A negative binomial regression model will be used for the analysis |
| | | instead. See section 5.4.2.2 for details. |
| Sections 5.4.3.2 | m-PASI | In the protocol section 11.3.4.1 it is described that the endpoint will be |
| | | summarised by visit. Since per protocol subjects will be withdrawn when |
| | | not achieving 'clear' or 'almost clear' according to PGA after rescue IMP, |
| | | the subset of subject's available values at the visits will be a selected |
| | | population (most likely are subjects who responds well to the IMP). Hence |
| | | summaries by visit will not be done. |
| | | The summaries will be done only for data capture at the start or the end of |
| | | a relapse period. See section 5.4.3.2. |
| Section 5.4.3.3 | Physician's Global Assessments of | This endpoint is added as compared to the protocol. |
| | disease severity | The summaries will be done only for data capture at the start or the end of |
| | | a relapse period. See section 5.4.3.3 for details. |



|------------------------------|-------------------|----------------|

| Section 5.4.3.5 | Time to when PASI75 is no longer | PASI and PGA are both tools for assessing the psoriasis severity and will |
|---|---|---|
| | fulfilled | therefore be mutually related. Since rescue IMP will be given to patients in |
| | | relapse (based on the PGA) y, the level of PASI might also be affected. |
| | | Therefore, the observed progress in PASI over time might be confounded |
| | | with the rescue IMP. For this reason, time to when PASI75 is no longer |
| | | fulfilled, will not be analysed (protocol section 11.3.4.3). |
| Section 5.4.3.6 | Time to first relapse according to m- | m-PASI and PGA are both tools for assessing the psoriasis severity and |
| | PASI | will therefore be mutually related. Since rescue IMP will be given to |
| | | patients in relapse (based on the PGA) y, the level of m-PASI might also be |
| | | affected. Therefore, the observed progress in m-PASI over time might be |
| | | confounded with the rescue IMP. For this reason, time to first relapse |
| | | according to m-PASI, will not be analysed (protocol section 11.3.4.4). |
| Section 5.4.3.8 | Target lesion/location scores | In the protocol section 11.3.4.6 it is described that the endpoint will be |
| | | summarised by visit. Since per protocol subjects will be withdrawn when |
| | | not achieving 'clear' or 'almost clear' according to PGA after rescue IMP, |
| | | the subset of subject's available values at the visits will be a selected |
| | | population (most likely are subjects who responds well to the IMP). Hence |
| | | summaries by visit will not be done. |
| | | The summaries will be done only for data capture at the start or the end of |
| | | a relapse period. See section 5.4.3.8. |



|------------------------------|-------------------|----------------|

| Section 5.4.3.9 | Body surface area | In the protocol section 11.3.4.7 it is described that the endpoint will be |
|---|---|---|
| | | summarised by visit. Since per protocol subjects will be withdrawn when |
| | | not achieving 'clear' or 'almost clear' according to PGA after rescue IMP, |
| | | the subset of subject's available values at the visits will be a selected |
| | | population (most likely are subjects who responds well to the IMP). Hence |
| | | summaries by visit will not be done. |
| | | The summaries will be done only for data capture at the start or the end of |
| | | a relapse period. See section 5.4.3.9. |
| Section 5.4.4.1 | Total DLQI score | In the protocol section 11.3.5.1 it is described that the endpoint will be |
| | | summarised by visit. Since per protocol subjects will be withdrawn when |
| | | not achieving 'clear' or 'almost clear' according to PGA after rescue IMP, |
| | | the subset of subject's available values at the visits will be a selected |
| | | population (most likely are subjects who responds well to the IMP). Hence |
| | | summaries by visit will not be done. |
| | | The summaries will be done only for data capture at the start or the end of |
| | | a relapse period. See section 5.4.4.1. |
| | | The analysis described in the protocol section 11.3.5.1 disregard the |
| | | possible differences in withdrawal patterns between the two treatment |
| | | groups. Instead multiple imputation for missing data and an MMRM |
| | | analysis will be done. See section 5.4.4.1 for details. |



|------------------------------|-------------------|----------------|

| Section 5.4.4.2 | EQ-5D-5L PSO | In the protocol section 11.3.5.2 it is described that the endpoint will be summarised by visit. Since per protocol subjects will be withdrawn when not achieving 'clear' or 'almost clear' according to PGA after rescue IMP, the subset of subject's available values at the visits will be a selected population (most likely are subjects who responds well to the IMP). Hence summaries by visit will not be done. The summaries will be done only for data capture at the start or the end of a relapse period. See section 5.4.4.2. |
|---|---|---|
| Section 5.4.4.4 | PSI | In the protocol section 11.3.5.1 it is described that the endpoint will be summarised over time. Since per protocol subjects will be withdrawn when not achieving 'clear' or 'almost clear' according to PGA after rescue IMP, the subset of subject's available values over time in the trial will be a selected population (most likely are subjects who responds well to the IMP). Hence summaries over time will not be done. The summaries will be done using AUC over trial phases. See section 5.4.4.4 for details. |
| | | The analysis described in the protocol section 11.3.5.4 disregard the possible differences in withdrawal patterns between the two treatment |



|------------------------------|-------------------|----------------|

| | | groups. Instead multiple imputation for missing data and an MMRM analysis will be done. See section 5.4.4.1 for details. |
|---|---|---|
| Section 5.4.4.5 | SGA | In the protocol section 11.3.5.5 it is described that the endpoint will be summarised by visit. Since per protocol subjects will be withdrawn when not achieving 'clear' or 'almost clear' according to PGA after rescue IMP, the subset of subject's available values at the visits will be a selected population (most likely are subjects who responds well to the IMP). Hence summaries by visit will not be done. The summaries will be done only for data capture at the start or the end of a relapse period. See section 5.4.4.5. |



|------------------------------|-------------------|----------------|

# Appendix I

Tables, Figures and Listings



|------------------------------|-------------------|----------------|

# **Tables and Figures, Baseline Characteristics and Investigational Product Data (Module 2)**

#### **Tables**

- Table 1-1 Disposition of subjects in the open-label phase: enrolled subjects
- Table 1-2 Disposition of subjects in the maintenance phase: randomised subjects
- Table 1-3 Reasons for leaving the trial during the open-label phase by last visit attended: enrolled subjects
- Table 1-4 Reasons for leaving the trial during the maintenance phase by last visit attended: randomised subjects
- Table 1-5 Age, height, weight, BMI and duration of psoriasis vulgaris: open-label safety analysis set
- Table 1-6 Age, height, weight, BMI and duration of psoriasis vulgaris: randomised subjects
- Table 1-7 Age by site: open-label safety analysis set
- Table 1-8 Age by site: randomised subjects
- Table 1-9 Age group, sex, race, ethnicity, and skin type: open-label safety analysis set
- Table 1-10 Age group, sex, race, ethnicity, and skin type: randomised subjects
- Table 1-11 Sex, race, and ethnicity by site: open-label safety analysis set
- Table 1-12 Sex, race, and ethnicity by site: randomised subjects
- Table 1-13 PGA at baseline: open-label safety analysis set
- Table 1-14 PGA at baseline: randomised subjects
- Table 1-15 PGA at baseline by site: open-label safety analysis set
- Table 1-16 PGA at baseline by site: randomised subjects
- Table 1-17 m-PASI and BSA involved at baseline: open-label safety analysis set
- Table 1-18 m-PASI and BSA involved at baseline: randomised subjects
- Table 1-19 m-PASI at baseline by site: open-label safety analysis set
- Table 1-20 m-PASI at baseline by site: randomised subjects
- Table 1-21 Vital signs at baseline: open-label safety analysis set
- Table 1-22 Vital signs at baseline: randomised subjects
- Table 1-23 Vitamin D at baseline: open-label safety analysis set
- Table 1-24 Vitamin D at baseline: randomised subjects
- Table 1-25 Location of psoriasis and location of other psoriasis at baseline: open-label safety analysis set



|------------------------------|-------------------|----------------|

- Table 1-26 Location of psoriasis and location of other psoriasis at baseline: randomised subjects
- Table 1-27 Concurrent diagnoses at baseline: open-label safety analysis set
- Table 1-28 Concurrent diagnoses at baseline: randomised subjects
- Table 1-29 Concomitant medication at baseline: open-label safety analysis set
- Table 1-30 Concomitant medication at baseline: randomised subjects
- Table 1-31 Previous and latest systemic anti-psoriatic therapy: open-label safety analysis set
- Table 1-32 Previous and latest systemic anti-psoriatic therapy: randomised subjects
- Table 1-33 Previous and latest topical anti-psoriatic therapy: open-label safety analysis set
- Table 1-34 Previous and latest topical anti-psoriatic therapy: randomised subjects
- Table 1-35 Duration of exposure during the open-label treatment phase: open-label phase safety analysis set
- Table 1-36 Duration of exposure during the maintenance phase: safety analysis set
- Table 1-37 Amount of investigational medicinal product used: open-label safety analysis set
- Table 1-38 Amount of investigational medicinal product and rescue medication used: safety analysis set
- Table 1-39 Cumulative amount of investigational medical product used up each scheduled visit: safety analysis set
- Table 1-40 Compliance with treatment instructions during open-label treatment phase: open-label safety analysis set
- Table 1-41 Compliance with treatment instructions during maintenance phase excluding periods of treatment with rescue medication: safety analysis set
- Table 1-42 Compliance with treatment instructions during periods of treatment with rescue medication: safety analysis set

#### **Figures**

- Figure 1-1 Discontinuation by reason during open-label phase: open-label safety analysis set
- Figure 1-2 Discontinuation by reason during maintenance phase: safety analysis set.
- Figure 1-3 Cumulative amount of amount of investigational medical product used: safety analysis set.

#### Tables and Figures, Efficacy Data (Module 3)

#### **Tables**



|------------------------------|-------------------|----------------|

#### **Primary Efficacy Endpoint**

- Table 2-1 Censored and uncensored observations for time to first confirmed relapse: full analysis set
- Table 2-2 Censored and uncensored observations for time to first confirmed relapse: per protocol analysis set
- Table 2-3 Number of subjects at risk of first relapse by scheduled visit: full analysis set
- Table 2-4 Number of subjects at risk of relapse by relapse by scheduled visit: per protocol analysis set
- Table 2-5 Statistical analysis of time to first relapse: full analysis set
- Table 2-6 Statistical analysis of time to first relapse: per protocol analysis set
- Table 2-7 Percentiles from estimated survival curves: full analysis set
- Table 2-8 Percentiles from estimated survival curves: per protocol analysis set
- Table 2-9 Summary of observation types—sensitivity analysis: full analysis set
- Table 2-10 Summary of observation types sensitivity analysis: per protocol analysis set
- Table 2-11 Sensitivity analysis of time to first relapse: full analysis set
- Table 2-12 Percentiles from estimated survival curves sensitivity analysis: full analysis set

#### **Secondary Efficacy Endpoints**

- Table 2-13 Observed proportion of days in remission: full analysis set
- Table 2-14 Observed proportion of days in remission: per protocol analysis set
- Table 2-15 Statistical analysis of proportion of days in remission: full analysis set
- Table 2-16 Statistical analysis of proportion of days in remission: per protocol analysis set
- Table 2-17 Sensitivity analysis of proportion of days in remission: full analysis set
- Table 2-18 Number of relapses during maintenance phase: full analysis set
- Table 2-19 Number of relapses during maintenance phase: per protocol analysis set
- Table 2-20 Statistical analysis of number of relapses during maintenance phase: full analysis set
- Table 2-21 Statistical analysis of number of relapses during maintenance phase: per protocol analysis set
- Table 2-22 Sensitivity analysis of number of relapses during maintenance phase (negative binomial model): full analysis set

#### **Exploratory Efficacy Endpoints**



|------------------------------|-------------------|----------------|

- Table 2-23 Comparison of proportions of subjects still at risk of first relapse at 26 weeks and 52 weeks after randomisation using z-test: full analysis set
- Table 2-24 Comparison of proportions of subjects still at risk of first relapse at 26 weeks and 52 weeks after randomisation using exact test: full analysis set
- Table 2-25 m-PASI by visit in open-label phase: open-label safety analysis set
- Table 2-26 Change in m-PASI from start to end of open-label phase: open-label safety analysis set
- Table 2-27 Percent change in m-PASI from start to end of open-label phase: open-label safety analysis set
- Table 2-28 m-PASI by visit not related to relapse: full analysis set
- Table 2-29 m-PASI by visit for start of relapse: full analysis set
- Table 2-30 m-PASI by visit for end of relapse: full analysis set
- Table 2-31 Change in m-PASI from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-32 Percent change in m-PASI from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-33 Physician's global assessment of disease severity by visit in open-label phase: open-label safety analysis set
- Table 2-34 Shift table for physician's global assessment of disease severity from start to end of open-label phase: open-label safety analysis set
- Table 2-35 Physician's global assessment of disease severity by visit not related to relapse: full analysis set
- Table 2-36 Physician's global assessment of disease severity by visit for start of relapse: full analysis set
- Table 2-37 Physician's global assessment of disease severity by visit for end of relapse: full analysis set
- Table 2-38 Shift table for physician's global assessment of disease severity from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-39 Subjects in remission by scheduled visit: full analysis set
- Table 2-40 Subjects achieving clear or almost clear after treatment of relapse by number of relapses: full analysis set
- Table 2-41 Target lesion/location scores by visit in open-label phase: open-label safety analysis set



|------------------------------|-------------------|----------------|

- Table 2-42 Shift tables for target lesion/location scores from start to end of open-label phase: open-label safety analysis set
- Table 2-43 Target lesion/location scores by visit not related to relapse: full analysis set
- Table 2-44 Target lesion/location scores by visit for start of relapse: full analysis set
- Table 2-45 Target lesion/location scores by visit for end of relapse: full analysis set
- Table 2-46 Shift table for target lesion/location scores from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-47 BSA by visit in open-label phase: open-label safety analysis set
- Table 2-48 Change in BSA from start to end of open-label phase: open-label safety analysis set
- Table 2-49 Percent change in BSA from start to end of open-label phase: open-label safety analysis set
- Table 2-50 BSA by visit not related to relapse: full analysis set
- Table 2-51 BSA by visit for start of relapse: full analysis set
- Table 2-52 BSA by visit for end of relapse: full analysis set
- Table 2-53 Change in BSA from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-54 Percent change in BSA from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-55 Number of active treatment days during maintenance phase: full analysis set

#### **Patient-Reported Outcomes**

- Table 2-56 DLQI by visit in open-label phase: open-label safety analysis set
- Table 2-57 Change in DLQI from start to end of open-label phase: open-label safety analysis set
- Table 2-58 Percent change in DLQI from start to end of open-label phase: open-label safety analysis set
- Table 2-59 DLQI by visit not related to relapse: full analysis set
- Table 2-60 DLQI by visit for start of relapse: full analysis set
- Table 2-61 DLQI by visit for end of relapse: full analysis set
- Table 2-62 Change in DLQI from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-63 Percent change in DLQI from start of relapse to end of relapse by visit for start of relapse: full analysis set



|------------------------------|-------------------|----------------|

- Table 2-64 Statistical analysis of DLQI; full analysis set
- Table 2-65 EQ-5D-5L-PSO by visit in open-label phase: open-label safety analysis set
- Table 2-66 Shift tables for EQ-5D-5L-PSO dimensions from start to end of open-label phase: open-label safety analysis set
- Table 2-67 Change in EQ-5D-5L-PSO index score from start to end of open-label phase: open-label safety analysis set
- Table 2-68 Percent change in EQ-5D-5L-PSO index score from start to end of open-label phase: open-label safety analysis set
- Table 2-69 EQ-5D-5L-PSO by visit not related to relapse: full analysis set
- Table 2-70 EQ-5D-5L-PSO by visit for start of relapse: full analysis set
- Table 2-71 EQ-5D-5L-PSO by visit for end of relapse: full analysis set
- Table 2-72 Shift table for EQ-5D-5L-PSO dimensions from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-73 Change in EQ-5D-5L-PSO index score from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-74 Percent change in EQ-5D-5L-PSO index score from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-75 Health on VAS score by visit in open-label phase: open-label safety analysis set
- Table 2-76 Change in health on VAS score from start to end of open-label phase: open-label safety analysis set
- Table 2-77 Percent change in health on VAS score from start to end of open-label phase: open-label safety analysis set
- Table 2-78 Health on VAS score by visit not related to relapse: full analysis set
- Table 2-79 Health on VAS score by visit for start of relapse: full analysis set
- Table 2-80 Health on VAS score by visit for end of relapse: full analysis set
- Table 2-81 Change in health on VAS score from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-82 Percent change in health on VAS score from start of relapse to end of relapse by visit for start of relapse: full analysis set
- Table 2-83 WPAI:PSO by visit in open-label phase: open-label safety analysis set
- Table 2-84 Change in WPAI:PSO from start to end of open-label phase: open-label safety analysis set
- Table 2-85 Percent change in WPAI:PSO from start to end of open-label phase: open-label safety analysis set



| Tria | al ID: <b>LP0053-1004</b> | Date: 15-JUL-2019 | Version: 1.0 |
|------|---------------------------|-------------------|----------------|

- Table 2-86 WPAI:PSO by visit: full analysis set
- Table 2-87 Total PSI score during open-label phase; open-label safety analysis set.
- Table 2-88 Change in total PSI score from start to end of open-label phase; open-label safety analysis set.
- Table 2-89 Percent change in total PSI score from start to end of open-label phase; open-label safety analysis set.
- Table 2-90 Total PSI score for time on rescue medication and time in remission during the first 28 weeks of the maintenance phase; full analysis set.
- Table 2-91 Statistical analysis of PSI; full analysis set
- Table 2-92 Subject's global assessment of disease severity by visit in open-label phase: open-label safety analysis set
- Table 2-93 Shift table for subject's global assessment of disease severity from start to end of open-label phase: open-label safety analysis set
- Table 2-94 Subject's global assessment of disease severity by visit not related to relapse: full analysis set
- Table 2-95 Subject's global assessment of disease severity by visit for start of relapse: full analysis set
- Table 2-96 Subject's global assessment of disease severity by visit for end of relapse: full analysis set
- Table 2-97 Shift tables for subject's global assessment of disease severity from start of relapse to end of relapse by visit for start of relapse: full analysis set

#### **Figures**

- Figure 2-1 Estimated survival curves with 95% confidence intervals for time to first relapse: full analysis set
- Figure 2-2 Estimated survival curves with 95% confidence intervals for time to first relapse: per protocol analysis set
- Figure 2-3 Estimated survival curves with 95% confidence intervals for time to first relapse sensitivity analysis: full analysis set
- Figure 2-4 Distribution of proportion of days in remission: full analysis set
- Figure 2-5 Distribution of proportion of days in remission: per protocol analysis set
- Figure 2-6 Distribution of number of relapses during maintenance phase: full analysis set
- Figure 2-7 Distribution of number of relapses during maintenance phase: per protocol analysis set
- Figure 2-8 Number of days in remission between relapses: full analysis set



|------------------------------|-------------------|----------------|

- Figure 2-9 Number of days in remission between relapses: per protocol analysis set
- Figure 2-10 Stacked plot over subjects in remission by visit: full analysis set
- Figure 2-11 Stacked plot over subjects in remission by visit: per protocol analysis set
- Figure 2-12 Stacked plot for efficacy after treatment of relapse: full analysis set
- Figure 2-13 Estimated treatment difference for DLQI by visit: full analysis set
- Figure 2-14 Estimated treatment difference for PSI by week: full analysis set

#### **Tables and Figures, Safety Data (Module 4)**

#### **Tables**

- Table 3-1 Overall summary of adverse events during open-label phase: open-label safety analysis set
- Table 3-2 Overall summary of adverse events during the total maintenance phase by randomised treatment: safety analysis set
- Table 3-3 Overall summary of adverse events during the first 28 weeks of the randomised phase by randomised treatment: safety analysis set
- Table 3-4 Overall summary of adverse events during the last 32 weeks of the randomised phase by randomised treatment: safety analysis set
- Table 3-5 Overall summary of adverse events during the total maintenance phase by randomised treatment and rescue medication: safety analysis set
- Table 3-6 Overall summary of adverse events during the first 28 weeks of the maintenance phase by randomised treatment and rescue medication: safety analysis set
- Table 3-7 Overall summary of adverse events during the last 24 weeks of the maintenance phase by randomised treatment and rescue medication: safety analysis set
- Table 3-8 Adverse events during the open-label phase by SOC and preferred term: open-label safety analysis set
- Table 3-9 Adverse events during the total randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-10 Adverse events during the first 28 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-11 Adverse events during the last 32 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-12 Adverse events during the total maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set



|------------------------------|-------------------|----------------|

- Table 3-13 Adverse events during the first 28 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-14 Adverse events during the last 24 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-15 Mild adverse events during open-label phase by SOC and preferred term: open-label safety analysis set
- Table 3-16 Mild adverse events during the total randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-17 Mild adverse events during the first 28 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-18 Mild adverse events during the last 32 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-19 Mild adverse events during the total maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-20 Mild adverse events during the first 28 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-21 Mild adverse events during the last 24 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-22 Moderate adverse events during open-label phase by SOC and preferred term: open-label safety analysis set
- Table 3-23 Moderate adverse events during the total randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-24 Moderate adverse events during the first 28 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-25 Moderate adverse events during the last 32 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-26 Moderate adverse events during the total maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-27 Moderate adverse events during the first 28 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-28 Moderate adverse events during the last 24 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-29 Severe adverse events during open-label phase by SOC and preferred term: open-label safety analysis set



|------------------------------|-------------------|----------------|

- Table 3-30 Severe adverse events during the total randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-31 Severe adverse events during the first 28 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-32 Severe adverse events during the last 32 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-33 Severe adverse events during the total maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-34 Severe adverse events during the first 28 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-35 Severe adverse events during the last 24 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-36 Related adverse events during the open-label phase by SOC and preferred term: open-label safety analysis set
- Table 3-37 Related adverse events during the total randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-38 Related adverse events during the first 28 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-39 Related adverse events during the last 24 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-40 Related adverse events during the total maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-41 Related adverse events during the first 28 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-42 Related adverse events during the last 24 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-43 Adverse events during the open-label phase by causal relationship to IMP, SOC, and preferred term: open-label safety analysis set
- Table 3-44 Adverse events during the total randomised phase by causal relationship to IMP, SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-45 Adverse events during the first 28 weeks of the randomised phase by causal relationship to IMP, SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-46 Adverse events during the remaining 32 weeks of the randomised phase by causal relationship to IMP, SOC, preferred term, and randomised treatment: safety analysis set



|------------------------------|-------------------|----------------|

- Table 3-47 Adverse events during the total maintenance phase by causal relationship to IMP, SOC, preferred term, randomised treatment and rescue medication: safety analysis set
- Table 3-48 Adverse events during the first 28 weeks of the maintenance phase by causal relationship to IMP, SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-49 Adverse events during the remaining 24 weeks of the maintenance phase by causal relationship to IMP, SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-50 Serious adverse events during the open-label phase by SOC and preferred term: open-label safety analysis set
- Table 3-51 Serious adverse events during the total randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-52 Serious adverse events during the first 28 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-53 Serious adverse events during the last 32 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-54 Serious adverse events during the total maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-55 Serious adverse events during the first 28 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-56 Serious adverse events during the last 24 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-57 Non-serious adverse events during the open-label phase by SOC and preferred term: open-label safety analysis set
- Table 3-58 Non-serious adverse events during the total randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-59 Non-serious adverse events during the first 28 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-60 Non-serious adverse events during the last 32 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-61 Non-serious adverse events during the total maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-62 Non-serious adverse events during the first 28 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set



|------------------------------|-------------------|----------------|

- Table 3-63 Non-serious adverse events during the last 24 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-64 Frequent adverse events (>=1%) during the open-label phase by SOC and preferred term: open-label safety analysis set
- Table 3-65 Frequent adverse events (>=1% in any treatment group) during the total randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-66 Frequent adverse events (>=1% in any treatment group) during the first 28 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-67 Frequent adverse events (>=1% in any treatment group) during the last 32 weeks of the randomised phase by SOC, preferred term, and randomised treatment: safety analysis set
- Table 3-68 Frequent adverse events (>=1% in any treatment group) during the total maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-69 Frequent adverse events (>=1% in any treatment group) during the first 28 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-70 Frequent adverse events (>=1% in any treatment group) during the last 24 weeks of the maintenance phase by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set
- Table 3-71 Summary of rebounds occurring within 2 months after discontinuing open-label phase treatment or relapse treatment: safety analysis set
- Table 3-72 Summary of rebounds occurring within 2 months after discontinuation of maintenance treatment: safety analysis set
- Table 3-73 Physician's assessment of local safety and tolerability by visit in open-label phase: open-label safety analysis set
- Table 3-74 Shift table for physician's assessment of local safety and tolerability from start to end of open-label phase: open-label safety analysis set
- Table 3-75 Physician's assessment of local safety and tolerability by visit not related to relapse: safety analysis set
- Table 3-76 Physician's assessment of local safety and tolerability by visit for start of relapse: safety analysis set



|------------------------------|-------------------|----------------|

- Table 3-77 Physician's assessment of local safety and tolerability by visit for end of relapse: safety analysis set
- Table 3-78 Shift table for physician's assessment of local safety and tolerability from start of relapse to end of relapse by visit for start of relapse: safety analysis set
- Table 3-79 Subject's assessment of local safety and tolerability by visit in open-label phase: open-label safety analysis set
- Table 3-80 Shift table for subject's assessment of local safety and tolerability from start to end of open-label phase: open-label safety analysis set
- Table 3-81 Subject's assessment of local safety and tolerability by visit not related to relapse: safety analysis set
- Table 3-82 Subject's assessment of local safety and tolerability by visit for start of relapse: safety analysis set
- Table 3-83 Subject's assessment of local safety and tolerability by visit for end of relapse: safety analysis set
- Table 3-84 Shift table for subject's assessment of local safety and tolerability from start of relapse to end of relapse by visit for start of relapse: safety analysis set
- Table 3-85 Serum-cortisol concentration at time 0 and at 30 and 60 minutes after ACTH-challenge test by visit in open-label phase: open-label HPA analysis set
- Table 3-86 Individual data for subjects with serum-cortisol concentration ≤18 mcg/dL at either 30 minutes or 60 minutes after ACTH-challenge in the open-label phase: open-label HPA analysis set
- Table 3-87 Subjects with serum-cortisol concentration ≤18 mcg/dL at both 30 and 60 minutes after ACTH-challenge test in the open-label phase: open-label HPA analysis set
- Table 3-88 Serum-cortisol concentration at time 0 and at 30 and 60 minutes after ACTH-challenge test by visit: HPA analysis set
- Table 3-89 Individual data for subjects with serum-cortisol concentration ≤18 mcg/dL at either 30 minutes or 60 minutes after ACTH-challenge during the maintenance phase: HPA analysis set
- Table 3-90 Subjects with serum-cortisol concentration ≤18 mcg/dL at both 30 and 60 minutes after ACTH-challenge test during the maintenance phase: HPA analysis set
- Table 3-91 Serum-cortisol concentration at time 0 and at 30 and at 60 minutes after ACTH-challenge in the follow-up phase: HPA analysis set
- Table 3-92 Change in vital signs from baseline to end of open-label phase: open-label safety analysis set



|------------------------------|-------------------|----------------|

- Table 3-93 Change in vital signs from baseline to end of open-label phase: safety analysis set
- Table 3-94 Change in vital signs from randomisation to end of maintenance phase: safety analysis set
- Table 3-95 Change in vital signs from randomisation to end of maintenance phase for subjects discontinuing the trial before 6 months after randomisation: safety analysis set
- Table 3-96 Change in vital signs from randomisation to end of maintenance phase for subjects discontinuing the trial on or after 6 months after randomisation: safety analysis set
- Table 3-97 Change in vital signs from randomisation to end of maintenance phase for subjects completing the maintenance phase: safety analysis set
- Table 3-98 Change in laboratory parameters from baseline to end of open-label phase: open-label safety analysis set
- Table 3-99 Change in laboratory parameters from baseline to end of open-label phase: safety analysis set
- Table 3-100 Change in laboratory parameters from randomisation to end of maintenance phase: safety analysis set
- Table 3-101 Change in laboratory parameters from randomisation to end of maintenance phase for subjects discontinuing the trial before 6 months after randomisation: safety analysis set
- Table 3-102 Change in laboratory parameters from randomisation to end of maintenance phase for subjects discontinuing the trial on or after 6 months after randomisation: safety analysis set
- Table 3-103 Change in laboratory parameters from randomisation to end of maintenance phase for subjects completing the maintenance phase: safety analysis set
- Table 3-104 Shift table for laboratory parameter categories at baseline against end of openlabel phase: open-label safety analysis set
- Table 3-105 Shift table for laboratory parameter categories at baseline against end of openlabel phase: safety analysis set
- Table 3-106 Shift table for laboratory parameter categories at randomisation against end of maintenance phase: safety analysis set
- Table 3-107 Shift table for laboratory parameter categories at randomisation against end of maintenance phase for subjects discontinuing the trial before 6 months after randomisation: safety analysis set



|------------------------------|-------------------|----------------|

Table 3-108 Shift table for laboratory parameter categories at randomisation against end of maintenance phase for subjects discontinuing the trial on or after 6 months after randomisation: safety analysis set

Table 3-109 Shift table for laboratory parameter categories at randomisation against end of maintenance phase for subjects completing the maintenance phase: safety analysis set

Table 3-110 Shift table for albumin corrected serum calcium

#### **Figures**

Figure 3-1 Mean plot of serum-cortisol concentration at time 0, and at 30 and 60 minutes after ACTH-challenge test for visit 1 and visit 2; open-label HPA analysis set

Figure 3-2 Mean plot of serum-cortisol concentration at time 0, and at 30 and 60 minutes after ACTH-challenge test by treatment for visit 2, visit 8 and visit 15; HPA analysis set

#### **Patient Data Listings (Appendix 1)**

1-6 Randomisation

1-7 Subjects receiving Investigational Product from Specific Batches

#### **Patient Data Listings (Appendix 2)**

Appendix 2.1: Discontinued Subjects

Listing 1-1. Screening Failures

Listing 1-2. Reasons for Withdrawal from Trial in the Open-Label Phase

Listing 1-3. Reasons for Withdrawal from Trial in the Maintenance Phase

Listing 1-4. Subjects not entering the maintenance phase

Appendix 2.2: Protocol Deviations

Listing 2-1. Protocol Deviations

Listing 2-2. Comments from CRF



|------------------------------|-------------------|----------------|

Appendix 2.3: Trial Analysis Sets

Listing 3-1. Trial Analysis Set

Listing 3-2. Reasons for Exclusion from Analysis Set

Appendix 2.4: Demographic Data

Listing 4-1. Demographics

Listing 4-2. Date/Age of First Diagnosis of Psoriasis

Listing 4-3. Actual Trial Period

Listing 4-4. Medical History

Listing 4-5. Concurrent Diagnoses at Baseline

Listing 4-6. Concomitant Medication

Listing 4-7. Concurrent Procedures

Listing 4-8. Previous Anti-Psoriatic Treatment

Listing 4-9. Location of Psoriasis

Listing 4-10. Location of other Psoriasis

Appendix 2.5: Compliance and/or Investigational Product Concentration Data

Listing 5-1. Administration of Investigational Product

Listing 5-2. Drug Accountability



|------------------------------|-------------------|----------------|

# Appendix 2.6: Efficacy Data

Listing 6-1. Dermatology Quality Life Index

Listing 6-2. EQ-5D-5L-PSO

Listing 6-3. Work Productivity and Activity Impairment: Psoriasis (WPAI:PSO)

Listing 6-4. Psoriasis Symptom Inventory (PSI)

Listing 6-5. Physician's Global Assessment of Disease Severity (PGA)

Listing 6-6. Physician's Assessment of the Extent and Severity of Clinical Signs (m-PASI)

Listing 6-7. Investigator's Assessment of Body Surface Area (BSA)

Listing 6-8. Subject's Global Assessment of Disease Severity (SGA)

Listing 6-9. Target Lesion/Location Score

Listing 6-10. Number of Active Treatment Days during the Maintenance Phase

Listing 6-11. Time to First Relapse

Listing 6-12. Proportion of Days in Remission

Listing 6-13. Number of Relapses

#### Appendix 2.7: Safety Data

Listing 7-1. Deaths

Listing 7-2. Serious Adverse Events

Listing 7-3. Subjects withdrawn from trial due to Adverse Events

Listing 7-4. Severe Adverse Events

Listing 7-5. Adverse Events



|------------------------------|-------------------|----------------|

- Listing 7-6. Adverse Events Associated with Long Term Corticosteroid Use
- Listing 7-7. Subjects Assessment of Local Safety and Tolerability
- Listing 7-8. Investigators Assessment of Local Safety and Tolerability
- Listing 7-9. Rebounds
- Appendix 2.8: Listing of Laboratory Values by Subject
- Listing 8-1. Physical Examination, Abnormal Findings
- Listing 8-2. Laboratory Measurements
- Listing 8-3. Abnormal Laboratory Measurements
- Listing 8-4. Clinically Significant Laboratory Measurements
- Listing 8-5. Vital Signs
- Listing 8-6. Clinically Significant Vital Signs
- Listing 8-7. ACTH Laboratory Measurements



|------------------------------|-------------------|----------------|

## Additional Tables for Results Reporting in Clinical Trial Data Registries

- Table 4-1 Non-serious AEs occurring in ≥1% subjects by MedDRA primary SOC and preferred term: open-label safety analysis set
- Table 4-2 Non-serious AEs occurring in in ≥1% subjects by MedDRA primary SOC and preferred term: safety analysis set
- Table 4-3 Serious AEs by MedDRA primary SOC and preferred term: open-label safety analysis set
- Table 4-4 Serious AEs by MedDRA primary SOC and preferred term: safety analysis set
- Table 4-5 Subject enrolment and treatment assigned: enrolled subjects and subjects assigned treatment



|------------------------------|-------------------|----------------|

# Appendix II

Shells



|------------------------------|-------------------|----------------|

| Shell 1: Disposition of subjects in the open-label phase: enrolled subjects |
|---|
| Shell 2: Disposition of subjects in the randomised phase: randomised subjects |
| Shell 3: Reasons for leaving the trial during the open-label phase by last visit attended: enrolled subjects |
| Shell 4: Reasons for leaving the trial during the maintenance phase by last visit attended: randomised subjects |
| Shell 5: <continuous variable(s)="">: open-label safety analysis set</continuous> |
| Shell 6: <continuous variable(s)="">: randomised subjects</continuous> |
| Shell 7: <continuous variable(s)=""> by <strata>: open-label safety analysis set</strata></continuous> |
| Shell 8: <continuous variable(s)=""> by <strata>: randomised subjects</strata></continuous> |
| Shell 9: <categorical variable(s)="">: open-label safety analysis set</categorical> |
| Shell 10: <categorical variable(s)="">: randomised subjects</categorical> |
| Shell 11: <categorical variable(s)=""> by <strata>: open-label safety analysis set</strata></categorical> |
| Shell 12: <categorical variable(s)=""> by <strata>: randomised subjects</strata></categorical> |
| Shell 13: Location of psoriasis and location of other psoriasis at baseline: open-label safety analysis set |
| Shell 14: Location of psoriasis and location of other psoriasis at baseline: randomised subjects |
| Shell 15: Concomitant medication: open-label safety analysis set |
| Shell 16: Concomitant medication: randomised subjects |
| Shell 17: Previous and latest systemic anti-psoriatic treatment: open-label safety analysis set |
| Shell 18: Previous and latest systemic anti-psoriatic treatment: randomised subjects |
| Shell 19: Concurrent diagnoses at baseline: open-label safety analysis set |
| Shell 20: Summary of observation types for time to first relapse – sensitivity analysis: <full analysis="" per="" protocol="" set=""></full> |



|------------------------------|-------------------|----------------|

| Shell 21: Censored and uncensored observations for time to first relapse: <full analysis="" per="" protocol="" set=""></full> |
|---|
| Shell 22: Number of subjects at risk of first relapse by scheduled visit: <full analysis="" per="" protocol="" set=""></full> |
| Shell 23:< Statistical/Sensitivity> analysis of time to first relapse: <full analysis="" per="" protocol="" set=""></full> |
| Shell 24: Percentiles from estimated survival curves < - sensitivity analysis>: <full analysis="" per="" protocol="" set=""></full> |
| Shell 25: Comparison of proportions of subjects still at risk of first relapse at 26 weeks and 52 weeks after randomisation: full analysis set |
| Shell 26: Observed proportion of days in remission: <full analysis="" per="" protocol="" set=""></full> |
| Shell 27: <statistical sensitivity=""> analysis of proportion of days in remission: <full analysis="" per="" protocol="" set=""></full></statistical> |
| Shell 28: Number of relapses during maintenance phase: <full analysis="" per="" protocol="" set=""></full> |
| Shell 29: <statistical sensitivity=""> analysis of number of relapses during maintenance phase &lt;(negative binomial model)&gt;: <full analysis="" per="" protocol="" set=""> 94</full></statistical> |
| Shell 30: <xxx> by visit in open-label phase: open-label safety analysis set95</xxx> |
| Shell 31: <change change="" percent=""> in <xxx> from start to end of open-label phase: open-label safety analysis set</xxx></change> |
| Shell 32: <xxx> by visit not related to relapse: full analysis set</xxx> |
| Shell 33: <xxx> by visit for start of relapse: full analysis set</xxx> |
| Shell 34: <xxx> by visit for end of relapse: full analysis set</xxx> |
| Shell 35: <change change="" percent=""> in <xxx> from start of relapse to end of relapse by visit for start of relapse: full analysis set</xxx></change> |
| Shell 36: <physician's subject's=""> global assessment of disease severity by visit in open-label phase: open-label safety analysis set</physician's> |
| Shell 37: Shift table for <physician's subject's=""> global assessment of disease severity from start to end of open-label phase: open-label safety analysis set</physician's> |



|------------------------------|-------------------|----------------|

| Shell 38: | <physician's subject's=""> Global Assessment of Disease Severity by visit not relate<br/>to relapse: full analysis set</physician's> | |
|---|---|---|
| Shell 39: | <physician's subject's=""> global assessment of disease severity by visit for start of relapse: full analysis set</physician's> | |
| Shell 40: | <physician's subject's=""> global assessment of disease severity by visit for end of relapse: full analysis set</physician's> | |
| Shell 41: | Shift table for <physician's subject's=""> global assessment of disease severity from start of relapse to end of relapse by visit for start of relapse: full analysis set</physician's> | |
| Shell 42: | WPAI:PSO by visit: full analysis set | 07 |
| Shell 43: | WPAI:PSO by visit: open-label safety analysis set | 09 |
| Shell 44: | Total PSI score during open-label phase; open-label safety analysis set 1 | 11 |
| Shell 45: | <change change="" percent=""> in total PSI score from start to end of open-label phase open-label safety analysis set</change> | |
| Shell 46: | Total PSI score for time on rescue medication and time in remission during the firs 28 weeks of the maintenance phase: full analysis set | |
| Shell 47: | Statistical analysis of PSI: full analysis set | 13 |
| Shell 48: | Statistical analysis of DLQI: full analysis set | 15 |
| Shell 49: | Shift table for EQ-5D-5L from start to end of open-label phase: open-label safety analysis set | 16 |
| Shell 50: | Shift table for EQ-5D-5L-PSO dimensions from start of relapse to end of relapse by visit for start of relapse: maintenance full analysis set | • |
| Shell 51: | Subjects in remission by scheduled visit: full analysis set | 23 |
| Shell 52: | Subjects achieving clear or almost clear after treatment of relapse by number of relapses: full analysis set | 24 |
| Shell 53: | Target lesion/location score by visit in open-label phase: open-label safety analysis set | |
| Shell 54: | Shift table for target lesion/location score from start to end of open-label phase: open-label safety analysis set | <b>2</b> 6 |
| Shell 55: | Target lesion/location score by visit not related to relapse: full analysis set 1 | 27 |



|------------------------------|-------------------|----------------|

| Shell 56: T | Target lesion/location score by visit for start of relapse: full analysis set | 28 |
|---|---|---|
| Shell 57: T | Carget lesion/location score by visit for end of relapse: full analysis set | 30 |
| Shell 58: S | thift table for target lesion/location score from start of relapse to end of relapse by visit for start of relapse: full analysis set | |
| Shell 59: C | Overall summary of adverse events during open-label phase: open-label safety analysis set | 34 |
| Shell 60: C | Overall summary of adverse events during <xxx> by randomised treatment: safe analysis set</xxx> | - |
| Shell 61: C | Overall summary of adverse events during <xxx> by randomised treatment and rescue medication: safety analysis set</xxx> | 36 |
| Shell 62: < | XXXX> during the open-label phase by SOC and preferred term: open-label safety analysis set | |
| Shell 63: < | XXX> during <xxx> by SOC, preferred term, and randomised treatment: safety analysis set</xxx> | |
| Shell 64: < | XXX> during <xxx> by SOC, preferred term, randomised treatment, and rescumedication: safety analysis set</xxx> | |
| Shell 65: A | Adverse events during the open-label phase by causal relationship to IMP, SOC, as preferred term: open-label safety analysis set | |
| Shell 66: A | Adverse events during <xxx> by causal relationship to IMP, SOC, preferred term and randomised treatment: safety analysis set</xxx> | |
| Shell 67: A | Adverse events during <xxx> by causal relationship to IMP, SOC, preferred term randomised treatment, and rescue medication: safety analysis set</xxx> | - |
| Shell 68: P | Physician's assessment of local safety and tolerability by visit in open-label phase open-label safety analysis set | |
| Shell 69: S | chift table for physician's assessment of local safety and tolerability from start to end of open-label phase: open-label safety analysis set | 45 |
| Shell 70: P | Physician's assessment of local safety and tolerability by visit not related to relaps safety analysis set | |
| Shell 71: P | Physician's assessment of local safety and tolerability by visit for start of relapse: safety analysis set | 47 |


|------------------------------|-------------------|----------------|

| Shell | 2: Physician's assessment of local safety and tolerability by visit for end of relapse: safety analysis set |
|---|---|
| Shell | 3: Shift table for physician's assessment of local safety and tolerability from start of relapse to end of relapse by visit for start of relapse: safety analysis set 14 |
| Shell | 4: Subject's assessment of local safety and tolerability by visit in open-label phase: open-label safety analysis set |
| Shell | 5: Shift table for subject's assessment of local safety and tolerability from start to end of open-label phase: open-label safety analysis set |
| Shell | 6: Subject's assessment of local safety and tolerability by visit not related to relapse: safety analysis set |
| Shell | 7: Subject's assessment of local safety and tolerability by visit for start of relapse: safety analysis set |
| Shell | 8: Subject's assessment of local safety and tolerability by visit for end of relapse: safety analysis set |
| Shell | 9; Shift table for subject's assessment of local safety and tolerability from start of relapse to end of relapse by visit for start of relapse: safety analysis set 15 |
| Shell | 0: Change in vital signs from baseline to end of open-label phase: open-label safety analysis set |
| Shell | 1: Change in vital signs from randomisation to end of maintenance phase <for subject="" xxx="">: safety analysis set</for> |
| Shell | 2: Change in laboratory parameters from baseline to end of open-label phase: open-label safety analysis set |
| Shell | 3: Change in laboratory parameters from randomisation to end of maintenance phase <for subjects="" xxx="">: safety analysis set</for> |
| Shell | 4: Shift table for laboratory parameter categories at baseline against end of open-label phase: open-label safety analysis set |
| Shell | 5: Shift table for laboratory parameter categories at randomisation against end of maintenance phase <for subjects="" xxx="">: safety analysis set</for> |
| Shell | 6: Compliance with treatment instructions during open-label treatment phase: open-label safety analysis |
| Shell | 7: Compliance with treatment instructions during maintenance phase excluding period of treatment with rescue medication: maintenance phase safety analysis set 16 |



|------------------------------|-------------------|----------------|

| Shell 88: Compliance with treatment instructions during periods of treatment with rescue medication: maintenance phase safety analysis set |
|---|
| Shell 89: Duration of exposure during the open-label treatment phase: open-label safety analysis set |
| Shell 90: Duration of exposure during the maintenance phase: safety analysis set |
| Shell 91: Amount of investigational medicinal product used during open-label treatment phase: open-label safety analysis set |
| Shell 92: Amount of investigational medicinal product used during maintenance phase: safety analysis set |
| Shell 93: Cumulative amount of investigational medical product used up to scheduled visits: maintenance phase safety analysis set |
| Shell 94: Serum-cortisol concentration at time 0 and at 30 and at 60 minutes after ACTH-challenge test by visit: open-label HPA analysis set |
| Shell 95: Individual data for subjects with serum cortisol concentration ≤18 mcg/dL at either 30 minutes or 60 minutes after ACTH-challenge: open-label HPA analysis set. 169 |
| Shell 96: Subjects with serum cortisol concentration ≤18 mcg/dL at both 30 and 60 minutes after ACTH-challenge in open-label phase; open-label HPA analysis set 170 |
| Shell 97: Serum-cortisol concentration at time 0 and at 30 and at 60 minutes after ACTH-challenge test by visit: HPA analysis set |
| Shell 98: Subjects with serum cortisol concentration ≤18 mcg/dL at both 30 and 60 minutes after ACTH-challenge in maintenance phase; HPA analysis set |
| Shell 99: Individual data for subjects with serum cortisol concentration ≤18 mcg/dL at either 30 minutes or 60 minutes after ACTH-challenge: HPA analysis set |
| Shell 100: Serum-cortisol concentration at time 0 and at 30 and at 60 minutes after ACTH-challenge in the follow-up phase: HPA analysis set |
| Shell 101: Summary of rebounds occurring within 2 months after discontinuing open-label phase treatment or relapse treatment: safety analysis set |
| Shell 102: Summary of rebounds occurring within 2 months after discontinuing of maintenance treatment: safety analysis set |



|------------------------------|-------------------|----------------|

Shell 1: Disposition of subjects in the open-label phase: enrolled subjects

| | Open-label LEO 90100 (n=xxx) | |
|---|---|---|
| | N (%) | Visit 2 (Week 4)<br>attendance<br>Yes / No |
| nrolled subjects | xx(xx.x) | xx / xx |
| Randomised subjects | xx(xx.x) | xx / xx |
| Withdrawn from trial during open-label phase | xx(xx.x) | xx / xx |
| Adverse event | xx(xx.x) | xx / xx |
| Death | xx(xx.x) | xx / xx |
| Lost to follow-up | xx(xx.x) | xx / xx |
| Withdrawal by subject | xx(xx.x) | xx / xx |
| Lack of efficacy | xx(xx.x) | xx / xx |
| Subject did not achieve treatment success | | |
| after initial 4 weeks treatment | xx(xx.x) | xx / xx |
| Other | xx(xx.x) | xx / xx |

N: Number of subjects, %: Percentage of subjects.

Shell 2: Disposition of subjects in the randomised phase: randomised subjects

| | All randomised subjects (n=xxx) | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|---|
| | N (%) | N (%) | N (%) |
| Randomised subjects | xx (100.0) | xx (100.0) | xx (100.0) |
| Full analysis set | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Safety analysis set | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Per protocol analysis set | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawn from trial during randomis | ed | | |
| phase | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal by subject | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lack of efficacy | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject did not achieve treatment success after initial 4 weeks | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject not clear or almost clear after treatment of relapse | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N: Number of subjects, %: Percentage of subjects.

<sup>1)</sup> Subjects randomised in error.



|------------------------------|-------------------|----------------|

Shell 3: Reasons for leaving the trial during the open-label phase by last visit attended: enrolled subjects

| | Open-label LEO 90100 |
|-------------------------------------------------|----------------------|
| | (n=xxx) |
| Reason for withdrawal | |
| Last visit attended | N (%) |
| Adverse event | |
| Visit 1 | xx(xx.x) |
| Visit 2 | xx(xx.x) |
| Death | |
| Visit 1 | xx(xx.x) |
| Visit 2 | xx(xx.x) |
| Lost to follow-up | |
| Visit 1 | xx(xx.x) |
| Visit 2 | xx(xx.x) |
| Withdrawal by subject | |
| Visit 1 | xx(xx.x) |
| Visit 2 | xx(xx.x) |
| Lack of efficacy | |
| Visit 1 | xx(xx.x) |
| Visit 2 | xx(xx.x) |
| Subject did not achieve treatment success after | |
| initial 4 weeks treatment | |
| Visit 1 | xx(xx.x) |
| Visit 2 | xx(xx.x) |
| Other | |
| Visit 1 | xx(xx.x) |
| Visit 2 | xx(xx.x) |

N: Number of subjects, %: Percentage of subjects.



|------------------------------|-------------------|----------------|

Shell 4: Reasons for leaving the trial during the maintenance phase by last visit attended: randomised subjects

| | All randomised<br>subjects<br>(n=xxx) | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|---|
| Reason for withdrawal<br>Last visit attended | N (%) | N (%) | N (%) |
| Adverse event | | | |
| Visit 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| • • • | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 15 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | | | |
| Visit 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit 15 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | | | |
| <as above=""></as> | | | |
| Subject did not achieve treatmer<br>success after initial 4 weeks | nt | | |
| - | nt | | |
| success after initial 4 weeks | nt | | |
| <pre>success after initial 4 weeks treatment¹ <as above=""></as></pre> | nt | | |
| success after initial 4 weeks treatment <sup>1</sup> | nt | | |
| success after initial 4 weeks treatment <sup>1</sup> <as above=""></as> | | xx (xx.x) | xx (xx.x) |
| success after initial 4 weeks treatment¹ <as above=""> Other</as> | xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| success after initial 4 weeks treatment¹ <as above=""> Other Visit 2 Visit 3</as> | xx (xx.x)<br>xx (xx.x) | xx (xx.x) | xx (xx.x) |
| success after initial 4 weeks treatment¹ <as above=""> Other Visit 2</as> | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| success after initial 4 weeks treatment¹ <as above=""> Other Visit 2 Visit 3 Visit 4 Visit 5</as> | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| success after initial 4 weeks treatment¹ <as above=""> Other Visit 2 Visit 3 Visit 4</as> | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| success after initial 4 weeks treatment¹ <as above=""> Other Visit 2 Visit 3 Visit 4 Visit 5 Visit 6</as> | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

N: Number of subjects, %: Percentage of subjects.

1) Subjects randomised in error.



|------------------------------|-------------------|----------------|

Shell 5: <Continuous variable(s)>: open-label safety analysis set

| | Open-label LEO 90100<br>(n=xxx) |
|--------------------|---------------------------------|
| nt var 1> | |
| Jumber of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | XX.X;XX.X |
| Min;Max | xx.x;xx.x |
| ont var K> | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min; Max | XX.X;XX.X |

Shell 6: <Continuous variable(s)>: randomised subjects

| | All randomised | | |
|---|---|---|---|
| | subjects | LEO 90100 | Vehicle |
| | (n=xxx) | (n=xxx) | (n=xxx) |
| Cont var 1> | | | |
| Number of subjects | xxx | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X | xx.x;xx.x |
| Min; Max | xx.x; xx.x | xx.x; xx.x | xx.x;xx.x |
| <pre><cont k="" var=""></cont></pre> | | | |
| Number of subjects | xxx | xxx | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |



|------------------------------|-------------------|----------------|

### Shell 7: <Continuous variable(s)> by <strata>: open-label safety analysis set

| | Open-label LEO 90100 |
|--------------------------------------|----------------------|
| | (n=xxx) |
| <pre><cont 1="" var=""></cont></pre> | |
| <pre><strata 1=""></strata></pre> | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | XX.X;XX.X |
| Min; Max | xx.x;xx.x |
| ••• | |
| <strata m=""></strata> | |
| Number of subjects | XXX |
| Mean(SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min;Max | xx.x;xx.x |
| <cont k="" var=""></cont> | |
| <strata 1=""></strata> | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min;Max | xx.x; xx.x |
| ••• | |
| <strata m=""></strata> | |
| Number of subjects | XXX |
| Mean(SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min; Max | xx.x;xx.x |



|------------------------------|-------------------|----------------|

Shell 8: <Continuous variable(s)> by <strata>: randomised subjects

| | All randomised subjects | LEO 90100<br>(n=xxx) | Vehicle |
|---|---|---|---|
| | (n=xxx) | | (n=xxx) |
| cont var 1> | | | |
| <pre><strata 1=""></strata></pre> | | | |
| Number of subjects | xxx | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX • X |
| Q1;Q3 | xx.x;xx.x | xx.x; xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x; xx.x | xx.x;xx.x |
| <strata m=""></strata> | | | |
| Number of subjects | XXX | xxx | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | XX.X;XX.X |
| Min; Max | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |
| • | | | |
| cont var K><br><strata 1=""></strata> | | | |
| Number of subjects | xxx | xxx | xxx |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X | XX.X;XX.X |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x; xx.x |
| <strata m=""></strata> | | | |
| Number of subjects | XXX | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X | xx.x |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |



|------------------------------|-------------------|----------------|

## Shell 9: <Categorical variable(s)>: open-label safety analysis set

| | Open-label LEO 90100 (n=xxx) |
|--------------------|------------------------------|
| Ccat var 1> | |
| Number of subjects | XXX |
| Category 1 | xxx (xx.x%) |
| ••• | xxx (xx.x%) |
| Category $k_1$ | xxx (xx.x%) |
| Ccat var K> | |
| Number of subjects | XXX |
| Category 1 | xxx (xx.x%) |
| ••• | xxx (xx.x%) |
| Category $k_K$ | xxx (xx.x%) |

## Shell 10: <Categorical variable(s)>: randomised subjects

| | All r | andomised | | | | |
|---|---|---|---|---|---|---|
| | su | bjects | LEC | 90100 | 7 | /ehicle |
| | (r | =xxx) | (r | n=xxx) | | (n=xxx) |
| Cat var 1> | | | | | | |
| Number of subjects | | XXX | | XXX | | XXX |
| Category 1 | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| ••• | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Category $k_1$ | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| <pre><cat k="" var=""></cat></pre> | | | | | | |
| Number of subjects | | XXX | | XXX | | XXX |
| Category 1 | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| ••• | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| $Category k_K$ | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |



|------------------------------|-------------------|----------------|

# Shell 11: <Categorical variable(s)> by <strata>: open-label safety analysis set

| | Open-label LEO 90100<br>(n=xxx) |
|------------------------------------|---------------------------------|
| 45.4 | |
| <pre><cat 1="" var=""></cat></pre> | |
| <strata 1=""></strata> | |
| Number of subjects | XXX |
| Category 1 | xxx (xx.x%) |
| | xxx (xx.x%) |
| Category $k_1$ | xxx (xx.x%) |
| ••• | |
| <strata m=""></strata> | |
| Number of subjects | XXX |
| Category 1 | xxx (xx.x%) |
| • • • | xxx (xx.x%) |
| Category $k_1$ | xxx (xx.x%) |
| <cat k="" var=""></cat> | |
| <strata 1=""></strata> | |
| Number of subjects | XXX |
| Category 1 | xxx (xx.x%) |
| ••• | xxx (xx.x%) |
| Category $k_K$ | xxx (xx.x%) |
| <strata m=""></strata> | |
| Number of subjects | XXX |
| Category 1 | xxx (xx.x%) |
| | xxx (xx.x%) |
| Category k <sub>K</sub> | xxx (xx.x%) |



|------------------------------|-------------------|----------------|

Shell 12: <Categorical variable(s)> by <strata>: randomised subjects

| | All randomised subjects | LEO 90100<br>(n=xxx) | Vehicle |
|---|---|---|---|
| | (n=xxx) | (II—AAA) | (n=xxx) |
| cat var 1> | | | |
| <strata 1=""></strata> | | | |
| Number of subjects | xxx | ××× | XXX |
| Category 1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| ••• | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Category $k_1$ | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| • • • | | | |
| <strata m=""></strata> | | | |
| Number of subjects | xxx | xxx | xxx |
| Category 1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| ••• | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Category $k_{\mathtt{M}}$ | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| cat var K> | | | |
| <strata 1=""></strata> | | | |
| Number of subjects | XXX | XXX | XXX |
| Category 1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| • • • | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Category $k_1$ | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <strata m=""></strata> | | | |
| Number of subjects | XXX | XXX | XXX |
| Category 1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| ••• | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| $Category k_{M}$ | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



|------------------------------|-------------------|----------------|

Shell 13: Location of psoriasis and location of other psoriasis at baseline: open-label safety analysis set

| | Open-label LEO 90100 (n=xxx) |
|----------------------------|------------------------------|
| ocation of psoriasis | |
| Number of subjects | XXX |
| Abdomen | xxx (xx.x%) |
| Chest | xxx (xx.x%) |
| Elbow | xxx (xx.x%) |
| Forearm incl. hand | xxx (xx.x%) |
| Knee | xxx (xx.x%) |
| Lower back | xxx (xx.x%) |
| Lower leg incl. foot | xxx (xx.x%) |
| Neck | xxx (xx.x%) |
| Upper arm | xxx (xx.x%) |
| Upper back | xxx (xx.x%) |
| Upper leg | xxx (xx.x%) |
| ocation of other psoriasis | |
| Number of subjects | XXX |
| Face | xxx (xx.x%) |
| Genitals | xxx (xx.x%) |
| Nails | xxx (xx.x%) |
| Palms | xxx (xx.x%) |
| Scalp | xxx (xx.x%) |
| Skin folds | xxx (xx.x%) |
| Soles | xxx (xx.x%) |



|------------------------------|-------------------|----------------|

Shell 14: Location of psoriasis and location of other psoriasis at baseline: randomised subjects

| Number of subjects xxx | | All randomised subjects (n=xxx) | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|---|---|
| Abdomen | ocation of psoriasis | | | |
| Chest | Number of subjects | xxx | XXX | XXX |
| Elbow | Abdomen | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Forearm incl. hand | Chest | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Knee xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Lower back xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Lower leg incl. foot xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Neck xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Upper arm xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Upper back xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Upper leg xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Number of subjects Xxx xxx xxx Face xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Genitals xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Nails xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Palms xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Scalp xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | Elbow | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Lower back | Forearm incl. hand | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Lower leg incl. foot | Knee | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Neck xxx (xx.x%) xxx (xx.x%) | Lower back | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Upper arm xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Upper back xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Upper leg xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Accation of other psoriasis Xxx xxx xxx Number of subjects Xxx xxx xxx Face xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Genitals xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Nails xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Palms xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Scalp xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | Lower leg incl. foot | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Upper back xxx (xx.x%) xxx (xx.x%) | Neck | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Upper leg xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Location of other psoriasis Xxx xxx xxx Number of subjects Xxx xxx xxx xxx Face xxx (xx.x%) xxx (xx | Upper arm | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Accation of other psoriasis Xxx xxx xxx< | Upper back | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Number of subjects Xxx xxx xxx Face xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Genitals xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Nails xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Palms xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Scalp xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | Upper leg | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Face xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Genitals xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Nails xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Palms xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Scalp xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | <del>-</del> | | | |
| Genitals xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Nails xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Palms xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Scalp xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | 3 | | | |
| Nails xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Palms xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Scalp xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | | , | , , , | , |
| Palms xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Scalp xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | 00111100110 | , , | , , , | , , |
| Scalp xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | | , | | , , |
| Skin folds xxx (xx.x%) xxx (xx.x%) xxx (xx.x%) | | , , | , , | , , |
| ( | 1 | ` ' | , , | , |
| | Skin folds<br>Soles | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |

Subjects may appear in more than one category.



|------------------------------|-------------------|----------------|

Shell 15: Concomitant medication: open-label safety analysis set

| Open-label LEO 9(n=xxx) | |
|-------------------------|------------------------|
| Medication (ATC code) | Number of subjects (%) |
| ACT1 | xx (xx.x) |
| ACT2 | xx(xx.x) |
| ACT3 | xx(xx.x) |
| ACT4 | xx(xx.x) |
| Preferred drug name | xx(xx.x) |

ATC: Anatomical Therapeutic Chemical Classification System.

Shell 16: Concomitant medication: randomised subjects

| | All randomised subjects (n=xxx) | LEO 90100 (n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|---|
| Medication (ATC code) | Number of subjects (%) | Number of subjects (%) | Number of subjects (%) |
| ACT1 | xx (xx.x) | xx(xx.x) | xx(xx.x) |
| ACT2 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| ACT3 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| ACT4 | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Preferred drug name | xx(xx.x) | xx(xx.x) | xx(xx.x) |

ATC: Anatomical Therapeutic Chemical Classification System.



| Tria | al ID: <b>LP0053-1004</b> | Date: 15-JUL-2019 | Version: 1.0 |
|------|---------------------------|-------------------|----------------|

Shell 17: Previous and latest systemic anti-psoriatic treatment: open-label safety analysis set

| | Open-label LEO 90100 (n=xxx) |
|-------------------------------------------|------------------------------|
| revious systemic anti-psoriatic treatment | |
| Number of subjects | XXX |
| Acitretin | xxx (xx.x%) |
| Adalimumab | xxx (xx.x%) |
| Apremilast | xxx (xx.x%) |
| Cyclosporin | xxx (xx.x%) |
| Etanercept | xxx (xx.x%) |
| Infliximab | xxx (xx.x%) |
| Methotrexate | xxx (xx.x%) |
| Phototherapy | xxx (xx.x%) |
| Secukinumab | xxx (xx.x%) |
| Ustekinumab | xxx (xx.x%) |
| Other | xxx (xx.x%) |
| atest systemic anti-psoriatic treatment | |
| Number of subjects | XXX |
| Acitretin | xxx (xx.x%) |
| Adalimumab | xxx (xx.x%) |
| Apremilast | xxx (xx.x%) |
| Cyclosporin | xxx (xx.x%) |
| Etanercept | xxx (xx.x%) |
| Infliximab | xxx (xx.x%) |
| Methotrexate | xxx (xx.x%) |
| Phototherapy | xxx (xx.x%) |
| Secukinumab | xxx (xx.x%) |
| Ustekinumab | xxx (xx.x%) |

Subjects may appear in more than one category.



|------------------------------|-------------------|----------------|

Shell 18: Previous and latest systemic anti-psoriatic treatment: randomised subjects

| | All randomised<br>subjects<br>(n=xxx) | | LEO 90100<br>(n=xxx) | | Vehicle<br>(n=xxx) | |
|---|---|---|---|---|---|---|
| Previous systemic anti-psoriatic | | | | | | |
| treatment | | | | | | |
| Number of subjects | | xxx | | xxx | | xxx |
| Acitretin | xxx | | ~~~ | (xx.x%) | ~~~ | (xx.x%) |
| Adalimumab | XXX | (xx.x%) | | (xx.x%) | | (xx.x%) |
| Apremilast | XXX | (xx.x%) | | (xx.x%) | | (xx.x%) |
| Cyclosporin | XXX | (xx.x%) | | (xx.x%) | | (xx.x%) |
| Etanercept | XXX | (xx.x%) | XXX | (xx.x%) | | (xx.x%) |
| Infliximab | XXX | (xx.x%) | XXX | (xx.x%) | | (xx.x%) |
| Methotrexate | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Phototherapy | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Secukinumab | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Ustekinumab | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Other | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| | | , | | , | | |
| Latest systemic anti-psoriatic | | | | | | |
| Number of subjects | | xxx | | xxx | | xxx |
| Acitretin | V V V | (xx.x%) | V V V | (xx.x%) | V V V | (xx.x%) |
| Adalimumab | XXX | (xx.x%) | | (xx.x%) | | (xx.x%) |
| Apremilast | XXX | (xx.x%) | XXX | (xx.x%) | | (xx.x%) |
| Cyclosporin | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Etanercept | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Infliximab | XXX | (xx.x%) | | (xx.x%) | XXX | |
| Methotrexate | XXX | (xx.x%) | | (xx.x%) | XXX | |
| Phototherapy | XXX | (xx.x%) | | (xx.x%) | XXX | |
| Secukinumab | XXX | (xx.x%) | | (xx.x%) | | (xx.x%) |
| Ustekinumab | XXX | (xx.x%) | | (xx.x%) | | (xx.x%) |
| Other | XXX | (xx.x%) | | (xx.x%) | | (xx.x%) |

Subjects may appear in more than one category.



|------------------------------|-------------------|----------------|

## Shell 19: Concurrent diagnoses at baseline: open-label safety analysis set

| | Open-label LEO 90100 |
|-------------------------------------|----------------------|
| System Organ Class (SOC) | (n=xxx) |
| Preferred term | N (%) |
| Total number of diagnoses | xxx |
| Number of subjects with a diagnosis | xxx |
| SOC 1 | xxx(xx.x) |
| Preferred term 1 | xxx(xx.x) |
| ••• | ••• |
| Preferred term $k_1$ | xxx(xx.x) |
| SOC 2 | xxx(xx.x) |
| Preferred term 1 | xxx(xx.x) |
| $\dots$ Preferred term $k_2$ | <br>xxx (xx.x) |
| 110101104 001 1.2 | ( / |
| ••• | |
| SOC M | xxx(xx.x) |
| Preferred term 1 | xxx(xx.x) |
| ••• | • • • |
| Preferred term $k_{	exttt{M}}$ | xxx(xx.x) |



|------------------------------|-------------------|----------------|

Shell 20: Summary of observation types for time to first relapse – sensitivity analysis: <full analysis set / per protocol analysis set>

| | LEO 90100<br>(n=xxx)<br>Subjects (%) | Vehicle<br>(n=xxx)<br>Subjects (%) |
|---|---|---|
| umber of subjects with: | | |
| No relapses <sup>1</sup> | xxx ( xx.x%) | xxx ( xx.x%) |
| Relapse confirmed at a scheduled visit <sup>2</sup> | xxx ( xx.x%) | xxx ( xx.x%) |
| Relapse confirmed at an unscheduled visit <sup>3</sup> | xxx (xx.x%) | xxx ( xx.x%) |
| otal | xxx (100.0%) | xxx (100.0%) |

<sup>1)</sup> No relapses corresponds to right-censored observations.

Shell 21: Censored and uncensored observations for time to first relapse: <full analysis set / per protocol analysis set>

| | LEO 90100<br>(n=xxx)<br>Subjects (%) | Vehicle<br>(n=xxx)<br>Subjects (%) |
|---|---|---|
| Number of subjects with: | | |
| | / 0.1 | / ) |
| No relapses1 | xxx ( xx.x%) | xxx ( xx.x%) |
| No relapses <sup>1</sup> Relapses confirmed <sup>2</sup> | xxx ( xx.x%)<br>xxx ( xx.x%) | xxx ( xx.x%) |

<sup>1)</sup> No relapses corresponds to censored observations.



<sup>2)</sup> Relapse confirmed at a scheduled visit corresponds to interval censored observations.

<sup>3)</sup> Relapse confirmed at an unscheduled visit corresponds to exact observations.

<sup>2)</sup> Relapses confirmed correspond to uncensored observations.

|------------------------------|-------------------|----------------|

Shell 22: Number of subjects at risk of first relapse by scheduled visit: <full analysis set / per protocol analysis set>

| | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|
| Time relative to randomisation | Subjects (%1) | Subjects (%1) |
| Randomisation, Visit 2 | | |
| Number of subjects attending the visit | XXX | XXX |
| Number of subjects still at risk of first relapse | xxx (xx.x%) | xxx (xx.x%) |
| 28 days², Visit 3 | | |
| Number of subjects attending the visit | XXX | XXX |
| Number of subjects still at risk of first relapse | xxx (xx.x%) | xxx (xx.x%) |
| 364 days <sup>2</sup> , Visit 15 | | |
| Number of subjects attending the visit | XXX | XXX |
| Number of subjects still at risk of first relapse | xxx (xx.x%) | xxx (xx.x%) |

<sup>1)</sup> Percents are calculated as number of subjects still at risk of first relapse divided by number of subjects in the <full analysis set / per protocol analysis set> multiplied by 100.

Shell 23:< Statistical/Sensitivity> analysis of time to first relapse: <full analysis set / per protocol analysis set>

| | LEO 90100 vs. vehicle |
|--------------------------------------------|-----------------------|
| Number of subjects randomised to LEO 90100 | xxx |
| Number of subjects randomised to Vehicle | xxx |
| Hazard ratio | xx.xx |
| 95% CI | xx.xx-xx.xx |
| p-value | 0.xxx or <0.001 |

Estimates are obtained from a proportional hazards model with treatment group, pooled sites, and disease severity at maintenance baseline (determined by PGA) as factors. <The model incorporates interval censoring>.



<sup>2)</sup> Number of days since randomisation assuming the scheduled visits happen every fourth week.

|------------------------------|-------------------|----------------|

Shell 24: Percentiles from estimated survival curves < - sensitivity analysis>: <full analysis set / per protocol analysis set>

| Percentiles | LEO 90100 | Vehicle |
|----------------------------------------------|-----------|---------|
| Estimated number of days after randomisation | (n=xxx) | (n=xxx) |
| 25% | | |
| Estimate | XXX | XXX |
| 95% CI | xxx-xxx | xxx-xxx |
| 50% | | |
| Estimate | XXX | XXX |
| 95% CI | XXX-XXX | XXX-XXX |
| 75% | | |
| Estimate | XXX | XXX |
| 95% CI | XXX-XXX | xxx-xxx |

The percentiles are obtained from the estimated survival curves. The percentiles describe the number of days after randomisation until a certain percent of subjects are no longer at risk. <The survival curves are estimated using a non-parametric maximum likelihood estimator, namely the Turnbull self-consistency algorithm.>



|------------------------------|-------------------|----------------|

Shell 25: Comparison of proportions of subjects still at risk of first relapse at 26 weeks and 52 weeks after randomisation: full analysis set

| Weeks after randomisation Proportion of subjects | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) | p-value <sup>1</sup> |
|---|---|---|---|
| 26 weeks | | | |
| Estimate | XX.XX | XX.XX | 0.xxx or <0.001 |
| 95% CI | xx.xx-xx.xx | xx.xx-xx.xx | |
| 52 weeks | | | |
| Estimate | XX.XX | XX.XX | 0.xxx or <0.001 |
| 95% CI | xx.xx-xx.xx | xx.xx-xx.xx | |

The proportion are obtained from the estimated survival curves.



<sup>1)</sup> The p-value is obtained from a z-test comparing LEO 90100 to vehicle.

|------------------------------|-------------------|----------------|

Shell 26: Observed proportion of days in remission: <full analysis set / per protocol analysis set>

| | LEO 90100 | Vehicle |
|---------------------------------|------------|------------|
| Proportion of days in remission | (n=xxx) | (n=xxx) |
| Number of subjects | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min;Max | xx.x;xx.x | xx.x;xx.x |

Shell 27: <Statistical / Sensitivity> analysis of proportion of days in remission: <full analysis set / per protocol analysis set>

| | LEO 90100 vs. vehicle |
|--------------------------------------------|-----------------------|
| Number of subjects randomised to LEO 90100 | xxx |
| Number of subjects randomised to vehicle | xxx |
| Treatment difference | xx.xx |
| 95% CI | xx.xx-xx.xx |
| p-value | 0.xxx or <0.001 |

Estimates are obtained using multiple imputation with 100 imputation and an ANOVA model with treatment group, pooled trial site, and disease severity at maintenance baseline as factors. Estimates are pooled using Rubin's rule to draw inference.



|------------------------------|-------------------|----------------|

Shell 28: Number of relapses during maintenance phase: <full analysis set / per protocol analysis set>

| | LEO 90100 | Vehicle |
|--------------------------|-------------|-------------|
| | (n=xxx) | (n=xxx) |
| PYE | XXX.X | xxx.x |
| Number of subjects | xxx | xxx |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min;Max | xx;xx | xx;xx |
| Total number of relapses | xxx | xxx |
| Rate | XX.X | XX.X |

PYE: Patient years of exposure, SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile, Rate: Number of relapses divided by patient years of exposure multiplied by 100.

Shell 29: <Statistical / Sensitivity> analysis of number of relapses during maintenance phase <(negative binomial model)>: <full analysis set / per protocol analysis set>

| | LEO 90100 vs. Vehicle |
|--------------------------------------------|-----------------------|
| Number of subjects randomised to LEO 90100 | xxx |
| Number of subjects randomised to Vehicle | xxx |
| Rate ratio | xx.xx |
| 95% CI | xx.xx-xx.xx |
| p-value | 0.xxx or <0.001 |

Estimates are obtained from a <Poisson regression model/negative binomial model> with treatment group, pooled site, and disease severity at maintenance baseline (determined by PGA) as factors, subject as random effect, and risk time as an offset.



|------------------------------|-------------------|----------------|

Shell 30: <xxx> by visit in open-label phase: open-label safety analysis set

| Visit | Open-label safety analysis set | Randomised subjects | Not randomised subjects |
|---|---|---|---|
| <xxx></xxx> | (n=xxx) | (n=xxx) | (n=xxx) |
| Visit 1 | | | |
| Number of subjects | XXX | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | XX.X;XX.X |
| Min;Max | xx.x;xx.x | xx.x;xx.x | XX.X;XX.X |
| Visit 2 | | | |
| Number of subjects | XXX | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X | XX.X;XX.X |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |



|------------------------------|-------------------|----------------|

Shell 31: <Change / Percent change> in <xxx> from start to end of open-label phase: open-label safety analysis set

| CChange / Percent change> from visit 1 to visit 2 | Open-label safety<br>analysis set<br>(n=xxx) | Randomised<br>subjects<br>(n=xxx) | Not randomised<br>subjects<br>(n=xxx) |
|---|---|---|---|
| Number of subjects | xxx | xxx | xxx |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | XX.X;XX.X |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |

Shell 32: <xxx> by visit not related to relapse: full analysis set

| Visit | LEO 90100 | Vehicle |
|--------------------|------------|------------|
| <xxx></xxx> | (n=xxx) | (n=xxx) |
| Visit 2 | | |
| Number of subjects | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | xx.x;xx.x | xx.x;xx.x |
| Visit 3 | | |
| Number of subjects | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | xx.x;xx.x | xx.x;xx.x |
| Visit 15 | | |
| Number of subjects | xxx | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | XX.X;XX.X |



|------------------------------|-------------------|----------------|

Shell 33: <xxx> by visit for start of relapse: full analysis set

| Visit interval | LEO 90100 | Vehicle |
|--------------------|------------|------------|
| <xxx></xxx> | (n=xxx) | (n=xxx) |
| Visit 2-visit 3 | | |
| Number of subjects | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| 01;03 | XX.X;XX.X | XX.X;XX.X |
| Min; Max | XX.X;XX.X | XX.X;XX.X |
| 11211, 11011 | | |
| /isit 3 | | |
| Number of subjects | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x |
| Visit 3-visit 4 | | |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | XX.X;XX.X | XX.X;XX.X |
| Min;Max | xx.x;xx.x | xx.x;xx.x |
| isit 4 | | |
| Number of subjects | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | XX.X;XX.X | xx.x;xx.x |
| Jisit 14-visit 15 | | |
| Number of subjects | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | xx.x;xx.x | XX.X;XX.X |
| otal | | |
| Number of relapses | XXX | XXX |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x; xx.x | XX.X;XX.X |
| Min;Max | XX.X;XX.X | XX.X;XX.X |



|------------------------------|-------------------|----------------|

Shell 34: <xxx> by visit for end of relapse: full analysis set

| Visit interval | LEO 90100 | Vehicle |
|--------------------|------------|------------|
| <xxx></xxx> | (n=xxx) | (n=xxx) |
| Jisit 3-visit 4 | | |
| Number of subjects | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x; xx.x | xx.x;xx.x |
| isit 4 | | |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| 01;03 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x; xx.x | xx.x;xx.x |
| isit 4-visit 5 | | |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x; xx.x | xx.x;xx.x |
| ••• | | |
| isit 15 | | |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x |
| isit 15-visit X | | |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | xx.x;xx.x | xx.x;xx.x |
| otal | | |
| Number of relapses | XXX | XXX |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x |



|------------------------------|-------------------|----------------|

Shell 35: <Change / Percent change> in <xxx> from start of relapse to end of relapse by visit for start of relapse: full analysis set

| <pre><change change="" percent=""> in <xxx></xxx></change></pre> | LEO 90100 | Vehicle |
|---|---|---|
| from start to end of relapse period | (n=xxx) | (n=xxx) |
| isit 2-visit 3 | | |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | XX.X;XX.X | XX.X;XX.X |
| Min; Max | XX.X;XX.X | XX.X;XX.X |
| HIII, Hax | AA.A, AA.A | AA.A, AA.A |
| isit 3 | | |
| Number of subjects | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | xx.x; xx.x | xx.x; xx.x |
| isit 3-visit 4 | | |
| Number of subjects | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x |
| •• | | |
| 7isit 14-visit 15 | | |
| Number of subjects | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | XX.X;XX.X | XX.X;XX.X |
| Min; Max | xx.x;xx.x | XX.X; XX.X |
| | | , |
| otal | | |
| Number of relapses | XXX | XXX |
| Number of subjects | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | XX.X;XX.X | XX.X;XX.X |



|------------------------------|-------------------|-----------------|

Shell 36: <Physician's / Subject's> global assessment of disease severity by visit in open-label phase: open-label safety analysis set

| Visit | | | |
|---|---|---|---|
| <physician's subject's=""></physician's> | Open-label safety | Randomised | Not randomised |
| Global Assessment of Disease | analysis set | subjects | subjects |
| Severity | (n=xxx) | (n=xxx) | (n=xxx) |
| <i>J</i> isit 1 | | | |
| Number of subjects | xxx | XXX | XXX |
| Clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <almost clear="" mild="" very=""></almost> | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Visit 2 | | | |
| Number of subjects | xxx | XXX | xxx |
| Clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| <almost clear="" mild="" very=""></almost> | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |



|------------------------------|-------------------|-----------------|

Shell 37: Shift table for <physician's / subject's> global assessment of disease severity from start to end of open-label phase: open-label safety analysis set

| | | | safet<br>set<br>(n=xxx | :) | | | Randomi<br>( | sed su<br>n=xxx) | bjects | | No | t rando<br>( | mised<br>n=xxx) | _ | ts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | | • | Visit | 2 | | | v | isit 2 | | | | v | isit 2 | • | |
| <pre><physician's assessment="" global="" of<="" pre="" subject's=""></physician's></pre> | > | | | | | | | | | | | | | | |
| Disease Severity | Clear | <ac th="" vm<=""><th>&gt;Mild</th><th>Mod</th><th>Sev</th><th>Clear</th><th><ac vm=""></ac></th><th>Mild</th><th>Mod</th><th>Sev</th><th>Clear</th><th><ac vm=""></ac></th><th>Mild</th><th>Mod</th><th>Sev</th></ac> | >Mild | Mod | Sev | Clear | <ac vm=""></ac> | Mild | Mod | Sev | Clear | <ac vm=""></ac> | Mild | Mod | Sev |
| Visit 1 | | | | | | | | | | | | | | | |
| Clear | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| <almost clear="" mild="" very=""></almost> | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

<ac: Almost clear/VM: Very mild>, Mod: Moderate, Sev: Severe



|------------------------------|-------------------|-----------------|

Shell 38: <Physician's / Subject's> Global Assessment of Disease Severity by visit not related to relapse: full analysis set

| <pre><physician's subject's=""> Global Assessment of Disease Severity</physician's></pre> | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|
| 7isit 2 | | |
| Number of subjects | XXX | XXX |
| Clear | xxx (xx.x%) | xxx (xx.x%) |
| <almost clear="" mild="" very=""></almost> | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| 7isit 15 | | |
| Number of subjects | XXX | XXX |
| Clear | xxx (xx.x%) | xxx (xx.x%) |
| <almost clear="" mild="" very=""></almost> | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |



|------------------------------|-------------------|-----------------|

Shell 39: <Physician's / Subject's> global assessment of disease severity by visit for start of relapse: full analysis set

| <pre><physician's subject's=""> Global Assessment</physician's></pre> | | 90100 | Vehicle | |
|---|---|---|---|---|
| of Disease Severity | (n= | =xxx) | ( | n=xxx) |
| Visit 2-visit 3 | | | | |
| Number of subjects | | xxx | | xxx |
| Clear | | (xx.x%) | xxx | (xx.x%) |
| <pre><almost clear="" mild="" very=""></almost></pre> | | (xx.x%) | | (xx.x%) |
| Mild | | (xx.x%) | | (xx.x%) |
| Moderate | | (xx.x%) | | (xx.x%) |
| Severe | | (xx.x%) | | (xx.x%) |
| Severe | AAA ( | (\DA • \D 0 ) | AAA | (AA.A0) |
| 7isit 3 | | | | |
| Number of subjects | | XXX | | XXX |
| Clear | XXX | (xx.x%) | XXX | (xx.x%) |
| <almost clear="" mild="" very=""></almost> | XXX | (xx.x%) | XXX | (xx.x%) |
| Mild | XXX | (xx.x%) | XXX | (xx.x%) |
| Moderate | XXX | (xx.x%) | XXX | (xx.x%) |
| Severe | XXX | (xx.x%) | XXX | (xx.x%) |
| /isit 3-visit 4 | | | | |
| Number of subjects | | xxx | | xxx |
| Clear | xxx | (xx.x%) | xxx | (xx.x%) |
| <pre><almost clear="" mild="" very=""></almost></pre> | | (xx.x%) | | (xx.x%) |
| Mild | | (xx.x%) | XXX | (xx.x%) |
| Moderate | | (xx.x%) | | (xx.x%) |
| Severe | | (xx.x%) | xxx | (xx.x%) |
| ••• | | , | | , |
| Visit 14-visit 15 | | | | |
| Number of subjects | | XXX | | xxx |
| Clear | | (xx.x%) | XXX | (xx.x%) |
| <pre><almost clear="" mild="" very=""></almost></pre> | | (xx.x%) | | (xx.x%) |
| Mild | | (xx.x%) | | (xx.x%) |
| Moderate | | (xx.x%) | | (xx.x%) |
| Severe | | (xx.x%) | | (xx.x%) |
| Number of relapses | | XXX | | XXX |
| Number of subjects | | xxx | | XXX |
| Clear | | (xx.x%) | xxx | (xx.x%) |
| <pre><almost clear="" mild="" very=""></almost></pre> | | (xx.x%) | | (xx.x%) |
| Mild | | (xx.x%) | | (xx.x%) |
| Moderate | | (xx.x%) | | (xx.x%) |
| Severe | | (xx.x%) | | (xx.x%) |



|------------------------------|-------------------|-----------------|

Shell 40: <Physician's / Subject's> global assessment of disease severity by visit for end of relapse: full analysis set

| <pre><physician's subject's=""> Global Assessment of Disease Severity</physician's></pre> | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|
| White O while A | | |
| Visit 3-visit 4 | | |
| Number of subjects | XXX | XXX |
| Clear | xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| <pre><almost clear="" mild="" very=""> Mild</almost></pre> | XXX (XX.X%) | xxx (xx.x%)<br>xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| 7isit 4 | | |
| Number of subjects | XXX | XXX |
| Clear | xxx (xx.x%) | |
| <pre><almost clear="" mild="" very=""></almost></pre> | xxx (xx.x <sub>5</sub> )<br>xxx (xx.x <sub>8</sub> ) | · |
| Mild | xxx (xx.x <sub>5</sub> )<br>xxx (xx.x <sub>8</sub> ) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | , , | xxx (xx.x%) |
| /isit 4-visit 5 | | |
| Number of subjects | XXX | XXX |
| Clear | xxx (xx.x%) | xxx (xx.x%) |
| <pre><almost clear="" mild="" very=""></almost></pre> | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| • • • | | |
| Visit 15 | | |
| Number of subjects | XXX | XXX |
| Clear | | xxx (xx.x%) |
| <almost clear="" mild="" very=""></almost> | xxx (xx.x%) | |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| isit 15-UNS <sup>1</sup> | | |
| Number of subjects | XXX | XXX |
| Clear | xxx (xx.x%) | xxx (xx.x%) |
| <pre><almost clear="" mild="" very=""></almost></pre> | xxx (xx.x%) | xxx (xx.x%) |
| Mild | | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Potal | | |
| Number of relapses | XXX | XXX |
| Number of subjects | XXX | XXX |
| Clear | xxx (xx.x%) | xxx (xx.x%) |
| <pre><almost clear="" mild="" very=""></almost></pre> | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |

<sup>1)</sup> Possible unscheduled visits (UNS) in the maintenance phase after visit 15.



|------------------------------|-------------------|-----------------|

Shell 41: Shift table for <physician's / subject's> global assessment of disease severity from start of relapse to end of relapse by visit for start of relapse: full analysis set

| | LEO 90100<br>(n=xxx) | | | | | Vehicle<br>(n=xxx) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Trinit for that of malana | End of relapse | | | End of relapse | | | | | | |
| Visit for start of relapse <physician's subject's=""> Global Assessment of Disease Severity</physician's> | Clear | <ac vm=""></ac> | Mild | Mod | Sev | Clear | <ac vm=""></ac> | Mild | Mod | Sev |
| Visit 2-visit 3 | | | | | | | | | | |
| Clear | xxx | xxx | XXX | XXX | xxx | xxx | XXX | XXX | xxx | xxx |
| <pre><almost clear="" mild="" very=""></almost></pre> | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | xxx | xxx | XXX | XXX | XXX | xxx |
| Moderate | xxx | XXX | XXX | XXX | xxx | xxx | XXX | XXX | xxx | xxx |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Visit 3 | | | | | | | | | | |
| Clear | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| <almost clear="" mild="" very=""></almost> | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Visit 3-visit 4 | | | | | | | | | | |
| Clear | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| <almost clear="" mild="" very=""></almost> | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| ••• | | | | | | | | | | |
| | | | | | | | | | | continu |



|------------------------------|-------------------|-----------------|

| | LEO 90100 (n=xxx) End of relapse | | | | | Vehicle<br>(n=xxx) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | End of relapse | | | | |
| Visit for start of relapse<br><physician's subject's=""> Global<br/>Assessment of Disease Severity</physician's> | Clear | <ac vm=""></ac> | Mild | Mod | Sev | Clear | <ac vm=""></ac> | Mild | Mod | Sev |
| Visit 14-visit 15 | | | | | | | | | | |
| Clear | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| <almost clear="" mild="" very=""></almost> | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| [otal | | | | | | | | | | |
| Clear | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| <almost clear="" mild="" very=""></almost> | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

<ac: Almost clear/VM: Very mild>, Mod: Moderate, Sev: Severe



|------------------------------|-------------------|-----------------|

Shell 42: WPAI:PSO by visit: full analysis set

| | | LEO 90100 | | | Vehicle | |
|---|---|---|---|---|---|---|
| | | In remission at | In relapse at | | In remission at | In relapse at |
| | Total | visit | visit | Total | visit | visit |
| Visit<br>WPAI:PSO Score | | | | | | |
| Visit 2 | | | | | | |
| Current work status | | | | | | |
| Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Absenteeism | | | | | | |
| N | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x; xx.x | xx.x; xx.x | xx.x;xx.x |
| Min;Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x; xx.x | xx.x; xx.x | xx.x;xx.x |
| Presenteeism | | | | | | |
| N | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x; xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| | | | | | | continued. |


|------------------------------|-------------------|-----------------|

| | | LEO 90100 | | | Vehicle | |
|---|---|---|---|---|---|---|
| | - | In remission at | In relapse at | - | In remission at | In relapse at |
| | Total | visit | visit | Total | visit | visit |
| Visit<br>WPAI:PSO Score | | | | | | |
| TWPI | | | | | | |
| N | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Min;Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| TAI | | | | | | |
| N | xxx | XXX | XXX | XXX | XXX | xxx |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Min;Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Visit 8 | | | | | | |
| <as above=""></as> | | | | | | |
| Visit 15 | | | | | | |
| <as above=""></as> | | | | | | |

SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile, TWPI: Total work productivity impairment, TAI: Total activity impairment.

Subjects are included in the relapse category in each treatment group if they have been on rescue medication during the past 7 days up to the visit.



|------------------------------|-------------------|-----------------|

Shell 43: WPAI:PSO by visit: open-label safety analysis set

| | Open-label safety | | |
|---|---|---|---|
| Visit | analysis set | Randomised subjects | Not randomised subjects |
| WPAI:PSO Score | (n=xxx) | (n=xxx) | (n=xxx) |
| Visit 1 | | | |
| Current work status | | | |
| Yes | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| No | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Absenteeism | | | |
| N (GE) | XXX | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X | xx.x;xx.x |
| Min;Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Presenteeism | | | |
| N | xxx | xxx | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | xx.x | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| TWPI | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | xx.x | xx.x |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Min;Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| I | | | continue |



|------------------------------|-------------------|-----------------|

| isit<br>WPAI:PSO Score | Open-label safety<br>analysis set<br>(n=xxx) | Randomised subjects (n=xxx) | Not randomised subjects (n=xxx) |
|---|---|---|---|
| TAI | | | |
| N | xxx | xxx | xxx |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x; xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| isit 2 | | | |
| <as above=""></as> | | | |

SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile, TWPI: Total work productivity impairment, TAI: Total activity impairment.



|------------------------------|-------------------|-----------------|

Shell 44: Total PSI score during open-label phase; open-label safety analysis set.

| | Open-label safety<br>analysis set | Randomised subjects | Not randomised subjects |
|---|---|---|---|
| Total PSI score (AUC) | (n=xxx) | (n=xxx) | (n=xxx) |
| Number of subjects | xxx | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Min; Max | XX.X;XX.X | xx.x;xx.x | xx.x;xx.x |

SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile, AUC: Area under the curve. AUC is calculated based on all the daily total PSI scores using the trapezoidal rule to approximate the area under and is normalised by the total number of days in the open-label phase.

Shell 45: <Change / Percent change> in total PSI score from start to end of open-label phase: open-label safety analysis set

| otal PSI score from visit 1 | Open-label safety analysis set | Randomised subjects | Not randomised subjects |
|---|---|---|---|
| to visit 2 | (n=xxx) | (n=xxx) | (n=xxx) |
| Number of subjects | xxx | xxx | xxx |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Min; Max | XX.X;XX.X | XX.X;XX.X | xx.x;xx.x |

SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile



|------------------------------|-------------------|-----------------|

Shell 46: Total PSI score for time on rescue medication and time in remission during the first 28 weeks of the maintenance phase: full analysis set

| | LEO 90100 | Vehicle |
|---------------------------|------------|------------|
| Total PSI score (AUC) | (n=xxx) | (n=xxx) |
| Time in remission | | |
| Number of subjects | XXX | xxx |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x; xx.x |
| Time in relapse | | |
| Number of subjects | XXX | xxx |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | XX.X;XX.X | XX.X;XX.X |
| Min; Max | xx.x;xx.x | xx.x;xx.x |
| Time in maintenance phase | | |
| Number of subjects | XXX | xxx |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | XX.X;XX.X | XX.X;XX.X |
| Min; Max | XX.X;XX.X | xx.x; xx.x |

SD: Standard deviation,  $Q1:1^{st}$  quartile,  $Q3: 3^{rd}$  quartile, AUC: Area under the curve.

Average PSI score is calculated as area under the curve (AUC) over the time intervals on rescue medication

and the time intervals in remission for each subject. AUC is calculated based on all the weekly total PSI scores using the trapezoidal rule to approximate the area under and is normalised by the total number of days remission or relapse, respectively.



|------------------------------|-------------------|-----------------|

## Shell 47: Statistical analysis of PSI: full analysis set

| Weeks from randomisation | LEO 90100 vs. vehicle |
|--------------------------------------------|-----------------------|
| Number of subjects wordenied to IEO 00100 | |
| Number of subjects randomised to LEO 90100 | XXX |
| Number of subjects randomised to vehicle | XXX |
| Randomisation | |
| Estimated means | |
| LEO 90100 | XX.XX |
| Vehicle | xx.xx |
| Treatment difference | xx.xx |
| 95% CI | xx.xx-xx.xx |
| p-value | 0.xxx or <0.001 |
| Week 4 | |
| Estimated means | |
| LEO 90100 | |
| Vehicle | |
| Treatment difference | |
| 95% CI | |
| p-value | |
| <u>.</u> | |
| | continued |



|------------------------------|-------------------|-----------------|

Weeks from randomisation LEO 90100 vs. vehicle

#### Week 28

Estimated means LEO 90100 Vehicle

Treatment difference 95% CI p-value

Estimates are obtained from a Mixed effect Model Repeat Measurement (MMRM) including treatment group, days from randomisation, interaction between treatment and time, relapse status, PSI total score at time of randomisation. Multiple imputation is used to impute missing assessment of PSI. Rubin's rule is used to pool the estimates for the inference.



|------------------------------|-------------------|-----------------|

### Shell 48: Statistical analysis of DLQI: full analysis set

| | LEO 90100 vs. vehicle |
|--------------------------------------------|-----------------------|
| Tumber of subjects randomised to LEO 90100 | xxx |
| umber of subjects randomised to vehicle | xxx |
| isit 2 | |
| stimated means | |
| LEO 90100 | XX.XX |
| Vehicle | xx.xx |
| reatment difference | xx.xx |
| 5% CI | xx.xx-xx.xx |
| -value | 0.xxx or <0.001 |
| isit 15 | |
| stimated means | |
| LEO 90100 | |
| Vehicle | |
| reatment difference | |
| 5% CI | |
| -value | |

Estimates are obtained from a Mixed effect Model Repeat measurement (MMRM) including treatment group, days from randomisation, interaction between treatment and time, relapse status, DLQI total score at time of randomisation. Multiple imputation is used to impute missing assessment of DLQI. Rubin's rule is used to pool the estimates for the inference.



| Trial ID: LP0053-1004 | Date: 15-JUL-2019 | Version: 1.0 |
|-----------------------|-------------------|-----------------|

Shell 49: Shift table for EQ-5D-5L from start to end of open-label phase: open-label safety analysis set

| | | Open-label safety analysis set Randomised su (n=xxx) (n=xxx) | | | | | - | ects | Not randomised subjects (n=xxx) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | | Vi | sit | 2 | | | v | isit | 2 | | | V | isit | 2 | |
| EQ-5D-5L | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 |
| /isit 1 | | | | | | | | | | | | | | | |
| Mobility | | | | | | | | | | | | | | | |
| 0: I have no problems walking | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight problems walking | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate problems walking | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems walking | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to walk | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Self-care | | | | | | | | | | | | | | | |
| 0: I have no problems washing or dressing myself | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight washing or dressing myself | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate washing or dressing myself | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe washing or dressing myself | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to wash or dress myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Usual activities | | | | | | | | | | | | | | | |
| 0: I have no problems doing my usual activities | XXX | XXX : | XXX | xxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight problems doing my usual activities | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate problems doing my usual activities | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems doing my usual activities | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to do my usual activities | XXX | XXX : | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |



|------------------------------|-------------------|-----------------|

| | - | n-lab<br>naly<br>(n= | | set | _ | Ran | | sed<br>n=xx: | _ | ects | ran | | Not<br>sed :<br>n=xx: | subj | ects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | | Vis | it | 2 | | | V | isit | 2 | | | V | isit | 2 | |
| EQ-5D-5L | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 |
| Pain/discomfort | | | | | | | | | | | | | | | |
| 0: I have no pain or discomfort | xxx | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight pain or discomfort | xxx | XXX X | XX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate pain or discomfort | xxx | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe pain or discomfort | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme pain or discomfort | XXX | XXX X | XX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Anxiety/depression | | | | | | | | | | | | | | | |
| 0: I am not anxious or depressed | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I am slightly anxious or depressed | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I am moderate problems walking | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems walking | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to walk | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Skin irritation | | | | | | | | | | | | | | | |
| 0: I have no itching | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight itching | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate itching | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe itching | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme itching | XXX | XXX X | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Self-confidence | | | | | | | | | | | | | | | |
| 0: I have no problems with self-confidence | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight problems with self-confidence | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate problems with self-confidence | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems with self-confidence | XXX | XXX X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme problems with self-confidence | XXX | XXX X | XXX X | XXX | xxx | XXX | xxx | xxx | xxx | xxx | XXX | xxx | XXX | XXX | XXX |

Column numbers refers to the numbering in each question.



|------------------------------|-------------------|-----------------|

# Shell 50: Shift table for EQ-5D-5L-PSO dimensions from start of relapse to end of relapse by visit for start of relapse: maintenance full analysis set

| | | LEO 90100<br>(n=xxx) | | | | | | Vehicle<br>(n=xxx) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | I | ind c | f re | laps | е | E | Ind c | f re | laps | e |
| isit<br>EO-5D-5L | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 |
| <u> </u> | 0 | | | | - | U | | | | - 4 |
| isit 2-visit 3 | | | | | | | | | | |
| Mobility | | | | | | | | | | |
| 0: I have no problems walking | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight problems walking | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate problems walking | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems walking | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to walk | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Self-care | | | | | | | | | | |
| 0: I have no problems washing or dressing myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight washing or dressing myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate washing or dressing myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe washing or dressing myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to wash or dress myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Usual activities | | | | | | | | | | |
| 0: I have no problems doing my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight problems doing my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate problems doing my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems doing my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to do my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | | | | | | СО | ntinu |



|------------------------------|-------------------|-----------------|

| | | | 0 90:<br>n=xx | | | | | ehic<br>n=xx | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | E | nd c | f re | laps | e | E | nd c | f re | laps | е |
| isit | | | | | | | | | | |
| EQ-5D-5L | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 |
| Pain/discomfort | | | | | | | | | | |
| 0: I have no pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Anxiety/depression | | | | | | | | | | |
| 0: I am not anxious or depressed | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I am slightly anxious or depressed | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I am moderate problems walking | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems walking | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to walk | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Skin irritation | | | | | | | | | | |
| 0: I have no itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Self-confidence | | | | | | | | | | |
| 0: I have no problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |



|------------------------------|-------------------|-----------------|

| | LEO 90100 Vehicle (n=xxx) (n=xxx) |
|-------------------------------------|----------------------------------------|
| | End of relapse |
| Visit | |
| EQ-5D-5L | 0 1 2 3 4 0 1 2 3 4 |
| Visit 3 | |
| Visit 3-visit 4 | |
| Visit 15 - UNS <sup>1</sup> | |
| •<br>• | |
| Total | |
| Mobility | |
| 0: I have no problems walking | XXX XX |
| 1: I have slight problems walking | XXX XX |
| 2: I have moderate problems walking | XXX XX |
| 3: I have severe problems walking | XXX XX |
| 4: I am unable to walk | xxx xx |



|------------------------------|-------------------|-----------------|

| | | | 0 90:<br>n=xx: | | | Vehicle (n=xxx) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | I | End c | f re | laps | e | E | Ind o | f re | laps | e |
| risit | | | | | | | | | | |
| EQ-5D-5L | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 |
| Self-care | | | | | | | | | | |
| 0: I have no problems washing or dressing myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight washing or dressing myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate washing or dressing myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe washing or dressing myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to wash or dress myself | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Usual activities | | | | | | | | | | |
| 0: I have no problems doing my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight problems doing my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate problems doing my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems doing my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to do my usual activities | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Pain/discomfort | | | | | | | | | | |
| 0: I have no pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme pain or discomfort | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Anxiety/depression | | | | | | | | | | |
| 0: I am not anxious or depressed | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I am slightly anxious or depressed | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I am moderate problems walking | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems walking | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I am unable to walk | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | | | | | | | co | ntinu |



|------------------------------|-------------------|-----------------|

| | | | 0 901<br>n=xxx | | | | | ehicl | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| | End of relapse | | | | | End of relapse | | | | |
| isit | | | | | | | | | | |
| EQ-5D-5L | 0 | 1 | 2 | 3 | 4 | 0 | 1 | 2 | 3 | 4 |
| Skin irritation | | | | | | | | | | |
| 0: I have no itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme itching | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Self-confidence | | | | | | | | | | |
| 0: I have no problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 1: I have slight problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 2: I have moderate problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3: I have severe problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4: I have extreme problems with self-confidence | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |



Column numbers refers to the numbering in each question.

1) Possible unscheduled visits (UNS) in the maintenance phase after visit 15.

|------------------------------|-------------------|-----------------|

# Shell 51: Subjects in remission by scheduled visit: full analysis set

| Visit | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|
| Visit 2 Number of subjects attending the visit Number of subjects in remission | xxx<br>xxx (xx.x%) | xxx<br>xxx (xx.x%) |
| Visit 3<br><as above=""></as> | | |
| <b>Visit 15</b> <as above=""></as> | | |



|------------------------------|-------------------|-----------------|

Shell 52: Subjects achieving clear or almost clear after treatment of relapse by number of relapses: full analysis set

| | LEO 90100 | Vehicle |
|---|---|---|
| Number of relapses | (n=xxx) | (n=xxx) |
| 1 <sup>st</sup> | | |
| Number of subjects with relapse<br>Number of subjects achieving clear or almost clear | xxx (xx.x%) | xxx (xx.x%) |
| $2^{ m nd}$ | | |
| <as above=""></as> | | |
| 3rd | | |
| <as above=""></as> | | |
| 4 <sup>th</sup><br><as above=""></as> | | |
| 5 <sup>th</sup><br><as above=""></as> | | |
| (ds dbove) | | |
| 6 <sup>th</sup> | | |
| <as above=""></as> | | |
| 7 <sup>th</sup> | | |
| <as above=""></as> | | |
| 8 <sup>th</sup> | | |
| <as above=""></as> | | |



|------------------------------|-------------------|-----------------|

Shell 53: Target lesion/location score by visit in open-label phase: open-label safety analysis set

| Farget lesion/location score<br>Visit | Ope<br>s<br>anal<br>(r | su | domised<br>bjects<br>n=xxx) | Not<br>randomised<br>subjects<br>(n=xxx) | | |
|---|---|---|---|---|---|---|
| Redness | | | | | | |
| Visit 1 | | | | | | |
| Number of subjects | | xxx | | XXX | | XXX |
| None | xxx | (xx.x%) | xxx | (xx.x%) | xxx | (xx.x%) |
| Mild | | (xx.x%) | | (xx.x%) | | , |
| Moderate | | (xx.x%) | | (xx.x%) | | . , |
| Severe | | (xx.x%) | | (xx.x%) | | , |
| Very severe | | (xx.x%) | | (xx.x%) | | . , |
| .017 00.010 | | (11111110) | | (1111 • 11 0 ) | | (1111 • 11 0 ) |
| Visit 2 | | | | | | |
| <as above=""></as> | | | | | | |
| hickness | | | | | | |
| Visit 1 | | | | | | |
| Number of subjects | | XXX | | XXX | | XXX |
| None | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Mild | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Moderate | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Severe | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Very severe | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Visit 2 | | | | | | |
| <as above=""></as> | | | | | | |
| Scaliness | | | | | | |
| Visit 1 | | | | | | |
| Number of subjects | | XXX | | XXX | | XXX |
| None | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Mild | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Moderate | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Severe | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Very severe | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (xx.x%) |
| Visit 2 | | | | | | |
| <as above=""></as> | | | | | | |



|------------------------------|-------------------|-----------------|

Shell 54: Shift table for target lesion/location score from start to end of open-label phase: open-label safety analysis set

| | | | l safe<br>set<br>(n=xxx | - | | | Randomi<br>( | sed subn=xxx) | ojects | | No | t rando | mised<br>(n=xxx | - | cts |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Visit | 2 | | | v | isit 2 | | | | 7 | /isit | 2 | |
| Visit | | | | | | | | | | | | | | | |
| Target lesion/location | | | | | | | | | | | | | | | |
| score | None | Mild | Mod | Sev | vs | None | Mild | Mod | Sev | vs | None | Mild | Mod | Sev | vs |
| Jisit 1 | | | | | | | | | | | | | | | |
| Redness | | | | | | | | | | | | | | | |
| None | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Very severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Thickness | | | | | | | | | | | | | | | |
| None | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Very severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Scaliness | | | | | | | | | | | | | | | |
| None | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Very severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Mod: Moderate, Sev: Severe, VS: Very severe



|------------------------------|-------------------|-----------------|

Shell 55: Target lesion/location score by visit not related to relapse: full analysis set

| arget lesion/location score Visit | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|
| tedness | | |
| Visit 2 | | |
| Number of subjects | XXX | XXX |
| None | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Very severe | xxx (xx.x%) | |
| Visit 15 | | |
| <as above=""></as> | | |
| hickness | | |
| Visit 2 | | |
| Number of subjects | XXX | XXX |
| None | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%) |
| Moderate | | |
| Severe | xxx (xx.x%) | |
| Very severe | xxx (xx.x%) | xxx (xx.x%) |
| Visit 15 | | |
| <as above=""></as> | | |
| caliness | | |
| Visit 2 | | |
| Number of subjects | XXX | XXX |
| None | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%) |
| Mild | XXX (XX.X%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%) |
| Severe | XXX (XX.X%) | xxx (xx.x%) |
| Very severe | xxx (xx.x%) | xxx (xx.x%) |
| ••• | | |
| Visit 15 | | |
| <as above=""></as> | | |



|------------------------------|-------------------|-----------------|

Shell 56: Target lesion/location score by visit for start of relapse: full analysis set

| edness Visit 2-visit 3 Number of subjects None Mild Moderate Severe Very severe Visit 3 <as above=""> Visit 3-visit 4</as> | xxx<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) | (n=xxx) |
|---|---|---|
| <pre>Visit 2-visit 3 Number of subjects None Mild Moderate Severe Very severe Visit 3 <as above=""></as></pre> | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) |
| Number of subjects None Mild Moderate Severe Very severe Visit 3 <as above=""></as> | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) |
| None Mild Moderate Severe Very severe Visit 3 <as above=""></as> | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) |
| None Mild Moderate Severe Very severe Visit 3 <as above=""></as> | xxx (xx.x%) | xxx (xx.x%) |
| Moderate Severe Very severe Visit 3 <as above=""></as> | xxx (xx.x%) | xxx (xx.x%) |
| Severe Very severe Visit 3 <as above=""></as> | xxx (xx.x%) | xxx (xx.x%) |
| Very severe Visit 3 <as above=""></as> | xxx (xx.x%) | xxx (xx.x%) |
| Visit 3 <as above=""></as> | xxx (xx.x%) | xxx (xx.x%) |
| <as above=""></as> | | |
| Wigit 2-wigit A | | |
| VISIC 3-VISIC 4 | | |
| <as above=""></as> | | |
| ••• | | |
| Visit 14-visit 15 | | |
| <as above=""></as> | | |
| Total | | |
| Number of relapses | XXX | XXX |
| Number of subjects | xxx | XXX |
| None | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) |
| Severe | | |
| Very severe | xxx (xx.x%) | xxx (xx.x%) |
| nickness | | |
| Visit 2-visit 3 | | |
| Number of subjects | XXX | XXX |
| None | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%)<br>xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Very severe | xxx (xx.x%) | xxx (xx.x%) |
| Visit 3 | | |
| <as above=""></as> | | |
| Visit 3-visit 4 | | |
| <as above=""></as> | | |
| ••• | | |
| Visit 14-visit 15 | | |
| <as above=""></as> | | |



|------------------------------|-------------------|-----------------|

| arget lesion/location score | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|
| Total | | |
| Number of relapses | xxx | XXX |
| Number of subjects | XXX | XXX |
| None | xxx (xx.x%) | , , |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Very severe | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%) |
| caliness | | |
| Visit 2-visit 3 | | |
| Number of subjects | XXX | XXX |
| None | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Very severe | xxx (xx.x%) | xxx (xx.x%) |
| Visit 3 | | |
| <as above=""></as> | | |
| Visit 3-visit 4 | | |
| <as above=""></as> | | |
| ••• | | |
| Visit 14-visit 15 | | |
| <as above=""></as> | | |
| Total | | |
| Number of relapses | XXX | XXX |
| Number of subjects | XXX | XXX |
| None | xxx (xx.x%) | , |
| Mild | xxx (xx.x%) | |
| Moderate | xxx (xx.x%) | |
| Severe | xxx (xx.x%) | · |
| Very severe | xxx (xx.x%) | xxx (xx.x%) |



|------------------------------|-------------------|-----------------|

Shell 57: Target lesion/location score by visit for end of relapse: full analysis set

| 'arget lesion/location score | LEO 90100 | Vehicle |
|---|---|---|
| Visit | (n=xxx) | (n=xxx) |
| ladaaa | | |
| edness<br>Visit 3-visit 4 | | |
| Number of subjects | | |
| - | XXX | XXX |
| None<br>Mild | xxx (xx.x%) | xxx (xx.x%) |
| | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Very severe | xxx (xx.x%) | xxx (xx.x%) |
| Visit 4 | | |
| <as above=""></as> | | |
| Visit 4-visit 5 | | |
| <as above=""></as> | | |
| ••• | | |
| Winit 15 | | |
| Visit 15 | | |
| <as above=""></as> | | |
| Visit 15-UNS <sup>1</sup> | | |
| <as above=""></as> | | |
| Total | | |
| Number of relapses | XXX | xxx |
| Number of subjects | XXX | xxx |
| None | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Very severe | xxx (xx.x%) | xxx (xx.x%) |
| hickness | | |
| Visit 3-visit 4 | | |
| Number of subjects | xxx | XXX |
| None | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%) |
| Very severe | xxx (xx.x%)<br>xxx (xx.x%) | xxx (xx.x%)<br>xxx (xx.x%) |
| Visit 4 | | |
| <as above=""></as> | | |
| Visit 4-visit 5 | | |
| <as above=""></as> | | |
| ••• | | |
| Visit 15 | | |
| <as above=""></as> | | |
| Visit 15-UNS <sup>1</sup> | | |
| <as above=""></as> | | |
| above/ | | contin |



| Trial ID: LP0053-1004 | Date: 15-JUL-2019 | Version: 1.0 |
|-----------------------|-------------------|-----------------|

| rget lesion/location score<br>Visit | LEO ( | Vehicle<br>(n=xxx) | | |
|---|---|---|---|---|
| Total | | | | |
| Number of relapses | X | xx | | XXX |
| Number of subjects | X | XX | | XXX |
| None | xxx ( | xx.x%) | XXX | (xx.x%) |
| Mild | xxx ( | xx.x%) | XXX | (xx.x%) |
| Moderate | xxx ( | xx.x%) | XXX | (xx.x%) |
| Severe | xxx ( | xx.x%) | XXX | (xx.x%) |
| Very severe | xxx ( | xx.x%) | XXX | (xx.x%) |
| aliness | | | | |
| Visit 3-visit 4 | | | | |
| Number of subjects | X | XX | | XXX |
| None | xxx ( | xx.x%) | XXX | (xx.x%) |
| Mild | xxx ( | xx.x%) | XXX | (xx.x%) |
| Moderate | xxx ( | xx.x%) | XXX | (xx.x%) |
| Severe | xxx ( | xx.x%) | XXX | (xx.x%) |
| Very severe | xxx ( | xx.x%) | XXX | (xx.x%) |
| Visit 4 | | | | |
| <as above=""></as> | | | | |
| Visit 4-visit 5 | | | | |
| <as above=""></as> | | | | |
| ••• | | | | |
| Visit 15 | | | | |
| <as above=""></as> | | | | |
| Visit 15-UNS <sup>1</sup> | | | | |
| <as above=""></as> | | | | |
| Total | | | | |
| Number of relapses | X | XX | | XXX |
| Number of subjects | X | XX | | XXX |
| None | xxx ( | xx.x%) | | (xx.x%) |
| Mild | xxx ( | xx.x%) | XXX | (xx.x% |
| Moderate | xxx ( | xx.x%) | XXX | (xx.x% |
| Severe | · | xx.x%) | XXX | (xx.x%) |
| Very severe | xxx ( | xx.x%) | xxx | (xx.x% |



|------------------------------|-------------------|-----------------|

Shell 58: Shift table for target lesion/location score from start of relapse to end of relapse by visit for start of relapse: full analysis set

| | | L | EO 90100<br>(n=xxx) | | | Vehicle<br>(n=xxx) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | End | of relap | se | End of relapse | | | | | |
| Target lesion/location score<br>Visit interval | None | Mild | Mod | Sev | vs | None | Mild | Mod | Sev | vs |
| Redness | | | | | | | | | | |
| Visit 2-visit 3 | | | | | | | | | | |
| None | xxx | xxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | xxx | XXX | xxx | XXX | XXX | xxx | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Very severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Visit 3 | | | | | | | | | | |
| None | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Very severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Visit 3-visit 4 | | | | | | | | | | |
| None | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Very severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| •• | | | | | | | | | | continu |



|------------------------------|-------------------|-----------------|

| | | I | EO 90100<br>(n=xxx) | | | Vehicle<br>(n=xxx) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | End | of relap | se | End of relapse | | | | | |
| arget lesion/location score | | | | | | | | | | |
| Visit interval | None | Mild | Mod | Sev | vs | None | Mild | Mod | Sev | VS |
| Visit 14-visit 15 | | | | | | | | | | |
| None | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Very severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Total | | | | | | | | | | |
| None | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | xxx |
| Very severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| ickness | | | | | | | | | | |
| <as above=""></as> | | | | | | | | | | |
| aliness | | | | | | | | | | |
| caliness<br><as above=""></as> | | | | | | | | | | |

Mod: Moderate, Sev: Severe, VS: Very severe



|------------------------------|-------------------|-----------------|--|

Shell 59: Overall summary of adverse events during open-label phase: open-label safety analysis set

| | 0 | pen-label LE<br>(n=xxx) | | |
|---|---|---|---|---|
| | N | (%) | E | R |
| PYE | XXX.XX | | | |
| Events | xxx | (xx.x) | XXX | xxx.x |
| Serious | XXX | (xx.x) | XXX | XXX.X |
| Severity | | | | |
| Mild | XXX | (xx.x) | XXX | XXX.X |
| Moderate | XXX | (xx.x) | XXX | XXX.X |
| Severe | XXX | (xx.x) | XXX | XXX.X |
| Related <sup>1</sup> to IMP | XXX | (xx.x) | XXX | XXX.X |
| Leading to withdrawal from trial | XXX | (xx.x) | XXX | XXX.X |
| Action taken with IMP | | | | |
| Dose not changed | XXX | (xx.x) | XXX | XXX.X |
| Dose reduced | XXX | (xx.x) | XXX | XXX.X |
| Dose increased | XXX | (xx.x) | XXX | XXX.X |
| Drug interrupted | XXX | (xx.x) | XXX | XXX.X |
| Drug withdrawn | XXX | (xx.x) | XXX | xxx.x |
| Not applicable | XXX | (xx.x) | XXX | XXX.X |
| Unknown | XXX | (xx.x) | XXX | xxx.x |
| Outcome | | | | |
| Fatal | XXX | (xx.x) | XXX | XXX.X |
| Not recovered/Not resolved | XXX | (xx.x) | XXX | XXX.X |
| Recovering/Resolving | XXX | (xx.x) | XXX | XXX.X |
| Recovered/Resolved | XXX | (xx.x) | XXX | XXX.X |
| Recovered/Resolved with sequelae | XXX | (xx.x) | XXX | XXX.X |
| Unknown | XXX | (xx.x) | XXX | XXX.X |

AEs collected during the exposure time in the initial open-label phase are shown. IMP: Investigational medicinal product, PYE: Patient years of exposure, N: Number of subjects with one or more events, %: Percentage of subjects with one or more events, E: Number of adverse events, R: Rate (number of adverse events divided by patient years of exposure multiplied by 100).



<sup>1)</sup> Considered possibly or probably related to trial product by the investigator.

|------------------------------|-------------------|-----------------|

Shell 60: Overall summary of adverse events during <XXX> by randomised treatment: safety analysis set

| | | LEO 9 | 0100 | | | Vehic | le | |
|---|---|---|---|---|---|---|---|---|
| | | (n=x | xx) | | | (n=xx | x) | |
| | N | (%) | E | R | N | (%) | E | R |
| PYE | xxx.xx | | | | xxx.xx | | | |
| Events | XXX | (xx.x) | XXX | XXX.X | xxx | (xx.x) | XXX | xxx.x |
| Serious | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Severity | | | | | | | | |
| Mild | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Moderate | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Severe | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Related <sup>1</sup> to IMP | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Leading to withdrawal from trial | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Action taken with IMP | | | | | | | | |
| Dose not changed | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Dose reduced | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Dose increased | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Drug interrupted | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Drug withdrawn | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Not applicable | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Unknown | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Outcome | | | | | | | | |
| Fatal | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Not recovered/Not resolved | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Recovering/Resolving | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Recovered/Resolved | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Recovered/Resolved with sequelae | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |
| Unknown | XXX | (xx.x) | XXX | XXX.X | XXX | (xx.x) | XXX | XXX.X |

AEs collected during the exposure time in the <total/first 28 weeks of the/remaining 24 weeks of the> maintenance phase are shown.

IMP: Investigational medicinal product, PYE: Patient years of exposure, N: Number of subjects with one or more events, %: Percentage of subjects with one or more events, E: Number of adverse events, R: Rate (number of adverse events divided by patient years of exposure multiplied by 100).

<sup>1)</sup> Considered possibly or probably related to IMP by the investigator.



|------------------------------|-------------------|-----------------|

Shell 61: Overall summary of adverse events during <XXX> by randomised treatment and rescue medication: safety analysis set

| | LEO 90100<br>(n= | remis | ssion | | Vehicle remission (n=xxx) | | | LEO 90100 relapse (n=xxx) | | | Vehicle relapse<br>(n=xxx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N (%) | E | R | N (%) | E | R | N (%) | E | R | N (%) | E | R |
| PYE | xxx.xx | | | xxx.xx | | | xxx.xx | | | XXX.XX | | |
| Events | xxx(xx.x) | xxx | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x |
| Serious | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Severity | | | | | | | | | | | | |
| Mild | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Moderate | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Severe | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Related <sup>1</sup> to IMP | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Leading to withdrawal from trial | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x |
| Action taken with IMP | | | | | | | | | | | | |
| Dose not changed | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Drug withdrawn | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Not applicable | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Unknown | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x |
| Outcome | | | | | | | | | | | | |
| Fatal | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x |
| Not recovered/Not resolved | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x |
| Recovering/Resolving | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x |
| | | | | | | | | | | | conti | inued |



|------------------------------|-------------------|-----------------|

| | LEO 90100 remission (n=xxx) | | | | Vehicle remission (n=xxx) | | | LEO 90100 relapse (n=xxx) | | | Vehicle relapse<br>(n=xxx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N (%) | E | R | N (%) | E | R | N (%) | E | R | N (%) | E | R |
| Recovered/Resolved | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | xxx | xxx.x | xxx(xx.x) | xxx | xxx.x |
| Recovered/Resolved with sequelae | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | xxx | xxx.x | xxx(xx.x) | XXX | xxx.x |
| Unknown | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | xxx | xxx.x |

AEs collected during the exposure time in the <total/first 28 weeks of the/remaining 24 weeks of the> maintenance phase are shown.

IMP: Investigational medicinal product, PYE: Patient years of exposure, N: Number of subjects with one or more events, %: Percentage of subjects with one or more events, E: Number of adverse events, R: Rate (number of adverse events divided by patient years of exposure multiplied by 100).

1) Considered possibly or probably related to IMP by the investigator.



|------------------------------|-------------------|-----------------|

Shell 62: <XXX> during the open-label phase by SOC and preferred term: open-label safety analysis set

| System Organ Class (SOC) | Open-label LEO 90100<br>(n=xxx) | | | |
|---|---|---|---|---|
| Preferred term | N | (%) | E | R |
| PYE | xxx.x | | | |
| All AEs | xxx | (xx.x) | XXX | XXX.XX |
| SOC 1 | xxx | (xx.x) | XXX | xxx.xx |
| Preferred term 1 | XXX | (xx.x) | XXX | xxx.xx |
| • • • | XXX | (xx.x) | XXX | XXX.XX |
| Preferred term $k_1$ | XXX | (xx.x) | XXX | XXX.XX |
| SOC 2 | xxx | (xx.x) | XXX | xxx.xx |
| Preferred term 1 | XXX | (xx.x) | XXX | XXX.XX |
| ••• | XXX | (xx.x) | XXX | XXX.XX |
| Preferred term $k_2$ | XXX | (xx.x) | XXX | XXX.XX |
| SOC M | XXX | (xx.x) | XXX | XXX.XX |
| Preferred term 1 | XXX | (xx.x) | XXX | XXX.XX |
| | XXX | (xx.x) | XXX | XXX.XX |
| Preferred term $k_{\mathtt{M}}$ | XXX | (xx.x) | XXX | XXX.XX |

AEs collected during the exposure time in the initial open-label phase are shown. Classification according to MedDRA xx.x. N: Number of subjects with one or more events, %: Percentage of subjects with one or more events, E: Number of adverse events, R: Rate (number of adverse events divided by patient years of exposure multiplied by 100).



|------------------------------|-------------------|-----------------|

Shell 63: <XXX> during <XXX> by SOC, preferred term, and randomised treatment: safety analysis set

| System Organ Class (SOC)<br>Preferred term | | | 90100<br>=xxx) | Vehicle<br>(n=xxx) | | | | |
|---|---|---|---|---|---|---|---|---|
| | N | (%) | E | R | N | (%) | E | R |
| PYE | xxx.x | | | | xxx.x | | | |
| All AEs | XXX | (xx.x) | XXX | xxx.xx | xxx | (xx.x) | XXX | XXX.XX |
| SOC 1 | xxx | (xx.x) | xxx | xxx.xx | XXX | (xx.x) | xxx | xxx.xx |
| Preferred term 1 | XXX | (xx.x) | XXX | XXX.XX | XXX | (xx.x) | XXX | XXX.XX |
| • • • | XXX | (xx.x) | XXX | XXX.XX | XXX | (xx.x) | XXX | XXX.XX |
| Preferred term $k_1$ | XXX | (xx.x) | XXX | xxx.xx | xxx | (xx.x) | XXX | XXX.XX |
| SOC 2 | XXX | (xx.x) | xxx | xxx.xx | xxx | (xx.x) | XXX | xxx.xx |
| Preferred term 1 | XXX | (xx.x) | XXX | XXX.XX | XXX | (xx.x) | XXX | XXX.XX |
| ••• | XXX | (xx.x) | XXX | XXX.XX | XXX | (xx.x) | XXX | xxx.xx |
| Preferred term $k_2$ | XXX | (xx.x) | XXX | xxx.xx | XXX | (xx.x) | XXX | XXX.XX |
| SOC M | xxx | (xx.x) | XXX | xxx.xx | xxx | (xx.x) | XXX | XXX.XX |
| Preferred term 1 | XXX | (xx.x) | XXX | XXX.XX | XXX | (xx.x) | XXX | XXX.XX |
| • • • | XXX | (xx.x) | XXX | XXX.XX | XXX | (xx.x) | XXX | XXX.XX |
| Preferred term $k_{\mathtt{M}}$ | XXX | (xx.x) | XXX | XXX.XX | XXX | (xx.x) | XXX | XXX.XX |

AEs collected during the exposure time in the <total/first 28 weeks of the/remaining 24 weeks of the> maintenance phase are shown. Classification according to MedDRA xx.x.



N: Number of subjects with one or more events, %: Percentage of subjects with one or more events, E: Number of adverse events, R: Rate (number of adverse events divided by patient years of exposure multiplied by 100).

|------------------------------|-------------------|-----------------|

Shell 64: <XXX> during <XXX> by SOC, preferred term, randomised treatment, and rescue medication: safety analysis set

| System Organ Class (SOC)<br>Preferred term | LEO 90100 remission (n=xxx) | | | | Vehicle remission (n=xxx) | | | LEO 90100 relapse<br>(n=xxx) | | | Vehicle relapse<br>(n=xxx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N (%) | E | R | N (%) | Е | R | N (%) | E | R | N (%) | E | R |
| PYE | XXX.X | | | XXX.X | | | XXX.X | | | XXX.X | | |
| All AEs | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |
| soc 1 | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X |
| Preferred term 1 | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X |
| | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |
| Preferred term $k_1$ | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |
| SOC 2 | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X |
| Preferred term 1 | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |
| | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |
| Preferred term $k_2$ | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |
| SOC M | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X |
| Preferred term 1 | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |
| | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |
| Preferred term $k_{	exttt{M}}$ | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | xxx.x | xxx(xx.x) | XXX | XXX.X | xxx(xx.x) | XXX | XXX.X |

AEs collected during the exposure time in the <total/first 28 weeks of the/remaining 24 weeks of the> maintenance phase are shown. Classification according to MedDRA xx.x. N: Number of subjects with one or more events, %: Percentage of subjects with one or more events, E: Number of adverse events, R: Rate (number of adverse events divided by patient years of exposure multiplied by 100).



|------------------------------|-------------------|-----------------|

Shell 65: Adverse events during the open-label phase by causal relationship to IMP, SOC, and preferred term: open-label safety analysis set

| | Open-label LEO 90100<br>(n=xxx) | | |
|---|---|---|---|
| System Organ Class (SOC) | NR | PO | PR |
| Preferred term | E | E | E |
| PYE | xxx.x | | |
| All AEs | XXX | XXX | XXX |
| SOC 1 | XXX | xxx | xxx |
| Preferred term 1 | xxx | XXX | XXX |
| ••• | xxx | XXX | XXX |
| Preferred term $k_1$ | XXX | XXX | XXX |
| ••• | | | |
| SOC M | xxx | xxx | xxx |
| Preferred term 1 | xxx | XXX | XXX |
| | XXX | XXX | XXX |
| Preferred term $k_{\mathtt{M}}$ | XXX | XXX | XXX |

AEs collected during the exposure time in the initial open-label phase are shown. Classification according to MedDRA xx.x. E: Number of adverse events, NR: Not Related, PO: Possibly Related, PR: Probably Related.



|------------------------------|-------------------|-----------------|

Shell 66: Adverse events during <XXX> by causal relationship to IMP, SOC, preferred term, and randomised treatment: safety analysis set

| | | LEO 90100<br>(n=xxx) | | Vehicle<br>(n=xxx) | | |
|---|---|---|---|---|---|---|
| System Organ Class (SOC) | NR | PO | PR | NR | PO | PR |
| Preferred term | E | E | E | E | E | E |
| PYE | xxx.x | | | xxx.x | | |
| All AEs | xxx | XXX | XXX | XXX | XXX | xxx |
| SOC 1 | XXX | xxx | XXX | xxx | xxx | xxx |
| Preferred term 1 | XXX | XXX | XXX | XXX | XXX | XXX |
| | XXX | XXX | XXX | XXX | XXX | XXX |
| Preferred term $k_1$ | xxx | XXX | XXX | xxx | xxx | xxx |
| SOC M | xxx | XXX | xxx | xxx | xxx | XXX |
| Preferred term 1 | XXX | XXX | XXX | XXX | XXX | XXX |
| | XXX | XXX | XXX | XXX | XXX | XXX |
| Preferred term $k_{\mathtt{M}}$ | XXX | XXX | xxx | xxx | XXX | XXX |

AEs collected during the exposure time in the <total/first 28 weeks of the/remaining 24 weeks of the> maintenance phase are shown. Classification according to MedDRA xx.x. E: Number of adverse events, NR: Not Related, PO: Possibly Related, PR: Probably Related.



|------------------------------|-------------------|-----------------|

Shell 67: Adverse events during <XXX> by causal relationship to IMP, SOC, preferred term, randomised treatment, and rescue medication: safety analysis set

| | LEO 90100 remission (n=xxx) | | | Vehi | Vehicle remission (n=xxx) | | | LEO 90100 relapse<br>(n=xxx) | | | Vehicle relapse (n=xxx) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class (SOC) | NR | PO | PR | NR | PO | PR | NR | PO | PR | NR | PO | PR |
| Preferred term | E | E | E | E | E | E | E | E | E | E | E | E |
| PYE | xxx.x | | | xxx.x | | | xxx.x | | | XXX.X | | |
| All AEs | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| SOC 1 | XXX | XXX | xxx | XXX | XXX | XXX | XXX | xxx | xxx | XXX | XXX | xxx |
| Preferred term 1 | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX | XXX |
| | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Preferred term $k_1$ | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| SOC M | xxx | xxx | xxx | xxx | xxx | xxx | xxx | XXX | xxx | XXX | XXX | XXX |
| Preferred term 1 | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Preferred term $k_{\mathtt{M}}$ | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

AEs collected during the exposure time in the <total/first 28 weeks of the/remaining 24 weeks of the> maintenance phase are shown. Classification according to MedDRA xx.x. E: Number of adverse events, NR: Not Related, PO: Possibly Related, PR: Probably Related.


| Trial I | D: <b>LP0053-1004</b> | Date: 15-JUL-2019 | Version: 1.0 |
|---------|-----------------------|-------------------|-----------------|

Shell 68: Physician's assessment of local safety and tolerability by visit in open-label phase: open-label safety analysis set

| Physician's assessment of local safety and<br>tolerability<br>Visit | Open-label safety analysis set (n=xxx) | Randomised subjects (n=xxx) | Not<br>randomise<br>subjects<br>(n=xxx) |
|---|---|---|---|
| Perilesional erythema | | | |
| Visit 1 | | | |
| Number of subjects | XXX | XXX | XXX |
| Absent | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Visit 2 <as above=""></as> | | | |
| Perilesional oedema | | | |
| <as above=""></as> | | | |
| Perilesional dryness | | | |
| <as above=""></as> | | | |
| Perilesional erosion | | | |
| <as above=""></as> | | | |



|------------------------------|-------------------|-----------------|

Shell 69: Shift table for physician's assessment of local safety and tolerability from start to end of open-label phase: open-label safety analysis set

| | | bjects<br>fety ana<br>(n=x | alysis s | | Rai | ndomised<br>(n=x | _ | s | Not ra | ndomise<br>(n=xx | _ | ects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Physician's assessment of local safety and | Visit 2 | | | Visit 2 | | | | Visit 2 | | | | |
| tolerability | Absent | Mild | Mod | Sev | Absent | Mild | Mod | Sev | Absent | Mild | Mod | Sev |
| Visit 1 | | | | | | | | | | | | |
| Perilesional erythema | | | | | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Perilesional oedema | | | | | | | | | | | | |
| <as above=""></as> | | | | | | | | | | | | |
| Perilesional dryness | | | | | | | | | | | | |
| <as above=""></as> | | | | | | | | | | | | |
| Perilesional erosion | | | | | | | | | | | | |
| <as above=""></as> | | | | | | | | | | | | |



|------------------------------|-------------------|-----------------|

# Shell 70: Physician's assessment of local safety and tolerability by visit not related to relapse: safety analysis set

| tolerability | LEO 90100 | Vehicle |
|-----------------------|-------------|-------------|
| Visit | (n=xxx) | (n=xxx) |
| Perilesional erytnema | | |
| Visit 2 | | |
| Number of subjects | xxx | XXX |
| Absent | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| ••• | | |
| Visit 15 | | |
| <as above=""></as> | | |
| Perilesional oedema | | |
| <as above=""></as> | | |
| Perilesional dryness | | |
| <as above=""></as> | | |
| Perilesional erosion | | |
| <as above=""></as> | | |



| Tı | rial ID: <b>LP0053-1004</b> | Date: 15-JUL-2019 | Version: 1.0 |
|----|-----------------------------|-------------------|-----------------|

Shell 71: Physician's assessment of local safety and tolerability by visit for start of relapse: safety analysis set

| colerability | LEO 90100 | Vehicle |
|-----------------------|-------------|-------------|
| Visit | (n=xxx) | (n=xxx) |
| Perilesional erythema | | |
| Visit 2-visit 3 | | |
| Number of subjects | XXX | XXX |
| Absent | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Visit 3 | | |
| <as above=""></as> | | |
| Visit 3-visit 4 | | |
| <as above=""></as> | | |
| ••• | | |
| Visit 14-visit 15 | | |
| <as above=""></as> | | |
| Total | | |
| Number of relapses | XXX | XXX |
| Number of subjects | XXX | XXX |
| Absent | xxx (xx.x%) | |
| Mild | xxx (xx.x%) | |
| Moderate | xxx (xx.x%) | |
| Severe | xxx (xx.x%) | xxx (xx.x%) |
| Perilesional oedema | | |
| <as above=""></as> | | |
| Perilesional dryness | | |
| <as above=""></as> | | |
| Perilesional erosion | | |
| <as above=""></as> | | |



|------------------------------|-------------------|-----------------|

Shell 72: Physician's assessment of local safety and tolerability by visit for end of relapse: safety analysis set

| tolerability | LEO 9010 | 0 Vehicle |
|---------------------------|------------------------|----------------|
| Visit | (n=xxx) | (n=xxx) |
| Perilesional erythema | | |
| Visit 3-visit 4 | | |
| Number of subjects | XXX | XXX |
| Absent | xxx (xx.x | |
| Mild | xxx (xx.x | %) xxx (xx.x%) |
| Moderate | xxx (xx.x<br>xxx (xx.x | %) xxx (xx.x%) |
| Severe | xxx (xx.x | %) xxx (xx.x%) |
| Visit 4 | | |
| <as above=""></as> | | |
| Visit 4-visit 5 | | |
| <as above=""></as> | | |
| ••• | | |
| Visit 15 | | |
| <as above=""></as> | | |
| Visit 15-UNS <sup>1</sup> | | |
| <as above=""></as> | | |
| Total | | |
| Number of relapses | XXX | XXX |
| Number of subjects | XXX | XXX |
| Absent | xxx (xx.x | %) xxx (xx.x%) |
| Mild | xxx (xx.x<br>xxx (xx.x | %) xxx (xx.x%) |
| Moderate | | |
| Severe | xxx (xx.x | %) xxx (xx.x%) |
| Perilesional oedema | | |
| <as above=""></as> | | |
| Perilesional dryness | | |
| <as above=""></as> | | |
| Perilesional erosion | | |
| <as above=""></as> | | |

<sup>1)</sup> Possible unscheduled visits (UNS) after Visit 15 in the maintenance phase.



|------------------------------|-------------------|-----------------|

Shell 73: Shift table for physician's assessment of local safety and tolerability from start of relapse to end of relapse by visit for start of relapse: safety analysis set

| | LEO 90100<br>(n=xxx) | | | Vehicle (n=xxx) End of relapse | | | | |
|---|---|---|---|---|---|---|---|---|
| hysician's assessment of local | End of relapse | | | | | | | |
| afety and tolerability<br>Visit | Absent | Mild | Mod | Sev | Absent | Mild | Mod | Sev |
| erilesional erythema<br>Visit 2-visit 3 | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Visit 3 | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX |
| Visit 3-visit 4 | | | | | | | | |
| Absent | XXX | xxx | XXX | XXX | XXX | XXX | xxx | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| •• | | | | | | | | continu |



|------------------------------|-------------------|-----------------|

| | | LEO 9<br>(n=x | | | | Vehic<br>(n=xx | _ | |
|---|---|---|---|---|---|---|---|---|
| | | End of | relapse | | | End of r | elapse | |
| Physician's assessment of local safety and tolerability | | | | | | | | |
| Visit | Absent | Mild | Mod | Sev | Absent | Mild | Mod | Sev |
| Visit 14-visit 15 | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX |
| Total | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Perilesional oedema | | | | | | | | |
| <as above=""></as> | | | | | | | | |
| Perilesional dryness | | | | | | | | |
| <as above=""></as> | | | | | | | | |
| Perilesional erosion <as above=""></as> | | | | | | | | |



|------------------------------|-------------------|-----------------|

Shell 74: Subject's assessment of local safety and tolerability by visit in open-label phase: open-label safety analysis set

| Subject's assessment of local safety and<br>tolerability<br>Visit | All subjects in open-label safety analysis set (n=xxx) | Randomised<br>subjects<br>(n=xxx) | Not<br>randomised<br>subjects<br>(n=xxx) |
|---|---|---|---|
| Application site burning or pain | | | |
| Visit 1 | | | |
| Number of subjects | XXX | XXX | XXX |
| Absent | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Visit 2 | | | |



|------------------------------|-------------------|-----------------|

Shell 75: Shift table for subject's assessment of local safety and tolerability from start to end of open-label phase: open-label safety analysis set

| <i>J</i> isit | open-lab | - | | | Ra | ndomised<br>(n=x: | - | .s | Not ra | ndomise<br>(n=xx | - | ects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject's assessment of | | Visi | .t 2 | | | Visi | t 2 | | | Visit | 2 | |
| local safety and<br>tolerability | Absent | Mild | Mod | Sev | Absent | Mild | Mod | Sev | Absent | Mild | Mod | Sev |
| isit 1 Application site burning | _ | | | | | | | | | | | |
| or pain | J | | | | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX | xxx | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | xxx | xxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |



|------------------------------|-------------------|-----------------|

Shell 76: Subject's assessment of local safety and tolerability by visit not related to relapse: safety analysis set

| Subject's assessment of local safety and tolerability Visit | | 90100<br>n=xxx) | Vehicle<br>(n=xxx) | |
|---|---|---|---|---|
| pplication site burning or pain | | | | |
| Visit 2 | | | | |
| Number of subjects | | XXX | | XXX |
| Absent | XXX | (xx.x%) | XXX | (xx.x%) |
| Mild | XXX | (xx.x%) | XXX | (xx.x%) |
| Moderate | XXX | (xx.x%) | XXX | (xx.x%) |
| Severe | XXX | (xx.x%) | XXX | (xx.x%) |
| Visit 15 | | | | |
| <as above=""></as> | | | | |



|------------------------------|-------------------|-----------------|

Shell 77: Subject's assessment of local safety and tolerability by visit for start of relapse: safety analysis set

| lerability | LEO 90100 | Vehicle |
|---------------------------------|------------|---------------|
| Visit | (n=xxx) | (n=xxx) |
| pplication site burning or pain | | |
| Visit 2-visit 3 | | |
| Number of subjects | XXX | XXX |
| Absent | xxx (xx.x% | |
| Mild | xxx (xx.x% | |
| Moderate | xxx (xx.x% | |
| Severe | xxx (xx.x% | |
| Visit 3 | | |
| <as above=""></as> | | |
| Visit 3-4 | | |
| <as above=""></as> | | |
| Visit 4 | | |
| <as above=""></as> | | |
| ••• | | |
| Visit 14-visit 15 | | |
| <as above=""></as> | | |
| Total | | |
| Number of relapses | XXX | XXX |
| Number of subjects | XXX | XXX |
| Absent | xxx (xx.x% | ) xxx (xx.x%) |
| Mild | xxx (xx.x% | ) xxx (xx.x%) |
| Moderate | xxx (xx.x% | ) xxx (xx.x%) |
| Severe | xxx (xx.x% | ) xxx (xx.x%) |



|------------------------------|-------------------|-----------------|

Shell 78: Subject's assessment of local safety and tolerability by visit for end of relapse: safety analysis set

| lerability | LEC | 90100 | 7 | <i>T</i> ehicle |
|---------------------------------|-----|---------|-----|-----------------|
| Visit | (r | n=xxx) | ( | (n=xxx) |
| oplication site burning or pain | | | | |
| Visit 3-visit 4 | | | | |
| Number of subjects | | XXX | | XXX |
| Absent | XXX | (xx.x%) | XXX | (xx.x%) |
| Mild | XXX | (xx.x%) | | (xx.x%) |
| Moderate | XXX | (xx.x%) | XXX | (xx.x%) |
| Severe | XXX | (xx.x%) | XXX | (xx.x%) |
| Visit 4 | | | | |
| <as above=""></as> | | | | |
| Visit 4-5 | | | | |
| <as above=""></as> | | | | |
| ••• | | | | |
| Visit 15 | | | | |
| <as above=""></as> | | | | |
| Visit 15-UNS <sup>1</sup> | | | | |
| <as above=""></as> | | | | |
| Total | | | | |
| Number of relapses | | xxx | | XXX |
| Number of subjects | | XXX | | XXX |
| Absent | XXX | (xx.x%) | XXX | (xx.x%) |
| Mild | | (xx.x%) | | (xx.x%) |
| Moderate | XXX | (xx.x%) | XXX | (xx.x%) |
| Severe | XXX | (xx.x%) | XXX | (xx.x%) |

<sup>1)</sup> Possible unscheduled visits (UNS) after visit 15 in the maintenance phase.



|------------------------------|-------------------|-----------------|

Shell 79; Shift table for subject's assessment of local safety and tolerability from start of relapse to end of relapse by visit for start of relapse: safety analysis set

| | | LEO 9<br>(n=x | | | | Vehic<br>(n=xx | | |
|---|---|---|---|---|---|---|---|---|
| Subject's assessment of local safety and tolerability | | End of 1 | relapse | | | End of r | elapse | |
| Visit | Absent | Mild | Mod | Sev | Absent | Mild | Mod | Sev |
| Application site burning or pain<br>Visit 2-visit 3 | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX |
| Visit 3 | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX |
| Visit 3-visit 4 | | | | | | | | |
| Absent | | | | | | | | |
| Mild | | | | | | | | |
| Moderate | | | | | | | | |
| Severe | | | | | | | | |
| • • • | | | | | | | | |
| Visit 14-visit 15 | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | xxx | xxx |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | xxx | xxx |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | xxx | xxx |
| | | | | | | | | continued |



|------------------------------|-------------------|-----------------|

| _ | | LEO 9<br>(n=x | | | | Vehic<br>(n=xx | _ | |
|---|---|---|---|---|---|---|---|---|
| Subject's assessment of local safety and tolerability | | End of 1 | elapse | | | End of re | elapse | |
| Visit | Absent | Mild | Mod | Sev | Absent | Mild | Mod | Sev |
| Total | | | | | | | | |
| Absent | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mild | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Moderate | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Severe | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |



|------------------------------|-------------------|-----------------|

Shell 80: Change in vital signs from baseline to end of open-label phase: open-label safety analysis set

| Vital sign | Open-label LEO 90100 |
|------------------------------|----------------------|
| Change | (n=xxx) |
| Parameter 1 ( <unit>)</unit> | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | XX.X;XX.X |
| Min; Max | xx.x; xx.x |
| Parameter 2 ( <unit>)</unit> | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min; Max | xx.x;xx.x |
| ••• | |
| Parameter k ( <unit>)</unit> | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | XX.X;XX.X |
| Min;Max | XX.X;XX.X |



|------------------------------|-------------------|-----------------|

Shell 81: Change in vital signs from randomisation to end of maintenance phase <for subjects XXX>: safety analysis set

| Vital sign | LEO 90100 | Vehicle |
|----------------------------------------------|------------|------------|
| Change | (n=xxx) | (n=xxx) |
| <parameter 1=""> (<unit>)</unit></parameter> | | |
| Number of subjects | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x; xx.x |
| Min; Max | xx.x;xx.x | xx.x; xx.x |
| <parameter 2=""> (<unit>)</unit></parameter> | | |
| Number of subjects | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x; xx.x | xx.x; xx.x |
| ••• | | |
| <parameter k=""> (<unit>)</unit></parameter> | | |
| Number of subjects | XXX | xxx |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min;Max | xx.x;xx.x | xx.x;xx.x |



|------------------------------|-------------------|-----------------|

Shell 82: Change in laboratory parameters from baseline to end of open-label phase: open-label safety analysis set

| Laboratory parameter | Open-label LEO 90100 |
|----------------------------------------------|----------------------|
| Change | (n=xxx) |
| ochemistry | |
| <parameter 1=""> (<unit>)</unit></parameter> | |
| Number of subjects | XXX |
| Mean (SD) | x.xx(x.xx) |
| Median | X.XX |
| Q1;Q3 | x.xx;x.xx |
| Min; Max | x.xx;x.xx |
| <parameter 2=""> (<unit>)</unit></parameter> | |
| Number of subjects | XXX |
| Mean(SD) | x.xx(x.xx) |
| Median | X.XX |
| Q1;Q3 | x.xx;x.xx |
| Min; Max | x.xx;x.xx |
| rinalysis | |
| <parameter 1=""> (<unit>)</unit></parameter> | |
| Number of subjects | XXX |
| Mean (SD) | x.xx(x.xx) |
| Median | X.XX |
| Q1;Q3 | x.xx;x.xx |
| Min;Max | x.xx;x.xx |
| <parameter 2=""> (<unit>)</unit></parameter> | |
| Number of subjects | XXX |
| Mean(SD) | x.xx(x.xx) |
| Median | X • XX |
| Q1;Q3 | X.XX; X.XX |
| Min; Max | x.xx;x.xx |



|------------------------------|-------------------|-----------------|

Shell 83: Change in laboratory parameters from randomisation to end of maintenance phase <for subjects XXX>: safety analysis set

| aboratory parameter | LEO 90100 | Vehicle |
|-------------------------------|------------|------------|
| Change | (n=xxx) | (n=xxx) |
| chemistry | | |
| Parameter 1> ( <unit>)</unit> | | |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| 01;03 | XX.X;XX.X | XX.X;XX.X |
| Min; Max | XX.X; XX.X | XX.X; XX.X |
| rilli, ridx | ΛΛ.Λ, ΛΛ.Λ | AA.A/ AA.A |
| Parameter 2> ( <unit>)</unit> | | |
| Number of subjects | xxx | xxx |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x; xx.x | XX.X;XX.X |
| nalysis | | |
| Parameter 1> ( <unit>)</unit> | | |
| Number of subjects | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | xx.x |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x |
| Parameter 2> ( <unit>)</unit> | | |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| 01;03 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | | |
| Min; Max | xx.x; xx.x | xx.x; xx. |



|------------------------------|-------------------|-----------------|

Shell 84: Shift table for laboratory parameter categories at baseline against end of open-label phase: open-label safety analysis set

| | | | Open-label<br>(n=x | | |
|---|---|---|---|---|---|
| | | | End of open- | label phase | |
| aboratory as | | | | | |
| Laboratory | parameter | Low | Normal | High | Missing |
| siochemistry | | | | | |
| <parameter< td=""><td>1&gt;</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td></parameter<> | 1> | XX | XX | XX | XX |
| Baseline | Low | XX | XX | XX | XX |
| Baseline | Normal | XX | XX | XX | XX |
| Baseline | High | XX | XX | XX | XX |
| Baseline | Missing | | | | |
| <parameter< td=""><td>2&gt;</td><td></td><td></td><td></td><td></td></parameter<> | 2> | | | | |
| • • • | | | | | |
| <b>Trinalysis</b> | | | | | |
| <parameter< td=""><td>1&gt;</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td></parameter<> | 1> | XX | XX | XX | XX |
| Baseline | Low | XX | XX | XX | XX |
| Baseline | Normal | XX | XX | XX | XX |
| Baseline | High | XX | XX | XX | XX |
| Baseline | Missing | | | | |
| <parameter< td=""><td>2&gt;</td><td></td><td></td><td></td><td></td></parameter<> | 2> | | | | |



|------------------------------|-------------------|-----------------|

Shell 85: Shift table for laboratory parameter categories at randomisation against end of maintenance phase <for subjects XXX>: safety analysis set

| | LEO 90100<br>(n=xxx) | | | Vehicle<br>(n=xxx) | | | | |
|---|---|---|---|---|---|---|---|---|
| | End | of maint | enance | phase | End of maintenance phase | | | |
| Laboratory assessment | | | | | | | | |
| Laboratory parameter | Low | Normal | High | Missing | Low | Normal | High | Missing |
| Biochemistry | | | | | | | | |
| <parameter 1=""></parameter> | | | | | | | | |
| Randomisation Low | XX | XX | XX | XX | XX | XX | XX | XX |
| Randomisation Normal | XX | XX | XX | XX | XX | XX | XX | XX |
| Randomisation High | XX | XX | XX | XX | XX | XX | XX | XX |
| Randomisation Missing | XX | XX | XX | XX | XX | XX | XX | XX |
| <parameter 2=""></parameter> | | | | | | | | |
| • • • | | | | | | | | |
| rinalysis | | | | | | | | |
| <parameter 1=""></parameter> | | | | | | | | |
| Randomisation Low | XX | XX | XX | XX | XX | XX | XX | XX |
| Randomisation Normal | XX | XX | XX | XX | XX | XX | XX | XX |
| Randomisation High | XX | XX | XX | XX | XX | XX | XX | XX |
| Randomisation Missing | XX | XX | XX | XX | XX | XX | XX | XX |
| <parameter 2=""></parameter> | | | | | | | | |

Shell 86: Compliance with treatment instructions during open-label treatment phase: open-label safety analysis

| | Open-label LEO 90100<br>(n=xxx) |
|---|---|
| Number of subjects in non-compliance with treatment | xxx(xx.x) |
| instructions<br>Number of daily IMP applications missed | xxx(xx.x) |
| Percentage of missed daily IMP applications: | *** (****) |
| >0% and <=10% | xx(xx.x) |
| >10% and <=20% | xx(xx.x) |
| >20% and <=30% | xx(xx.x) |
| >30% | xx(xx.x) |



|------------------------------|-------------------|-----------------|

Shell 87: Compliance with treatment instructions during maintenance phase excluding periods of treatment with rescue medication: maintenance phase safety analysis set

| xxx (n=xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | x.x) (.x) (.x) (.x) (.x) |
|---|---|
| x) | <.x) <.x) <.x) |
| x) | <.x) <.x) <.x) |
| x) | x.x)<br>x.x) |
| x) | x.x)<br>x.x) |
| x) | x.x)<br>x.x) |
| x) | x.x)<br>x.x) |
| x) xx(xx | x.x) |
| | • |
| x) xx (xx | (.x) |
| x xx | Х |
| x.x) | x.x) |
| x xx | Х |
| x.x) | x.x) |
| , | |

Shell 88: Compliance with treatment instructions during periods of treatment with rescue medication: maintenance phase safety analysis set

| | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|
| o of daily IMP applications missed ercentage of missed daily IMP pplications: | xx (xx.x) | xx(xx.x) |
| >0% and <=10% | xx(xx.x) | xx(xx.x) |
| >10% and <=20% | xx(xx.x) | xx(xx.x) |
| >20% and <=30% | xx(xx.x) | xx(xx.x) |
| >30% | xx(xx.x) | xx(xx.x) |



|------------------------------|-------------------|-----------------|

### Shell 89: Duration of exposure during the open-label treatment phase: open-label safety analysis set

| | Open-label LEO 90100<br>(n=xxx) |
|--------------------|---------------------------------|
| ration of exposure | |
| Number of days | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min; Max | xx.x;xx.x |

SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile.

#### Shell 90: Duration of exposure during the maintenance phase: safety analysis set

| | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|--------------------|----------------------|--------------------|
| ration of exposure | | |
| Number of days | xxx | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx.x | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | XX.X;XX.X | xx.x;xx.x |

SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile.

#### Shell 91: Amount of investigational medicinal product used during open-label treatment phase: open-label safety analysis set

| | Open-label LEO 90100<br>(n=xxx) |
|--------------------|---------------------------------|
| Amount of IMP used | |
| Number of subjects | xxx |
| Mean(SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min;Max | XX.X;XX.X |

SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile.

The amount of IMP used is normalised by the number of days in the open-label phase for each



|------------------------------|-------------------|-----------------|



|------------------------------|-------------------|-----------------|

Shell 92: Amount of investigational medicinal product used during maintenance phase: safety analysis set

| | | 90100<br>xxx) | _ | icle<br>xxx) |
|--------------------|------------|---------------|------------|--------------|
| | Total IMP | Rescue IMP | Total IMP | Rescue IMP |
| Number of subjects | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Q1 <b>;</b> Q3 | XX.X;XX.X | XX.X;XX.X | XX.X;XX.X | xx.x;xx.x |
| Min;Max | xx.x;xx.x | XX.X;XX.X | xx.x;xx.x | xx.x;xx.x |

SD: Standard deviation, Q1: 1st quartile, Q3: 3rd quartile.

The amount of IMP used for each subject is normalised by the number of days in the maintenance phase or number of days in remission, respectively.

Shell 93: Cumulative amount of investigational medical product used up to scheduled visits: maintenance phase safety analysis set

| | LEO 90100 | Vehicle |
|--------------------|------------|------------|
| | (n=xxx) | (n=xxx) |
| 7isit 3 | | |
| Number of subjects | XXX | xxx |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min;Max | xx.x;xx.x | xx.x; xx.x |
| ••• | | |
| Visit 15 | | |
| Number of subjects | XXX | xxx |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | XX.X;XX.X | xx.x;xx.x |



| Trial ID: LP0053-1004 | Date: 15-JUL-2019 | Version: 1.0 |
|-----------------------|-------------------|-----------------|

Shell 94: Serum-cortisol concentration at time 0 and at 30 and at 60 minutes after ACTH-challenge test by visit: open-label HPA analysis set

| | Open-label LEO 90100 |
|---------------------------------------|----------------------|
| | (n=xxx) |
| it 1 | |
| min (before ACTH-challenge test) | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min; Max | xx.x;xx.x |
| 0 min after ACTH-challenge test | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min; Max | xx.x; xx.x |
| 0 min after ACTH-challenge test | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | XX.X;XX.X |
| Min; Max | XX.X; XX.X |
| , | , |
| it 2 min (before ACTH-challenge test) | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | XX.X; XX.X |
| Min; Max | XX.X; XX.X |
| 1111,1101 | ^^,^,^^ |
| 0 min after ACTH-challenge test | |
| Number of subjects | XXX |
| Mean (SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | xx.x;xx.x |
| Min; Max | xx.x;xx.x |
| 0 min after ACTH-challenge test | |
| Number of subjects | XXX |
| Mean(SD) | xx.x(xx.x) |
| Median | XX.X |
| Q1;Q3 | XX.X;XX.X |
| Min; Max | XX.X;XX.X |



|------------------------------|-------------------|-----------------|

Shell 95: Individual data for subjects with serum cortisol concentration ≤18 mcg/dL at either 30 minutes or 60 minutes after ACTH-challenge: open-label HPA analysis set.

| | *** | Ourselle bine | Serum cortisol concentration | Change in serum cortisol concentration from time 0 | DG2 (0) |
|---|---|---|---|---|---|
| Subject | Visit | Sample time | (mcg/dL) | (mcg/dL) | BSA (%) |
| <subject id=""></subject> | Visit xx | 0 min | XX.X | | XX.X |
| | | 30 min | XX.X | XX.X | |
| | | 60 min | XX.X | XX.X | |
| | Visit xx | 0 min | XX.X | | XX.X |
| | | 30 min | XX.X | XX.X | |
| | | 60 min | XX.X | XX.X | |
| | | 0 1 | | | |
| <subject id=""></subject> | Visit xx | | XX.X | | XX.X |
| | | 30 min | XX.X | XX.X | |
| | | 60 min | XX.X | XX.X | |
| | Visit xx | 0 min | XX.X | | XX.X |
| | | 30 min | XX.X | XX.X | |
| | | 60 min | XX.X | XX.X | |



|------------------------------|-------------------|-----------------|

Shell 96: Subjects with serum cortisol concentration ≤18 mcg/dL at both 30 and 60 minutes after ACTH-challenge in open-label phase; open-label HPA analysis set

| | Open-label LEO 90100 |
|-----------------------------------------|------------------------|
| | (n=xxx) |
| Visit | |
| Serum Cortisol Concentration (mcg/dL) | Number of subjects (%) |
| Visit 1 | |
| 30 min after ACTH challenge test | |
| ≤18 mcg/dL | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) |
| Total | xx(xx.x) |
| 60 min after ACTH challenge test | |
| ≤18 mcg/dL | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) |
| Total | xx(xx.x) |
| 30 and 60 min after ACTH challenge test | |
| ≤18 mcg/dL | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) |
| Total | xx (xx.x) |
| Visit 2 | |
| 30 min after ACTH challenge test | |
| ≤18 mcg/dL | xx (xx.x) |
| >18 mcg/dL | xx(xx.x) |
| Total | xx(xx.x) |
| 60 min after ACTH challenge test | |
| ≤18 mcg/dL | xx (xx.x) |
| >18 mcg/dL | xx(xx.x) |
| Total | xx(xx.x) |
| 30 and 60 min after ACTH challenge test | |
| ≤18 mcg/dL | xx (xx.x) |
| >18 mcg/dL | xx(xx.x) |
| Total | xx(xx.x) |
| 10001 | 111 (111 · 11) |



|------------------------------|-------------------|-----------------|

Shell 97: Serum-cortisol concentration at time 0 and at 30 and at 60 minutes after ACTH-challenge test by visit: HPA analysis set

| ### Sit 8 ### Min (before ACTH-challenge test) Number of subjects | | All randomised subjects in the HPA axis group (n=xxx) | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|---|---|
| Number of subjects | ait 2 | | | |
| Number of subjects | | | | |
| Mean (SD) xx.x(xx.x) xx.x(xx. | _ | ***** | 171717 | 171717 |
| Median xx.x < | 3 | | | |
| Q1;Q3 | • • | , , | | |
| ### Min; Max | | | | |
| Number of subjects | | | | • |
| Number of subjects xxx | 20 min often ACMU challenge toot | · | · | · |
| Mean (SD) xx.x (xx.x) xx.x (xx.x) xx.x (xx.x) Median- xx.x xx.x x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x xx.x;xx.x Min;Max xx.x;xx.x xx.x | <del>_</del> | VVV | YYV | <b>**</b> |
| Median- xx.x xx.x xx.x Q1/Q3 xx.x,xxx.x xx.x,xxx.x xx.x,xxx.x Min;Max xx.x,xxx.x xx.x,xxx.x xx.x,xxx.x S0 min after ACTH-challenge test xxx xx.x xx.x Nedian xx.x xx.x xx.x xx.x Median xx.x xx.x xx.x xx.x Min;Max xx.x,xxx.x xx.x,xxx.x xx.x,xxx.x Sit 8 xx.x xx.x xx.x xx.x Number of subjects xx xx.x xx.x xx.x Median xx.x xx.x xx.x xx.x Median xx.x xx.x xx.x xx.x Min;Max xx.x,xxx.x xx.x,xxx.x xx.x,xxx.x 30 min after ACTH-challenge test xx xx xx.x xx.x Number of subjects xx xx.x xx.x xx.x Mean (SD) xx.x,xxxx xx.x xx.x xx.x Mean (SD) xx.x,xxxx | | | | |
| Q1;Q3 | | | | |
| Min; Max | | | | |
| Number of subjects | | | | |
| Number of subjects xxx xxx xxx xxx xxx xxxx xxx xxxx | • | | , | , |
| Mean (SD) xx.x (xx.x) xx.x (xx.x) xx.x (xx.x) xx.x x | <del>_</del> | VVV | VVV | ~~~ |
| Median xx.x < | _ | | | |
| Q1;Q3 | | | | |
| Min; Max xx.x;xx.x xx.x;xx.x xx.x;xx.x Sit 8 0 min (before ACTH-challenge test) xxx xxx.x xx.x | | | | |
| D min (before ACTH-challenge test) XXX < | | | | XX.X;XX.X |
| 0 min (before ACTH-challenge test) Number of subjects xxx | ai+ 0 | | | |
| Number of subjects xxx xxx xxx xxx xxx xxxx xxx | | | | |
| Mean(SD) xx.x(xx.x) xx.x(xx.x) xx.x(xx.x) Median xx.x xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x xx.x;xx.x Min;Max xxx xxx xxx xxx Mean(SD) xx.x(xx.x) xx.x(xx.x) xx.x(xx.x) Median xx.x xx.x xx.x xx.x Min;Max xx.x;xx.x xx.x;xx.x xx.x;xx.x xx.x;xx.x 60 min after ACTH-challenge test xxx xxx xxx xxx Number of subjects xxx xxx xxx xxx Mean(SD) xx.x(xx.x) xx.x(xx.x) xx.x(xx.x) Median xx.x xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x | | ~~~ | VVV | ~~~ |
| Median xx.x < | | | | |
| Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x xx.x;xx.x 30 min after ACTH-challenge test xxx xxx xxx Number of subjects xxx xx.x (xx.x) xx.x (xx.x) Mean (SD) xx.x (xx.x) xx.x (xx.x) xx.x (xx.x) Median xx.x (xx.x) xx.x;xx.x xx.x;xx.x Min;Max xx.x;xx.x xx.x;xx.x xx.x;xx.x 50 min after ACTH-challenge test xx xx xx Number of subjects xx xx xx xx Mean (SD) xx.x (xx.x) xx.x (xx.x) xx.x (xx.x) Median xx.x xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x | | | | |
| Min; Max xx.x; xx.x xx.x; xx.x xx.x; xx.x 30 min after ACTH-challenge test xxx xxx xxx Number of subjects xx.x (xx.x) xx.x (xx.x) xx.x (xx.x) Median xx.x xx.x xx.x xx.x Q1;Q3 xx.x; xx.x xx.x; xx.x xx.x; xx.x xx.x; xx.x Min; Max xx.x; xx.x xx.x; xx.x xx.x; xx.x xx.x; xx.x 50 min after ACTH-challenge test xxx xxx xxx xxx Number of subjects xxx xxx xx.x (xx.x) xx.x (xx.x) Median xx.x xx.x xx.x xx.x Q1;Q3 xx.x; xx.x xx.x; xx.x xx.x; xx.x | | | | |
| Number of subjects | | | | · |
| Number of subjects xxx xxx xxx xxx xxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxx xxx xxx xxx xxx xxx xxx xxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx xxxx <t< td=""><td>20</td><td></td><td></td><td></td></t<> | 20 | | | |
| Mean(SD) xx.x(xx.x) xx.x(xx.x) xx.x(xx.x) Median xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x Min; Max xx.x;xx.x xx.x;xx.x xx.x;xx.x 50 min after ACTH-challenge test xxx xxx xxx Number of subjects xxx xxx xxx Mean(SD) xx.x(xx.x) xx.x(xx.x) xx.x(xx.x) Median xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x | <del>_</del> | VVV | VVV | VVV |
| Median xx.x < | - | | | |
| Q1;Q3 xx.x;xx.x xx.x | | | | |
| Min; Max xx.x;xx.x xx.x;xx.x xx.x;xx.x 50 min after ACTH-challenge test xxx xxx xxx Number of subjects xxx xxx xxx Mean (SD) xx.x (xx.x) xx.x (xx.x) xx.x (xx.x) Median xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x | | | | |
| Mumber of subjects xxx xxx xxx Mean(SD) xx.x(xx.x) xx.x(xx.x) xx.x(xx.x) Median xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x | | | | |
| Number of subjects xxx xxx xxx Mean(SD) xx.x(xx.x) xx.x(xx.x) xx.x(xx.x) Median xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x | | 222 • 22 / 222 • 22 | 222 • 22 / 222 • 23 | 222 • 22 2222 • 22 |
| Mean (SD) xx.x(xx.x) xx.x(xx.x) xx.x(xx.x) Median xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x | | | | |
| Median xx.x xx.x xx.x Q1;Q3 xx.x;xx.x xx.x;xx.x xx.x;xx.x | 2 | | | |
| Q1;Q3 | | | | , , |
| | | XX.X | XX.X | XX.X |
| Min; Max xx.x; xx.x xx.x; xx.x xx.x; xx.x | | XX.X;XX.X | XX.X;XX.X | XX.X;XX.X |
| | Min; Max | XX.X;XX.X | XX.X;XX.X | XX.X;XX.X |



| Trial ID: LP0053-1004 | Date: 15-JUL-2019 | Version: 1.0 |
|-----------------------|-------------------|-----------------|

| | All randomised | LEO 90100<br>(n=xxx) | Vehicle |
|---|---|---|---|
| | subjects in<br>the HPA axis<br>group<br>(n=xxx) | | (n=xxx) |
| isit 15 | | | |
| 0 min (before ACTH-challenge test) | | | |
| Number of subjects | xxx | xxx | xxx |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| 01;03 | XX.X;XX.X | XX.X;XX.X | XX.X;XX.X |
| Min;Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| 30 min after ACTH-challenge test | | | |
| Number of subjects | XXX | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | xx.x |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| 60 min after ACTH-challenge test | | | |
| Number of subjects | XXX | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x | xx.x;xx.x |
| Min; Max | XX.X;XX.X | XX.X;XX.X | xx.x;xx.x |



| Trial ID: LP0053-1004 | Date: 15-JUL-2019 | Version: 1.0 |
|-----------------------|-------------------|-----------------|

Shell 98: Subjects with serum cortisol concentration ≤18 mcg/dL at both 30 and 60 minutes after ACTH-challenge in maintenance phase; HPA analysis set

| | All randomised subjects in the HPA axis group (n=xxx) | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|---|
| Visit<br>Serum Cortisol Concentration (mcg/dL | Number of subjects (%) | Number of subjects (%) | Number of subjects (%) |
| Visit 2 | | | |
| 30 min after ACTH challenge test | | | |
| ≤18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Total | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 60 min after ACTH challenge test | | | |
| ≤18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Total | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 30 and 60 min after ACTH challenge test | | | |
| ≤18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Total | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| <br>Visit 8 | | | |
| 30 min after ACTH challenge test | | | |
| ≤18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Total | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 60 min after ACTH challenge test | | | |
| ≤18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 30 and 60 min after ACTH challenge | | | |
| test | | | |
| ≤18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | • • | continued |



|------------------------------|-------------------|-----------------|

| | All randomised subjects in the HPA axis group (n=xxx) | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|---|
| isit | Number of | Number of | Number of |
| Serum Cortisol Concentrati | ion (mcg/dL) subjects (%) | subjects (%) | subjects (%) |
| isit 15 | | | |
| 30 min after ACTH challend | re test | | |
| ≤18 mcg/dL | xx (xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx (xx.x) | xx(xx.x) | xx(xx.x) |
| Total | xx (xx.x) | xx(xx.x) | xx(xx.x) |
| 60 min after ACTH challend | ge test | | |
| ≤18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Total | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| 30 and 60 min after ACTH o | challenge | | |
| est | | | |
| ≤18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >18 mcg/dL | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| >10 mcg/an | 2121 (2121 • 21) | () | ( |



|------------------------------|-------------------|-----------------|

Shell 99: Individual data for subjects with serum cortisol concentration ≤18 mcg/dL at either 30 minutes or 60 minutes after ACTH-challenge: HPA analysis set.

| Subject | Visit | Sample time | Serum cortisol concentration (mcg/dL) | Change in<br>serum cortisol<br>concentration<br>from time 0<br>(mcg/dL) | BSA (%) |
|---|---|---|---|---|---|
| | | <del>_</del> | | <del>-</del> | |
| | 771 - 1 | 0 | | | |
| <subject id=""></subject> | Visit XX | | XX.X | | XX.X |
| | | 30 min | XX.X | XX.X | |
| | | 60 min | XX.X | XX.X | |
| | Visit xx | 0 min | XX.X | | XX.X |
| | | 30 min | XX.X | XX.X | |
| | | 60 min | XX.X | XX.X | |
| <subject id=""></subject> | Visit xx | 0 min | XX.X | | XX.X |
| | | 30 min | XX.X | XX.X | |
| | | 60 min | XX.X | XX.X | |
| | Visit xx | 0 min | XX.X | | XX.X |
| | | 30 min | XX.X | XX.X | |
| | | 60 min | XX.X | XX.X | |



| Trial ID: LP0053-1004 | Date: 15-JUL-2019 | Version: 1.0 |
|-----------------------|-------------------|-----------------|

Shell 100: Serum-cortisol concentration at time 0 and at 30 and at 60 minutes after ACTH-challenge in the follow-up phase: HPA analysis set

| | All randomised subjects in the HPA axis group (n=xxx) | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|---|
| ollow-up visit 2 | | | |
| 0 min (before ACTH-challenge | | | |
| est) | | | |
| Number of subjects | XXX | XXX | XXX |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X | xx.x;xx.x |
| Min;Max | xx.x;xx.x | XX.X;XX.X | XX.X;XX.X |
| Number of subjects Mean(SD) Median- | xxx<br>xx.x(xx.x)<br>xx.x | xxx<br>xx.x(xx.x)<br>xx.x | xxx<br>xx.x(xx.x)<br>xx.x |
| 01;03 | XX.X;XX.X | xx.x;xx.x | XX.X;XX.X |
| Min;Max | XX.X;XX.X | XX.X;XX.X | XX.X;XX.X |
| 60 min often ACMU challenge | | | |
| 60 min after ACTH-challenge | | | |
| est | xxx | xxx | xxx |
| est<br>Number of subjects | XXX<br>XX.X(XX.X) | xxx<br>xx.x(xx.x) | xxx<br>xx.x(xx.x) |
| Number of subjects Mean(SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| est<br>Number of subjects | | | |



|------------------------------|-------------------|-----------------|

Shell 101: Summary of rebounds occurring within 2 months after discontinuing openlabel phase treatment or relapse treatment: safety analysis set

| | LEO 90100 | Vehicle |
|---------------------------------------|------------|------------|
| | (n=xxx) | (n=xxx) |
| Nithin 2 months after discontinuation | on of | |
| ppen-label treatment: | | |
| Number of rebounds | XXX | XXX |
| Number of subjects | XXX | xxx |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min;Max | xx.x;xx.x | xx.x;xx.x |
| Within 2 months after discontinuation | on of | |
| relapse treatment: | | |
| Number of rebounds | XXX | XXX |
| Number of subjects | XXX | XXX |
| Mean (SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | xx.x;xx.x |
| Min; Max | xx.x;xx.x | xx.x;xx.x |

Shell 102: Summary of rebounds occurring within 2 months after discontinuing of maintenance treatment: safety analysis set

| | LEO 90100<br>(n=xxx) | Vehicle<br>(n=xxx) |
|---|---|---|
| Within 2 months after discontinuation of | | |
| maintenance treatment: | | |
| Number of rebounds | XXX | XXX |
| Number of subjects | xxx | xxx |
| Mean(SD) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X |
| Q1;Q3 | xx.x;xx.x | XX.X;XX.X |
| Min; Max | xx.x;xx.x | xx.x;xx.x |



## Signature Page for TMF-000023733 v1.0

| Reason for signing: Approved | Manage | (s) |
|---|---|---|
| | Name: PPD | |
| | Capacit | |
| | Date of signature: 15-Jul-2019 08:57:51 GMT+0000 | |
| | - | |
| Reason for signing: Approved | Manage | dict(s) |
| | Name: PPD | |
| | Capacit | |
| | Date of signature: 15-Jul-2019 09:16:48 GMT+0000 | |
| Reason for signing: Approved | QC App | |
| | QC App<br>Name: PPD | |
| | Capacit | |
| | Date of signature: 15-Jul-2019 09:20:55 GMT+0000 | |

Electronic signatures made within eTMF LEO are considered to be a legally binding equivalent of traditional handwritten signatures.